CLINICAL STUDY PROTOCOL: SP-624-201 A

**Study Title:** 

A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Efficacy of SP-624 in the Treatment of Adults

with Major Depressive Disorder

**Sponsor:** Sirtsei Pharmaceuticals, Inc.

**Phase of Development:** Phase 2

NCT Number NCT04479852

**Protocol Number:** SP-624-201

Protocol Version: Amendment 3

**Protocol Version Number:** 4.0

Protocol Version Date: 26 May 2021

# CLINICAL STUDY PROTOCOL: SP-624-201

Study Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled

Study of the Safety and Efficacy of SP-624 in the Treatment of

Adults with Major Depressive Disorder

Study Drug: SP-624

IND Number:

**Sponsor:** Sirtsei Pharmaceuticals, Inc.

**Phase of Development:** Phase 2

**Protocol Number:** SP-624-201

**Protocol Version:** Amendment 3

**Protocol Version Number:** 4.0

**Protocol Version Date:** 26 May 2021

## **Version History**

| Version<br>Number | Version Date | Comment |
|-------------------|-------------------|-------------|
| 1.0 | 09 July 2020 | Original |
| 2.0 | 17 September 2020 | Amendment 1 |
| 3.0 | 27 January 2021 | Amendment 2 |
| 4.0 | 26 May 2021 | Amendment 3 |

## **CONFIDENTIALITY STATEMENT**

This protocol is the property of Sirtsei Pharmaceuticals, Inc. and is a confidential communication. Acceptance implies an agreement not to disclose information contained herein that is not otherwise publicly available, except for use by an institutional review board (IRB) for the purpose of obtaining approval to conduct the study. The IRB is requested and expected to maintain confidentiality. This document may not be used or published in whole or in part without the consent of Sirtsei Pharmaceuticals, Inc.

# INVESTIGATOR'S PROTOCOL AGREEMENT PAGE

Note: A signed copy of this page will be collected and filed in both the Sponsor and Investigator trial master files prior to the commencement of this study.

- I have read the SP-624-201 protocol and agree to conduct the study as outlined.
- I have received and read the Investigator's Brochure for SP-624.
- I agree to maintain the confidentiality of all information received or developed in connection with this protocol.
- I will personally oversee the conduct of this study as outlined herein and will make all reasonable efforts to complete the study within the time designated.
- I will provide all key study personnel under my supervision with copies of the protocol and access to all information provided by Sirtsei Pharmaceuticals, Inc.. I will discuss this material with them to ensure that they are fully informed about SP-624, the safety parameters, and the conduct of the study in general.
- I am aware that, before commencement of this study, the institutional review board responsible for such matters must approve this protocol in the clinical facility where it will be conducted.
- I agree to make all reasonable efforts to adhere to the attached protocol.
- I, or my designee, agree to be present at the site initiation visit. In addition, I will ensure the presence of all key study personnel under my supervision at this meeting.
- I agree to provide all subjects with informed consent forms, as required by government and International Council for Harmonisation regulations.
- I further agree to report to Sirtsei Pharmaceuticals, Inc. any adverse experiences in accordance with the terms of this protocol and Food and Drug Administration (FDA) regulation 21 Code of Federal Regulations (CFR) 312.64.

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| <br>Date |

# SPONSOR EMERGENCY CONTACT INFORMATION

## **Reporting of Serious Adverse Events (SAEs)**

Any SAE occurring in a study subject must be reported to the Sponsor within 24 hours.

See Section 8.1.2 (Serious Adverse Events) for definition and reporting procedure for SAEs.

All relevant information must be captured, preferably on an SAE Report Form, and submitted via email within 24 hours to each of the individuals listed in Table 1.

Request email confirmation of receipt, and if not confirmed, follow-up by phone to confirm receipt.

**Table 1:** Emergency Contact Information

| Role in Study | Name | Email Address | Telephone Number |
|----------------------------------|------|---------------|------------------|
| Sponsor Clinical Study<br>Leader | | | |
| Sponsor Medical Monitor | | | |

Sirtsei Pharmaceuticals, Inc. Protocol No: SP-624-201

Amendment 3

 Version: 4.0 – 26 May 2021

## PROTOCOL SYNOPSIS

## Name of Sponsor/Company:

Sirtsei Pharmaceuticals, Inc.

## Name of Investigational Product:

SP-624 (oral capsules)

## **Name of Active Ingredient:**

Code Name: SP-624

## Title of Study:

A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Efficacy of SP-624 in the Treatment of Adults with Major Depressive Disorder

## **Phase of development:**

Phase 2

### **Study center(s):**

Approxmiately 40 sites in the United States

### **Planned Study Duration:**

The planned study duration encompasses the estimated time from the Screening of the first subject to the estimated time the last subject completes the Week 6 Follow-Up Visit.

- Estimated date first subject Screened: September 2020
- Estimated date of last subject first visit: October 2021
- Estimated date of last subject last visit: November 2021

## **Objectives:**

## **Primary:**

• Evaluate the efficacy of SP-624 administered once-daily for up to 4 weeks compared to placebo in the treatment of adults with major depressive disorder (MDD)

### **Secondary:**

- Evaluate the safety and tolerability of SP-624 administered once-daily for up to 4 weeks compared to placebo in the treatment of adults with MDD
- Characterize the population pharmacokinetics (PK) of SP-624 in plasma when administered orally to subjects with MDD

Amendment 3

## **Study Design:**

This is a Phase 2, multicenter, double-blind, randomized, placebo-controlled study of the safety and efficacy of SP-624 in the treatment of adult subjects with MDD as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). Following the successful completion of a Screening Phase, subjects will be randomized to one of two treatment groups in a 1:1 ratio and will receive SP-624 or placebo over a treatment period of four weeks (Treatment Group #1: SP-624 20 mg/day; Treatment Group #2: Placebo).

Approximately 300 subjects (150 per treatment group) will be enrolled into the study. Each subject will complete Screening, Baseline, Treatment, and Follow-up Visits.

Prior to initiating the 4-week treatment period, subjects will complete a Screening/Baseline period of up to 28 days, during which time all Screening assessments will be performed, and any current depression medications discontinued. All Screening assessments should be completed before discontinuing any current depression medications. Subjects will return for a Baseline Visit to complete efficacy and safety assessments. During the treatment period, subjects will return to the investigative site to complete efficacy and safety assessments at the end of Weeks 1, 2, 3, and 4. After the final dose of study drug, subjects will complete a follow-up period of two weeks and will return at the end of Weeks 5 and 6. Subjects may be treated with anti-depressant medications according to physician recommendations after completion of the Week 5 Visit.

Unless there are any outstanding safety issues that require follow-up, subjects will be discharged from the study at the Week 6 Visit.

## **Number of subjects (planned):**

Approximately 300 adult subjects with MDD as defined by DSM-5; 150 subjects per treatment group at approximately 40 centers.

## **Duration of Subject Participation:**

Subjects will receive double-blind treatment for up to 4 weeks, following a Screening/Baseline period of up to 28 days. After the treatment period, subjects will complete a 2-week follow-up period. The planned study duration for each subject will be approximately 70 days.

Sirtsei Pharmaceuticals, Inc.


Protocol No: SP-624-201


Amendment 3

## Investigational Product, Dosage, and Mode of Administration:

Each dose of SP-624 will be supplied as two capsules, each containing 10 mg of active pharmaceutical ingredient (API). Matching placebo capsules identical in shape and color to the active capsules will also be used.

- Treatment Group #1: Two 10 mg capsules SP-624 each morning for 4 weeks
- Treatment Group #2: Two capsules placebo each morning for 4 weeks

If the two capsule dose is not well tolerated, the dose can be decreased to one capsule per dose after Week 1.

Study drug will be packaged in weekly blister cards (Weeks 1-4 of dosing), with each blister card containing 20 capsules of study drug (two capsules per dose for seven days of dosing, plus three extra days of dosing as a provision for study visit scheduling). Weekly blister cards will be assembled in subject kits containing four blister cards for use during the treatment period. Each kit will be labeled with a 3-part label that specifies the randomization number, cautionary statement, and storage conditions. Each blister card will have a one-part label that specifies the randomization number, week, number of capsules, cautionary statement, and storage conditions.

Each study drug dose should be taken orally, once daily at approximately the same time each morning. Study drug doses should be taken on an empty stomach before breakfast, and no food should be consumed for at least 1 hour after dosing. High fat foods at breakfast (e.g., bacon, cheese, eggs, etc.) should be avoided. Morning liquids such as coffee or tea are allowed without any additives (eg, cream, sugar, etc).

If dosing on an empty stomach is not practical or not well tolerated, then a low fat, low calorie breakfast 2 hours before dosing, or 30-60 minutes after dosing, is acceptable. If dosing remains not well tolerated, then subjects should dose 30 minutes after a low fat, low calorie meal.

## **Inclusion Criteria:**

To be eligible for this study, a subject must meet all of the following inclusion criteria:

- 1. Willing and able to provide written informed consent to participate in the study.
- 2. Males and females, aged 18 to 65 years, inclusive.
- 3. In generally good physical health, in the opinion of the Investigator.
- 4. Body mass index (BMI) must be  $\geq 18$  and  $\leq 40 \text{ kg/m}^2$
- 5. Females of reproductive potential and males with partners of reproductive potential must agree to remain abstinent or use adequate and reliable contraception throughout the study and for at least 30 days after the last dose of study drug.
  - a. Adequate contraception is defined as continuous use of double-barrier method (e.g., condom and spermicide or diaphragm and spermicide), oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, or intrauterine device.
  - b. Non-reproductive potential is defined as surgically sterile, undergone tubal ligation or vasectomy, or postmenopausal (defined as at least 12 months of spontaneous amenorrhea).
  - c. Subjects of reproductive potential but whose <u>sole</u> partner is of non-reproductive potential, or whose <u>sole</u> partner is of the same sex, are not required to maintain abstinence or contraception.

Sirtsei Pharmaceuticals, Inc.


Amendment 3

d. Subjects must agree to refrain from sperm and oocyte donation for at least 90 days after the last dose of study drug.

- 6. Meets DSM-5 criteria for moderate to severe MDD, as confirmed by the Mini International Neuropsychiatric Interview (MINI). Subjects with a diagnosis of co-morbid generalized anxiety disorder (GAD) may be included if MDD is the primary diagnosis.
- 7. Montgomery-Asberg Depression Rating Scale (MADRS) total score ≥ 27 at both Screening and Baseline.
- 8. History of inadequate or non-response to at least one adequate treatment, but no more than three of the same class of antidepressant, (i.e., an adequate dose for at least six weeks) for the current episode, in the opinion of the Investigator. NOTE: If immediately prior to this episode starting, treatment was working to the point of remission, but then the depression worsened, subject should not be enrolled. For example, subject should not have been on an antidepressant and in remission prior to the start of the current episode.
- 9. Willing and able to comply with the study design schedule and other requirements.

### **Exclusion Criteria:**

A subject who meets any of the following exclusion criteria will not be enrolled in the study:

- 1. Female who is pregnant, breastfeeding, or less than six months postpartum at Screening.
- History or presence of major bowel resection, total gastrectomy, or diabetes, and/or history or
  presence of any clinically significant medical condition, disease, or surgical history that
  could, in the opinion of the Investigator, jeopardize the safety of the subject or validity of the
  study data, or interfere with the absorption, distribution, metabolism, or excretion of the study
  drug.
- 3. A current DSM-5 diagnosis of depression with peripartum onset, panic disorder, obsessive compulsive disorder, post-traumatic stress disorder, anorexia nervosa, or bulimia nervosa.
- 4. A history of or current DSM-5 diagnosis of MDD with psychotic features, any schizophrenia spectrum and other psychotic disorders, bipolar disorder, or personality disorder.
- 5. History of treatment with electroconvulsive therapy (ECT), vagus nerve stimulation, deep brain stimulation, or transcranial magnetic stimulation within six months of Screening.
- 6. Current episode of depression exceeds 2 years or is less than six weeks from Screening.
- 7. History of inadequate or non-response, in the opinion of the Investigator, to an adequate treatment regimen of two or more classes of antidepressants during the current episode.
- 8. Subjects treated with an antipsychotic during the current episode should be excluded.
- 9. Subjects who meet DSM-5 criteria for moderate or severe substance use disorder for any substance except nicotine or caffeine, within 12 months of Screening. Subjects with a urine drug screen positive for suspected substance of abuse will be excluded. Urine drug screen positive for cannabinoids is not exclusionary if the subject does not meet criteria for moderate or severe substance use disorder.
- 10. Will require initiation of psychotherapy during the study period, in the Investigator's opinion. If a subject has been in ongoing psychotherapy for a minimum of three months, the therapy may continue if it remains unchanged. Cognitive behavioral therapy is excluded.

Sirtsei Pharmaceuticals, Inc.


Amendment 3

11. Poses a current or future suicidal risk, in the Investigator's opinion, or has a history of suicidal behavior within the past 12 months, and/or subject answers "yes" to "Suicidal Ideation" Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the Columbia-Suicide Severity Rating Scale (C-SSRS) assessment during the six months prior to the Screening period and/or at Baseline.

- 12. Failure to discontinue all psychoactive medications or psychoactive supplements including antidepressants and mood stabilizers, within a time period prior to Baseline corresponding to at least five half-lives of the medication in question.
- 13. Presence of a clinically significant abnormality on physical examination or electrocardiogram (ECG), including a corrected QT interval using Fridericia's formula (QTcF) >450 msec for males and >470 msec for females. Note: ECG may be repeated once at both Screening and Baseline for confirmatory purposes.
- 14. Presence or history of any known clinically significant cardiovascular disorders including, but not limited to: coronary artery disease, heart failure, valvular heart disease, cardiomyopathies, myocardial infarction, chamber enlargement or hypertrophy, or orthostatic hypotension.
- 15. Presence of uncontrolled hypertension, defined as consistent systolic blood pressure (SBP) >160 mmHg or consistent diastolic blood pressure (DBP) >95 mmHg despite present therapy. Note: Blood pressure measurements may be repeated twice at both Screening and Baseline for confirmatory purposes.
- 16. Screening laboratory value(s) outside the laboratory reference range that are considered to be clinically significant by the Investigator (clinical chemistry, hematology, coagulation, and urinalysis). Note: Screening labs may be repeated once for confirmatory purposes.
- 17. Screening liver function tests (ALT, AST, Alkaline phosphatase) > 2x the upper limit of normal
- 18. Known history of current or chronic Hepatitis B or Hepatitis C infection, or a known history of human immunodeficiency virus (HIV) infection. Subjects with a history of treated Hepatitis C infection where liver function tests are within normal limits may participate.
- 19. Subjects with a history of seizures or seizure disorder.

  Note: Subjects with a history of only febrile seizures, limited to up to two episodes, are permitted.
- 20. Clinically significant acute infection, other than mild viral or bacterial infections from which the subject has fully recovered (e.g., common cold, localized skin infection, etc.), within the two weeks prior to Baseline.
- 21. Major trauma or surgery in the 12 weeks prior to Screening or at any time between Screening and randomization.
- 22. Presence or history of malignancy within the last five years. Note: History of adequately treated basal cell or squamous cell carcinoma of the skin or in situ cervical cancer is allowed.
- 23. History of an anaphylactic allergic reaction to previous medication.
- 24. Blood or plasma donation within 30 days of randomization, or planned donations or elective surgery during the study or during the 60 days following the study.
- 25. Subjects who, in the opinion of the Investigator, are not suitable candidates for the study.

Amendment 3

26. Individuals who are currently enrolled in or have participated in a clinical trial (i.e., received study drug) involving an investigational product within 60 days or within five half-lives of the investigational product (whichever is longer) prior to Baseline.

## **Study Endpoints:**

## **Primary Efficacy Endpoint:**

• Change from Baseline to Week 4 in MADRS total score

## **Secondary Efficacy Endpoints:**

- Change from Baseline to Weeks 1, 2, and 3 in MADRS total score
- Change from Baseline to Weeks 1, 2, 3, and 4 in Clinical Global Impression Severity (CGI-S) total score
- Change from Baseline to Week 5 and change from Week 4 to Week 5 in MADRS total score and CGI-S total score
- Change from Baseline to Week 2 and Week 4 in the 17-item Hamilton Depression Rating Scale (HAM-D-17) total score
- Change from Baseline to Week 2 and Week 4 in the Sheehan Disability Scale (SDS)
- Change from Baseline to Week 2 and Week 4 in the Quick Inventory of Depressive Symptomology Self Report (QIDS-SR)
- Change from Baseline to Week 2 and Week 4 in the Quality of Life Enjoyment and Satisfaction Questionnaire – Short Form (Q-LES-Q-SF)

## **Safety Endpoints:**

- Adverse Events (AEs)
- Clinical safety laboratory tests (serum chemistry [including thyroid function], hematology, coagulation, and urinalysis tests)
- Vital signs (blood pressure, pulse rate, and oral body temperature)
- Body weight
- 12-lead ECGs
- Physical examinations
- C-SSRS

## **PK Endpoints:**

A total of four blood samples will be collected from each subject for the measurement of plasma concentrations of SP-624 at the following visits:

- Visit 2 (Day -1)
- Visit 3 (Week 1): Pre-Dose
- Visit 4 (Week 2): Pre-Dose or approximately 2 to 10 hours post-dose (whichever is more convenient for the subject)

Sirtsei Pharmaceuticals, Inc.


Amendment 3

• Visit 6 (Week 4): approximately 2 to 10 hours post-dose

If a subject missed the dose the day before a scheduled "pre-dose" sample collection, study personnel should instead collect a post-dose sample at that visit. Should a subject inadvertently dose prior to a scheduled "pre-dose" sample collection at Week 1 or Week 2, study personnel should collect a post-dose sample.

In the event that samples cannot be conveniently collected for a given subject according to the scheduled sampling times specified above, study personnel should attempt to collect at least one predose sample and at least one post-dose sample during the course of the study.

Date and time of most recent dose prior to PK sample collection, date and time of PK sample collection, and meal information relative to most recent dose, will be recorded on days of PK sample collection.

Plasma samples will be analyzed for SP-624 concentration using a validated bioanalytical method.

An aliquot of each subject's post-dose samples may be used by the bioanalytical laboratory for metabolite profiling. Potential metabolites will be identified using mass spectrometry techniques; and if conducted, these data will be summarized in a separate bioanalytical report.



## **Statistical Methods and Sample Size Justification:**

## **Analysis Populations:**

Within each population, analyses will be performed comparing subjects and by-treatment assignment (SP-624 vs placebo).

- All Subjects Population all subjects who sign informed consent and are assigned a unique subject identification number. This population will be used to summarize disposition.
- Modified Intent-to-Treat (mITT) Population all subjects who are randomized to receive
  treatment, receive at least one dose of study drug, and have a Baseline and at least one
  post-dose efficacy assessment. This population will be the primary population used to
  summarize demographics, baseline characteristics, medical history, treatment history, and
  all efficacy outcomes. Subjects will be analyzed according to randomized treatment
  group.
- Per Protocol (PP) Population All subjects in the mITT population who received assigned study drug as randomized, completed the Week 4 assessments without any major protocol violations, and have 75-125% compliance. The PP population will be used as an additional population for summaries of efficacy outcomes.

- Safety Population all subjects in the mITT population who receive at least one dose of study drug. Safety subjects will be summarized according to the treatment they actually received. This population will be used to summarize all safety assessments.
- PK Population all subjects who receive active study drug and have evaluable PK data based on actual treatment received, protocol compliance, adequate numbers of samples, and successful sample assays.

## **Sample Size Justification:**

Recent studies of MDD using change from Baseline in MADRS total scores suggest that placebo will yield an approximately nine unit decrease over four weeks with a standard deviation (SD) of around 9.2. SP-624 is expected to yield at least a 12 unit decrease in MADRS total score over four weeks with a similar SD of around 9.2. A minimum of 150 subjects per treatment arm (300 total) would be needed to detect a treatment difference of three units with 80% statistical power. The sample size was estimated using NQuery 8 (V8.5.2.0) two group test of equal means (MTT0-1: www.statsols.com).

## **Efficacy:**

The primary efficacy variable is change from Baseline in MADRS total score at Week 4, for testing superiority of SP-624 vs. placebo. This variable will be analyzed using a Mixed Model for Repeated Measures (MMRM), with change from Baseline in MADRS total score at each visit as the response variable. The MMRM model will include age, weight, and baseline MADRS total score as covariates, with factors for treatment, visit (Weeks 1, 2, 3, and 4; as a categorical variable), treatment by visit interaction term, gender, and site as a fixed effect. An unstructured covariance matrix will be used for the within-subject correlation. Kenward-Rogers approximation will be used to calculate the denominator degrees of freedom. The primary efficacy endpoint will be calculated using an estimate statement. Subjects from low enrolling sites may be pooled in order to help with model convergence. In the event of a model which fails to converge, analysis strategies will be detailed in the statistical analysis plan (SAP) which will be used to complete the analysis of the primary endpoint. This will include different model assumptions (e.g., restricted maximum likelihood vs maximum likelihood, covariance structure, and removing variables from the model [especially if they are associated with a high degree of missing values]).

### Safety:

Laboratory parameters, vital sign data, and ECG results will be summarized by treatment group and presented in tabular and graphic formats where appropriate. Appropriate change from Baseline calculations will be provided to detect any significant changes in laboratory parameters, vital sign values, ECG results, and C-SSRS results, but no formal statistical tests are planned.

### **Pharmacokinetic Assessments:**

Plasma concentration data for SP-624 will be listed and summarized using descriptive statistics. If data allow, results will be used for other analyses (e.g., PopPK) which will be presented in a separate report.

The population PK analysis of SP-624 will be performed using a nonlinear mixed effects model (NONMEM). This analysis will provide estimates of population PK parameters such as CL/F, Vz/F, etc. and a measure of their variability. Pharmacokinetic parameters of individual subjects (e.g., AUC[0-tau], Cavg, Cmax) may be estimated and their correlation with relevant covariates (e.g., body weight, gender, concomitant medications) will be explored. The population PK analysis plan will be prepared separately.

Plasma concentration data will remain blinded until the unblinding of the clinical database at the end of the study.

# **SCHEDULE OF EVENTS**

**Table 2:** Schedule of Events

| Study Period | Screening /<br>Washout | Baseline | Treatment Period | | | | Follow-up Period | |
|---|---|---|---|---|---|---|---|---|
| Study Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
| Study Day / Week | Day<br>-28 to -2 | Day -1 | Week 1<br>(Day 7 ± 3<br>days) | Week 2<br>(Day 14 ± 3<br>days) | Week 3<br>(Day 21 ± 3<br>days) | Week 4 /<br>Prema-<br>ture D/C<br>(Day 28 ± 3<br>days) | Week 5<br>(7 days ±3<br>days post<br>Week 4<br>Visit) | Week 6<br>(14 days<br>±3 days<br>post<br>Week 4<br>Visit) |
| <b>Event/Assessment</b> | | | | | | | | |
| Clinic Visit <sup>1</sup> | X | X | X | X | X | X | X | X |
| Informed Consent | X | | | | | | | |
| Inclusion/Exclusion | X | X | | | | | | |
| Diagnosis Confirmation and<br>Treatment History | X | | | | | | | |
| Demographics, Medical History | X | X | | | | | | |
| Height and Weight <sup>2</sup> | X | X | | | | X | | |
| Physical Exam <sup>3</sup> | X | X | X | X | X | X | X | |
| C-SSRS <sup>4</sup> | X | X | X | X | X | X | X | X |
| Pregnancy Test <sup>5</sup> | X | X | | | | X | | |
| Urine Drug Screen | X | | | | | | | |
| Clinical Safety Labs <sup>6</sup> | X | X | | X | | X | X | |
| Vital Signs <sup>7</sup> | X | X | X | X | X | X | X | X |
| 12-Lead ECG <sup>8</sup> | X | X | X | X | X | X | X | |
| MADRS | X | X | X | X | X | X | X | |
| CGI – S | X | X | X | X | X | X | X | |
| HAM-D, SDS, QIDS-SR; Q-<br>LES-Q-SF | | X | | X | | X | | |
| Randomization | | X | | | | | | |
| Dispensation / Collection /<br>Accountability of Study Drug | | X | X | X | X | X | | |
| Plasma PK Blood Sampling | | X | X | X | | X | | |
| Prior and Con Med Record | X | X | X | X | X | X | X | X |
| AE Monitoring | X | X | X | X | X | X | X | X |


Abbreviations: AE=adverse event; con med=concomitant medication; CGI-S=clinical global impression-severity; C-SSRS=Columbia-Suicide Severity Rating Scale; ECG=electrocardiogram; MADRS=Montgomery-Asberg Depression Rating Scale; PK=pharmacokinetics; Premature D/C=Premature Discontinuation from treatment; QIDS-SR=Quick Inventory of Depressive Symptomology – Self Report; Q-LES-Q-SF=Quality of Life Enjoyment and Satisfaction Questionnaire – Short Form; SDS=Sheehan Disability Scale

- <sup>1</sup> If a clinic visit is not possible (e.g., due to illness), a remote visit may be conducted to complete all assessments that can be done remotely and assess for adverse events and concomitant medications. The Screening, Baseline, and Week 4/Premature Discontinuation Visits cannot be done remotely. The sponsor should be contacted prior to conducting any remote visits whenever possible.
- <sup>2</sup> Height and body weight at Visit 1. Body weight only at Visit 2 and Visit 6/Premature Discontinuation.
- <sup>3</sup> Physical examinations will include a review of the following body systems: general appearance, skin and extremities, ear/eyes/nose/throat, head/neck, heart/chest, abdomen, musculoskeletal, and neurological.
- <sup>4</sup> Baseline/Screening Version at Visit 1; Since Last Visit Version at Visits 2-8.
- <sup>5</sup> All females; Serum pregnancy test at Visit 1 and Visit 6 (or Premature Discontinuation); Urine pregnancy test at Visit 2 if urine pregnancy test at Visit 2 is positive, a confirmatory serum pregnancy test will be conducted.
- <sup>6</sup> Clinical safety labs include clinical chemistry, hematology, coagulation, and urinalysis. Labs should be collected in a fasting state. Urinalysis not required at Visit 4 (Week 2 visit).
- <sup>7</sup> Vital signs include blood pressure, pulse rate, and oral body temperature. Vital signs to be assessed in a sitting position after three mins or more of quiet sitting.
- 8 Two ECGs to be collected at the Baseline Visit separated by approximately 10 minutes. One ECG collected at all other visits.

# TABLE OF CONTENTS

| TITLE P. | AGE | 1 |
|----------|------------------------------------------------|----|
| INVEST | IGATOR'S PROTOCOL AGREEMENT PAGE | 2 |
| SPONSO | R EMERGENCY CONTACT INFORMATION | 3 |
| PROTOC | COL SYNOPSIS | 4 |
| SCHEDU | JLE OF EVENTS | 12 |
| TABLE ( | OF CONTENTS | 14 |
| 1. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 21 |
| 2. | INTRODUCTION | 25 |
| 2.1. | Major Depressive Disorder | 25 |
| 2.2. | Investigational Product | 25 |
| 2.2.2. | Non-clinical Studies. | 26 |
| 2.2.3. | Clinical Studies | 27 |
| 2.2.3.1. | SP-624-101 | 27 |
| 2.2.3.2. | SP-624-102 | 28 |
| 2.3. | SP-624 Development Plan | 29 |
| 2.3.1. | Rationale for Dose | 29 |
| 2.3.2. | Benefit and Risk Assessment. | 29 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 31 |
| 3.1. | Objectives | 31 |
| 3.1.1. | Primary Objective | 31 |
| 3.1.2. | Secondary Objectives | 31 |
| 3.2. | Endpoints | 31 |
| 3.2.1. | Efficacy Endpoints | 31 |
| 3.2.1.1. | Primary Endpoint | 31 |
| 3.2.1.2. | Secondary Endpoints | 31 |
| 3.2.2. | Safety Endpoints | 31 |
| 3.2.3. | Pharmacokinetic Endpoints | 32 |
| 3.2.4. | | |
| 1 | INVESTIGATIONAL DI AN | 22 |

| 4.1. | Overall Study Design | 33 |
|---|---|---|
| 4.1.1. | Screening Period and Baseline Visit | 33 |
| 4.1.2. | Treatment and Follow-up Periods | 33 |
| 4.2. | Randomization and Blinding | 35 |
| 4.2.1. | Subject Identification and Randomization to Treatment | 35 |
| 4.2.2. | Blinding | 35 |
| 4.2.3. | Emergency Unblinding | 35 |
| 4.3. | Study Centers and Personnel | 35 |
| 4.4. | Number of Subjects | 36 |
| 4.5. | Study Duration | 36 |
| 5. | SELECTION AND WITHDRAWAL OF SUBJECTS | 37 |
| 5.1. | Subject Recruitment, Enrollment, and Identification | 37 |
| 5.2. | Subject Inclusion Criteria | 37 |
| 5.3. | Subject Exclusion Criteria | 38 |
| 5.4. | Subject Withdrawal from the Study | 40 |
| 5.5. | Premature Termination of the Study | 40 |
| 6. | STUDY TREATMENTS, MATERIALS, AND MANAGEMENT | 41 |
| 6.1. | Description of Study Drug | 41 |
| 6.2. | Acquisition of Study Drug Supplies | 41 |
| 6.3. | Subject Treatment Assignment | 41 |
| 6.4. | Study Drug Administration. | 41 |
| 6.5. | Treatment Compliance | 42 |
| 6.6. | Study Drug Accountability | 42 |
| 6.7. | Study Drug Storage and Stability | 43 |
| 6.8. | Prior and Concomitant Medications | 43 |
| 7. | STUDY PROCEDURES AND ASSESSMENTS | 46 |
| 7.1. | Schedule of Events | 46 |
| 7.2. | Study-Specific Procedures | 46 |
| 7.2.1. | Informed Consent | 46 |
| 7.2.2. | Demographic Information, Medical History/Current Medical Conditions, and Treatment History | 46 |
| 7.2.3. | Mini International Neuropsychiatric Interview | 47 |

| 7.2.4. | Assessment of Efficacy | 47 |
|---|---|---|
| 7.2.4.1. | Montgomery-Asberg Depression Rating Scale | 47 |
| 7.2.4.2. | Clinical Global Impression – Severity | 47 |
| 7.2.4.3. | Hamilton-Depression Rating Scale (17-item) | 47 |
| 7.2.4.4. | Sheehan Disability Scale | 48 |
| 7.2.4.5. | Quick Inventory of Depressive Symptomology – Self Report | 48 |
| 7.2.4.6. | Quality of Life Enjoyment and Satisfaction Questionnaire – Short Form | 48 |
| 7.2.5. | Assessment of Safety | 48 |
| 7.2.5.1. | Physical Examination | 48 |
| 7.2.5.2. | Vital Signs, Height, and Weight Measurements | 49 |
| 7.2.5.3. | 12-lead Electrocardiograms | 49 |
| 7.2.5.4. | Pregnancy Test | 49 |
| 7.2.5.5. | Clinical Safety Laboratory Assessments | 50 |
| 7.2.5.6. | Blood Volume Collection Summary | 50 |
| 7.2.5.7. | Columbia-Suicide Severity Rating Scale | 53 |
| 7.2.6. | Assessment of Pharmacokinetics | 53 |
| 7.2.6.1. | Pharmacokinetics | 53 |
| 7.2.6.2. | | 54 |
| 7.2.7. | Biological Sample Retention and Destruction | 54 |
| 8. | ADVERSE EVENTS, SERIOUS ADVERSE EVENTS, AND OTHER REPORTABLE EVENTS | 55 |
| 8.1. | Adverse Events | 55 |
| 8.1.1. | Clinical Safety Assessment Abnormalities | 55 |
| 8.1.2. | Serious Adverse Event (SAE) | 55 |
| 8.1.3. | Suspected and Unexpected Serious Adverse Reactions | 56 |
| 8.1.4. | Evaluation of Adverse Events | 56 |
| 8.1.4.1. | Adverse Event Term/Diagnosis | 56 |
| 8.1.4.2. | Date and Time of Adverse Event Onset and Resolution | 57 |
| 8.1.4.3. | Relationship to Study Drug | 57 |
| 8.1.4.4. | Intensity Categorization | 57 |
| 8.1.4.5. | Action Taken for Adverse Event | 58 |
| 8.1.4.6. | Outcome of Adverse Event. | 58 |

| 8.1.5. | Reporting of Serious Adverse Events | 59 |
|---|---|---|
| 8.1.6. | Other Reportable Events | 60 |
| 9. | STATISTICS | 61 |
| 9.1. | Determination of Sample Size | 61 |
| 9.2. | Analysis Populations | 61 |
| 9.3. | Description of Statistical Methods | 62 |
| 9.3.1. | General Approach | 62 |
| 9.3.2. | Interim Analysis. | 62 |
| 9.3.3. | Summary of Demographics, Baseline Characteristics, Medical History, and Treatment History | 62 |
| 9.3.4. | Summary of Efficacy | 62 |
| 9.3.4.1. | Primary Efficacy Endpoint Analysis | 62 |
| 9.3.4.2. | Secondary Efficacy Endpoint Analysis | 63 |
| 9.3.5. | Sensitivity Analyses | 64 |
| 9.3.6. | Summary of Pharmacokinetics | 64 |
| 9.3.7. | | 65 |
| 9.3.8. | Concomitant Medications | 65 |
| 9.3.9. | Summary of Safety and Tolerability | 65 |
| 9.3.9.1. | Adverse events | 65 |
| 9.3.9.2. | Vital Signs and ECGs | 66 |
| 9.3.9.3. | Clinical Laboratory Assessments | 66 |
| 9.3.9.4. | Physical Exams | 66 |
| 9.3.9.5. | C-SSRS | 66 |
| 10. | SPONSOR'S AND INVESTIGATOR'S RESPONSIBILITIES | 67 |
| 10.1. | Sponsor's Responsibilities | 67 |
| 10.2. | Investigator's Responsibilities | 67 |
| 11. | ETHICS | 68 |
| 11.1. | Ethical Conduct of the Study | 68 |
| 11.2. | Ethics Review | 68 |
| 11.3. | Written Informed Consent | 68 |
| 12. | DATA HANDLING AND RECORD KEEPING | 69 |
| 12.1. | Data Collection and Recording. | 69 |

| 12.2. | Retention of Records | 69 |
|---|---|---|
| 12.3. | Protocol Deviations | 69 |
| 12.4. | Publication Policy | 69 |
| 12.5. | Data Quality Assurance | 70 |
| 12.6. | Data Management | 70 |
| 13. | LIST OF REFERENCES | 71 |
| 13.1. | Publications Referenced | 71 |
| 13.2. | Sponsor Documents and Study Reports Referenced | 71 |
| 13.2.1. | Investigator's Brochure | 71 |
| 13.2.2. | Pharmacology Studies | 71 |
| 14. | APPENDICES | 72 |
| APPENDI | X A. MONTGOMERY-ASBERG DEPRESSION RATING SCALE | 73 |
| APPENDI | X B. CLINICAL GLOBAL IMPRESSION – SEVERITY | 77 |
| APPENDI | X C. 17-ITEM HAMILTON DEPRESSION RATING SCALE | 78 |
| APPENDI | X D. SHEEHAN DISABILITY SCALE | 83 |
| APPENDI | X E. THE QUICK INVENTORY OF DEPRESSIVE SYMPTOMOLOGY – SELF REPORT | 85 |
| APPENDI | X F. QUALITY OF LIFE ENJOYMENT AND SATISFACTION QUESTIONNAIRE – SHORT FORM | 87 |
| APPENDI | X G. COLUMBIA – SUICIDE SEVERITY RATING SCALE – BASELINE/SCREENING VERSION | 89 |
| APPENDI | X H. COLUMBIA – SUICIDE SEVERITY RATING SCALE – SINCE<br>LAST VISIT VERSION | 92 |

# LIST OF TABLES


| Table 1: | Emergency Contact Information | 3 |
|---|---|---|
| Table 2: | Schedule of Events | 12 |
| Table 3: | Abbreviations | 21 |
| Table 4: | Restricted and Prohibited Medications | 44 |
| Table 5: | Clinical Safety Laboratory Analytes | 51 |
| Table 6: | Estimation of Blood Volumes Required from Screening through the End of the Follow-up Period | 50 |
| | the ronow up remod | |

| Sirtsei Pharmaceuticals, Inc. |
|-------------------------------|
| Amendment 3 |


# LIST OF FIGURES

| Figure 1: | Study Schematic | 34 | ļ |
|-----------|-----------------|----|---|
| _ | | | |

# 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

The following abbreviations and terms are used in this study protocol.

**Table 3:** Abbreviations

| Abbreviation | Explanation |
|---|---|
| AE | Adverse event |
| ALT | Alanine aminotransferase |
| ANCOVA | Analysis of covariance |
| API | Active pharmaceutical ingredient |
| AST | Aspartate aminotransferase |
| AUC | Area under the plasma concentration-time curve |
| AUC[0-tau] | Area under the plasma concentration-time curve during the 24-hour dosing interval |
| BMI | Body mass index |
| BOCF | Baseline observation carried forward |
| bpm | Beats per minute |
| BUN | Blood urea nitrogen |
| С | Celsius |
| Cavg | Average plasma concentration |
| CBC | Complete blood count |
| CFR | Code of Federal Regulations |
| CGI-S | Clinical Global Impression – Severity |
| CL/F | Apparent systemic clearance |
| CLss/F | Apparent systemic clearance after oral dosing at steady state |
| cm | Centimeter(s) |
| Cmax | Observed maximum serum concentration |
| CRF | Case report form |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| DBP | Diastolic blood pressure |
| DMP | Data management plan |
| DNA | Deoxyribonucleic acid |
| DSM-5 | Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition |
| ECG | Electrocardiogram |

| Abbreviation | Explanation |
|--------------|----------------------------------------------|
| ECT | Electroconvulsive therapy |
| eGFR | Estimated glomerular filtration rate |
| FCS | Fully conditional specification |
| FDA | Food and Drug Administration |
| g | Gram(s) |
| GAD | Generalized anxiety disorder |
| GCP | Good Clinical Practice |
| GGT | Gamma-glutamyltransferase |
| GLP | Good Laboratory Practice |
| GMP | Good Manufacturing Practice |
| h | Hour(s) |
| HAM-D-17 | 17-item-Hamilton Depression Rating Scale |
| hCG | Human chorionic gonadotropin |
| HED | Human equivalent dose |
| HDL | High-density lipoprotein |
| HIV | Human immunodeficiency virus |
| ICF | Informed consent form |
| ICH | International Council for Harmonisation |
| IND | Investigational New Drug |
| INR | International normalized ratio |
| IRB | Institutional Review Board |
| LDH | Lactate dehydrogenase |
| LDL | Low-density lipoprotein |
| LOCF | Last observation carried forward |
| LTFU | Lost to follow up |
| MADRS | Montgomery-Asberg Depression Rating Scale |
| MAR | Missing at random |
| MCH | Mean corpuscular hemoglobin |
| MCHC | Mean corpuscular hemoglobin concentration |
| MCV | Mean cell volume |
| MDD | Major depressive disorder |
| MedDRA | Medical Dictionary for Regulatory Activities |

| Abbreviation | Explanation |
|---|---|
| mg | Milligram(s) |
| mL | Milliliter(s) |
| mm | Millimeter(s) |
| min | Minutes |
| MINI | Mini International Neuropsychiatric Interview |
| mITT | Modified intent-to-treat |
| MMRM | Mixed model for repeated measures |
| MNAR | Missing not at random |
| MPV | Mean platelet volume |
| MVN | Multivariate normal distribution |
| NAD+ | Nicotinamide-adenine dinucleotide coenzyme |
| ng | Nanogram(s) |
| NONMEM | Nonlinear mixed effects model |
| PI | Principal Investigator |
| PK | Pharmacokinetic(s) |
| PP | Per protocol |
| PT | Prothrombin time |
| PTT | Partial thromboplastin time |
| QA | Quality assurance |
| QIDS-SR | Quick Inventory of Depressive Symptomology – Self-Report |
| Q-LES-Q-SF | Quality of Life Enjoyment and Satisfaction Questionnaire – Short Form |
| QTcF | Corrected QT interval using Fridericia's formula |
| RBC | Red blood cells |
| RDW | Red cell distribution width |
| REML | Restricted maximum likelihood |
| RNA | Ribonucleic acid |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SBP | Systolic blood pressure |
| SD | Standard deviation |
| SDS | Sheehan Disability Scale |

 Version: 4.0 – 26 May 2021 Amendment 3

| Abbreviation | Explanation |
|--------------|-----------------------------------------------------------|
| SIGH-D | HAM-D-17 – Structured Interview Guide Version |
| SIGMA | MADRS – Structured Interview Guide Version |
| SOE | Schedule of Events |
| SOPs | Standard operating procedures |
| SUSAR | Suspected and unexpected serious adverse reaction |
| t½ | Terminal phase half-life |
| TEAE | Treatment-emergent adverse event |
| tmax | Time to reach maximum concentration |
| TSH | Thyroid stimulating hormone |
| ULN | Upper limit of normal |
| Vz/F | Apparent volume of distribution during the terminal phase |
| WBC | White blood cell |
| WHO | World Health Organization |

##  Version: 4.0 – 26 May 2021

## 2. INTRODUCTION

# 2.1. Major Depressive Disorder

Major depressive disorder, also known as unipolar or major depression, is characterized by a persistent feeling of sadness or a lack of interest in outside stimuli. The unipolar connotes a difference between MDD and bipolar depression, which refers to an oscillating state between depression and mania. Major depressive disorder is solely focused on the "lows," or the negative emotions and symptoms that are experienced (adapted from Lieber 2020). Depression is among the top public health concerns worldwide, causing significant disability and disease burden. In 2012, it was estimated that 16 million people were living with depression in the United States. The aim of antidepressant therapy is symptom remission or the reinstatement of euthymia—often defined as a score ≤7 on the total Hamilton Depression Rating Scale. Response, traditionally defined as a >50% decrease in the score from Baseline on a depression rating scale (commonly, the Hamilton Depression Rating Scale), has proven to be an inadequate goal, as many patients meeting the criteria for response will continue to have residual symptoms and functional impairments. Moreover, unremitted patients report poorer quality of life and are at a higher risk for relapse and recurrence of depression. Specifically, in the Sequenced Treatment Alternatives to Relieve Depression (STAR\*D) trial—the largest randomized depression study to date—68% of responders relapsed within the first year following treatment, compared with 47% of remitters who relapsed. In addition, when more treatment steps are needed, lower acute remission rates and higher relapse rates are to be expected. Indeed, one third of the STAR\*D cohort never remitted, even after four consecutive treatment trials. The remission rate was a mere 27.5% in Phase 1 treatment with citalogram, based on HAM-D scores, and 32.9% based on the Quick Inventory of Depressive Symptomology – Self-Report (QIDS-SR) scores (adapted from Ionescu et al., 2015). New antidepressant treatments with new mechanisms of action are needed to treat MDD.

# 2.2. Investigational Product



# 2.2.2. Non-clinical Studies





## 2.2.3. Clinical Studies

## 2.2.3.1. SP-624-101

SP-624 was assessed in a single, oral dose study, SP-624-101. The doses assessed following an overnight fast were 3 mg, 10 mg, and 30 mg. Additionally, 10 mg was assessed in a food effect cohort following an overnight fast and 30 minutes after a high fat meal. Each cohort in the first part of the study (non-food effect) comprised of eight subjects each, of whom six subjects per


cohort received single oral doses of SP-624 and two subjects received placebo. In the food effect part of the study, a separate cohort of eight subjects received SP-624 once under fasting conditions and once under fed conditions.

Orally administered SP-624 was well-tolerated after each dose.

There were no severe AEs, SAEs, deaths, or AEs leading to withdrawal in this study.

No placebo subjects reported an AE, and three SP-624 subjects reported at least one AE. One subject in the 3 mg dose group reported headache and insomnia, one subject in the 10 mg food effect fasted dose group reported headache, and one subject in the 10 mg food effect fed dose group reported vessel puncture site pain. All AEs were assessed as mild in intensity and not related to study drug.

Shifts in laboratory values appeared to be transient, and no patterns of clinical significance were observed. There were no laboratory values in the study that were deemed clinically significant by the Principal Investigator (PI).

There were no apparent patterns of mean change from Baseline in vital signs to suggest any effect from SP-624. There were no clinically relevant changes from Baseline in ECG parameters.

SP-624 displayed linear, dose-proportional PK when dosed following an overnight fast. At all dose levels SP-624 appeared to have a distinct absorption profile with some absorption occurring over the first two hours followed by a spike to the Cmax. Geometric mean plasma half-lives were similar across dose levels at 7.1, 6.8 and 6.8 hours for the 3, 10 and 30 mg cohorts, respectively. Volumes of distribution (Vz/F) were similar between cohorts (175, 230, and 209 liters) and displayed low inter-subject variability. Apparent systemic clearance (CL/F) values were consistent between cohorts (17.1, 23.6, and 21.4 L/h) with low variability.

When administered 30 minutes after a high fat meal (10 mg oral dose), plasma exposure to SP-624 was unchanged as assessed by area under the curve (AUC), but mean Cmax was decreased by approximately 30% and mean tmax was delayed from 2.25 hours to 5.13 hours.

## 2.2.3.2. SP-624-102

SP-624 was assessed in a multiple dose study, SP-624-102. The doses assessed were 3 mg, 10 mg, and 20 mg. The 3 and 10 mg doses were orally administered, once daily, for five days. The 20 mg dose was orally administered, once daily, for 10 days. Cohorts 1 and 2 (3 mg and 10 mg) comprised eight subjects each, of whom six received SP-624 and two received placebo. Cohort 3 comprised seven subjects, of whom five received SP-624 and two received placebo.

Orally administered SP-624 was well-tolerated after each dose. No safety concerns were identified for electrocardiography, vital signs, safety laboratories or adverse events for any cohort of subjects.

There were no severe AEs, SAEs, deaths, or AEs leading to withdrawal in this study.

No placebo subjects reported an AE, and five SP-624 subjects reported a total of 12 AEs. All AEs were reported by single subjects. All AEs were assessed as mild in intensity with the exception of arthralgia that was reported twice for one subject in the 3 mg SP-624 dose group;

once at mild intensity and once at moderate intensity. No AEs were assessed as probably related to study drug; eight AEs were assessed as possibly related: pallor (3 mg QD), procedural dizziness (3 mg QD), defecation urgency (20 mg QD), diarrhea (20 mg QD), melanocytic nevus (20 mg QD), oropharyngeal discomfort (20 mg QD), tongue blistering (20 mg QD), and tongue discomfort (20 mg QD).

AUC and Cmax values increased in proportion to dose during multiple dosing of SP-624 at dose levels of 3, 10, and 20 mg per day. Cmax exceeded predicted efficacious plasma concentrations of 3.28 ng/mL at all doses. t½ and CLss/F remained constant as the dose was increased. There was little or no accumulation during 5 days of dosing at 3, 10, and 20 mg SP-624 or 10 days of dosing at 20 mg SP-624.

# 2.3. SP-624 Development Plan

Sirtsei Pharmaceuticals, Inc. plans to investigate the safety and efficacy of SP-624 in this pilot, double-blind, placebo controlled, multicenter study in adults with moderate to severe MDD. The study will evaluate the safety and efficacy of a 4-week, multidose regimen of SP-624 versus placebo in approximately 300 subjects.

Pending the efficacy and safety profile observed from this study, additional nonclinical and clinical studies will be conducted.

## 2.3.1. Rationale for Dose



### 2.3.2. Benefit and Risk Assessment

SP-624 was well tolerated at a dose of 20 mg per day for 10 days in study SP-624-102. There were no SAEs, AEs leading to discontinuation, or severe AEs. There were no changes of


concern in clinical laboratory findings, physical exams, vital signs, ECGs, or mental status. Steady state Cmax values were well in excess of predicted efficacious concentrations.

It is concluded that the dose of SP-624 planned in this study, together with the safety monitoring procedures, has a low foreseeable risk of inflicting harm or injury to study participants. This is the first study of SP-624 in subjects with MDD and the study may provide initial evidence of efficacy. The Sponsor believes that the potential benefit of SP-624 for MDD and good tolerability profile supports conduct of this clinical study.

#### **3.** STUDY OBJECTIVES AND ENDPOINTS

#### **Objectives** 3.1.

#### **Primary Objective** 3.1.1.

Evaluate the efficacy of SP-624 administered once-daily for up to 4 weeks compared to placebo in the treatment of adults with MDD.

#### 3.1.2. **Secondary Objectives**

- Evaluate the safety and tolerability of SP-624 administered once-daily for up to 4 weeks compared to placebo in the treatment of adults with MDD; and
- Characterize the population PK of SP-624 in plasma when administered orally to subjects with MDD.

#### 3.2. **Endpoints**

#### 3.2.1. **Efficacy Endpoints**

#### 3.2.1.1. **Primary Endpoint**

Change from Baseline to Week 4 in MADRS total score

#### 3.2.1.2. **Secondary Endpoints**

- Change from Baseline to Weeks 1, 2, and 3 in MADRS total score
- Change from Baseline to Weeks 1, 2, 3, and 4 in CGI S total score
- Change from Baseline to Week 5 and change from Week 4 to Week 5 in MADRS total score and CGI-S total score
- Change from Baseline to Week 2 and Week 4 in the HAM-D-17 total score
- Change from Baseline to Week 2 and Week 4 in the SDS
- Change from Baseline to Week 2 and Week 4 in the QIDS-SR
- Change from Baseline to Week 2 and Week 4 in the Q-LES-Q-SF

#### 3.2.2. **Safety Endpoints**

- **AEs**
- Clinical safety laboratory tests (serum chemistry [including thyroid function], hematology, coagulation, and urinalysis tests)
- Vital signs (blood pressure, pulse rate, and oral body temperature)
- Body weight
- 12-lead ECGs


- Physical examinations
- C-SSRS

# 3.2.3. Pharmacokinetic Endpoints

A total of four blood samples will be collected from each subject for the measurement of plasma concentrations of SP-624 at the following visits:

- Visit 2 (Day -1)
- Visit 3 (Week 1): Pre-Dose
- Visit 4 (Week 2): Pre-Dose or approximately 2 to 10 hours post-dose (whichever is more convenient for the subject)
- Visit 6 (Week 4): approximately 2 to 10 hours post-dose



##  Version: 4.0 – 26 May 2021

## 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design

This is a Phase 2, multicenter, double-blind, randomized, placebo-controlled study of the safety and efficacy of SP-624 in the treatment of adult subjects with MDD as defined by the DSM-5. Following the successful completion of a Screening Phase, subjects will be randomized to one of two treatment groups in a 1:1 ratio and will receive SP-624 or placebo over a treatment period of four weeks (Treatment Group #1: SP-624 20 mg/day; Treatment Group #2: Placebo).

Approximately 300 subjects (150 per treatment group) will be enrolled into the study. Each subject will complete Screening, Baseline, Treatment, and Follow-up Visits.

The Schedule of Events (SOE) to be completed for subjects in the study is provided in Table 2.

An overview of the study schematics is displayed in Figure 1. Study periods are detailed below.

# 4.1.1. Screening Period and Baseline Visit

A Screening period of up to 28 days (Day -28 to Day -2) and a Baseline Visit (Day -1) will precede initiation of the Treatment Period. During the Screening Period, all Screening assessments will be completed and any current depression medications will be discontinued. All Screening assessments should be completed before discontinuing any current depression medications. An adequate number of subjects will be screened to ensure the planned number of subjects is enrolled (approximately 300 subjects).

The Screening Period may be extended for extenuating circumstances, such as when additional time is needed for medication taper/washout or to repeat laboratory testing, with the approval of the medical monitor.

Subjects who continue to satisfy all entry criteria at the Baseline Visit will be randomized in a 1:1 ratio to one of two treatment groups (Treatment Group #1: SP-624 20 mg/day; Treatment Group #2: placebo). At the completion of the Baseline Visit, randomized subjects will be dispensed study drug and will be instructed to begin dosing the next morning (Day 1).

## 4.1.2. Treatment and Follow-up Periods

Subjects will be scheduled to return to the clinic for safety and efficacy assessments at the end of Weeks 1, 2, 3, 4, and 5 as specified in the SOE (Table 2). After the final dose of study drug, subjects will complete a Follow-up Period of two weeks and will return at the end of Weeks 5 and 6. Subjects may be treated with anti-depressant medications according to physician recommendations after completion of the Week 5 Visit unless a clinically significant lab value is identified at the Week 4 Visit. If a clinically significant lab value is identified at the Week 4 Visit, consult with the Medical Monitor to determine if the lab value needs to be followed prior to initiating new therapy.

Unless there are any outstanding safety issues that require follow-up, subjects will be discharged from the study at the Week 6 Visit.


Figure 1: Study Schematic



##  Version: 4.0 – 26 May 2021

# 4.2. Randomization and Blinding

## 4.2.1. Subject Identification and Randomization to Treatment

A unique subject identification number (sometimes referred to as the Screening number and different from the randomization number) should be assigned to each subject who signs an informed consent form (ICF). The subject identification number should be used on all case report forms (CRFs) and in all correspondence between sites, the Sponsor, Institutional Review Boards (IRBs), and the Food and Drug Administration (FDA).

Sirtsei Pharmaceuticals or designee will generate a randomization scheme with appropriate blocking. Randomization numbers will be 3 digits starting with 101. When the decision is made to randomize a subject to treatment, the Investigator should pick the next available randomization number from the study drug kits assigned to the site. The subject randomization number will be recorded in the CRF, linking the subject's unique subject identification number to the subject's assigned randomization number.

## 4.2.2. Blinding

The study will be conducted under double-blind conditions, meaning the Investigator, study center personnel, study subjects, and Sponsor will be unaware of the treatment assignment for the subjects.

## 4.2.3. Emergency Unblinding

If an emergency situation occurs that, in the Investigator's opinion, cannot be adequately treated without knowing the identity of the study medication, the study treatment assignment can be unblinded via the tamper-evident covered disclosure panel attached to the study drug kit.

Every effort will be made to contact the Sponsor Medical Monitor prior to breaking the blind. If this is not possible and the situation is an emergency, the Investigator may break the blind for only the subject(s) involved in the emergency situation and must contact the Sponsor Medical Monitor as soon as possible (see Table 1 for Medical Monitor contact information).

In any case of emergency unblinding, pertinent information including the date and reasons for breaking the blind must be documented in the subject CRF and in the site and Sponsor study files.

# 4.3. Study Centers and Personnel

The study will be conducted at approximately 40 investigative sites located in the United States.

The PI at each site will be a licensed physician or clinical psychologist experienced in conducting studies in MDD. For those sites where a clinical psychologist is the PI, one of the sub-Investigators must be a licensed physician. The PI will be responsible for delegating study responsibilities to only those key site personnel who have the appropriate level of education, training and experience, including medical expertise and good clinical practice (GCP) training, as applicable for their assigned role in the study.

The clinical research facility at each investigative site will have adequate facilities and equipment to conduct the study procedures, and to allow for close supervision of study subjects,
Sirtsei Pharmaceuticals, Inc. Protocol No: SP-624-201 Amendment 3  Version: 4.0 – 26 May 2021

including immediate access to equipment and appropriately qualified staff to respond in the case of an acute medical emergency.

# 4.4. Number of Subjects

Approximately 300 adult subjects with MDD as defined by DSM-5 will be enrolled with approximately 150 subjects per treatment group.

# 4.5. Study Duration

Subjects will receive double-blind treatment for up to 4 weeks, following a Screening/washout period of up to 28 days. After the treatment period, subjects will complete a 2-week follow-up period. The planned study duration for each subject will be approximately 70 days.

###  Version: 4.0 – 26 May 2021

### 5. SELECTION AND WITHDRAWAL OF SUBJECTS

# 5.1. Subject Recruitment, Enrollment, and Identification

Subject recruitment and enrollment will be organized and overseen by the Investigator at the site following approval of the study protocol, ICF, and any study specific advertisements/recruitment materials by the respective IRB.

Subjects will be recruited via advertisements, physician referral, and from databases kept by the research center.

A sufficient number of subjects will be screened in order to ensure that a total of approximately 300 subjects who satisfy the entry criteria are randomized to treatment.

Each subject's signed and dated ICF to participate in the study must be obtained before conducting any study-related procedures. All subjects who sign an ICF will be given a unique Screening identification number and their study status will be tracked on a study Screening and Enrollment log maintained in the Investigator study files.

# **5.2.** Subject Inclusion Criteria

To be eligible for this study, subjects must meet all of the following inclusion criteria.

- 1. Willing and able to provide written informed consent to participate in the study.
- 2. Males and females, aged 18 to 65 years, inclusive.
- 3. In generally good physical health, in the opinion of the Investigator.
- 4. Body mass index must be  $\geq 18$  and  $\leq 40 \text{ kg/m}^2$
- 5. Females of reproductive potential and males with partners of reproductive potential must agree to remain abstinent or use adequate and reliable contraception throughout the study and for at least 30 days after the last dose of study drug.
  - a. Adequate contraception is defined as continuous use of double-barrier method (e.g., condom and spermicide or diaphragm and spermicide), oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, or intrauterine device.
  - b. Non-reproductive potential is defined as surgically sterile, undergone tubal ligation or vasectomy, or postmenopausal (defined as at least 12 months of spontaneous amenorrhea).
  - c. Subjects of reproductive potential but whose <u>sole</u> partner is of non-reproductive potential, or whose <u>sole</u> partner is of the same sex, are not required to maintain abstinence or contraception.
  - d. Subjects must agree to refrain from sperm and oocyte donation for at least 90 days after the last dose of study drug.
- 6. Meets DSM-5 criteria for moderate to severe MDD, as confirmed by the MINI. Subjects with a diagnosis of co-morbid GAD may be included if MDD is the primary diagnosis.
- 7. Montgomery-Asberg Depression Rating Scale total score ≥ 27 at both Screening and Baseline.

Sirtsei Pharmaceuticals, Inc.


8. History of inadequate or non-response to at least one adequate treatment, but no more than three of the same class of antidepressant, (i.e., an adequate dose for at least six weeks) for the current episode, in the opinion of the Investigator. NOTE: If immediately prior to this episode starting, treatment was working to the point of remission, but then the depression worsened, subject should not be enrolled. For example, subject should not

have been on an antidepressant and in remission prior to the start of the current episode.

9. Willing and able to comply with the study design schedule and other requirements.

# 5.3. Subject Exclusion Criteria

Amendment 3

A subject who meets any of the following exclusion criteria will not be enrolled in the study:

- 1. Female who is pregnant, breastfeeding, or less than six months postpartum at Screening.
- 2. History or presence of major bowel resection, total gastrectomy, or diabetes, and/or history or presence of any clinically significant medical condition, disease, or surgical history that could, in the opinion of the Investigator, jeopardize the safety of the subject or validity of the study data, or interfere with the absorption, distribution, metabolism, or excretion of the study drug.
- 3. A current DSM-5 diagnosis of depression with peripartum onset, panic disorder, obsessive compulsive disorder, post-traumatic stress disorder, anorexia nervosa, or bulimia nervosa.
- 4. A history of or current DSM-5 diagnosis of MDD with psychotic features, any schizophrenia spectrum and other psychotic disorders, bipolar disorder, or personality disorder.
- 5. History of treatment with ECT, vagus nerve stimulation, deep brain stimulation, or transcranial magnetic stimulation within six months of Screening.
- 6. Current episode of depression exceeds 2 years or is less than six weeks from Screening.
- 7. History of inadequate or non-response, in the opinion of the Investigator, to an adequate treatment regimen of two or more classes of antidepressants during the current episode.
- 8. Subjects treated with an antipsychotic during the current episode should be excluded.
- 9. Subjects who meet DSM-5 criteria for moderate or severe substance use disorder for any substance except nicotine or caffeine, within 12 months of Screening. Subjects with a urine drug screen positive for suspected substance of abuse will be excluded. Urine drug screen positive for cannabinoids is not exclusionary if the subject does not meet criteria for moderate or severe substance use disorder.
- 10. Will require initiation of psychotherapy during the study period, in the Investigator's opinion. If a subject has been in ongoing psychotherapy for a minimum of three months, the therapy may continue if it remains unchanged. Cognitive behavioral therapy is excluded.
- 11. Poses a current or future suicidal risk, in the Investigator's opinion, or has a history of suicidal behavior within the past 12 months, and/or subject answers "yes" to "Suicidal Ideation" Item 4 (active suicidal ideation with some intent to act, without specific plan)

Sirtsei Pharmaceuticals, Inc.


Amendment 3

or Item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment during the six months prior to the Screening period and/or at Baseline.

- 12. Failure to discontinue all psychoactive medications or psychoactive supplements including antidepressants and mood stabilizers, within a time period prior to Baseline corresponding to at least five half-lives of the medication in question.
- 13. Presence of a clinically significant abnormality on physical examination or ECG, including a QTcF >450 msec for males and >470 msec for females. Note: ECG may be repeated once at both Screening and Baseline for confirmatory purposes.
- 14. Presence or history of any known clinically significant cardiovascular disorders including, but not limited to: coronary artery disease, heart failure, valvular heart disease, cardiomyopathies, myocardial infarction, chamber enlargement or hypertrophy, or orthostatic hypotension.
- 15. Presence of uncontrolled hypertension, defined as consistent SBP >160 mmHg or consistent DBP >95 mmHg despite present therapy. Note: Blood pressure measurements may be repeated twice at both Screening and Baseline for confirmatory purposes.
- 16. Screening laboratory value(s) outside the laboratory reference range that are considered to be clinically significant by the Investigator (clinical chemistry, hematology, coagulation, and urinalysis). Note: Screening labs may be repeated once for confirmatory purposes.
- 17. Screening liver function tests (ALT, AST, Alkaline phosphatase) > 2x the upper limit of normal.
- 18. Known history of current or chronic Hepatitis B or Hepatitis C infection, or a known history of HIV infection. Subjects with a history of treated Hepatitis C infection where liver function tests are within normal limits may participate.
- 19. Subjects with a history of seizures or seizure disorder.

  Note: Subjects with a history of only febrile seizures, limited to up to two episodes, are permitted.
- 20. Clinically significant acute infection, other than mild viral or bacterial infections from which the subject has fully recovered (e.g., common cold, localized skin infection, etc.), within the two weeks prior to Baseline.
- 21. Major trauma or surgery in the 12 weeks prior to Screening or at any time between Screening and randomization.
- 22. Presence or history of malignancy within the last five years. Note: History of adequately treated basal cell or squamous cell carcinoma of the skin or in situ cervical cancer is allowed.
- 23. History of an anaphylactic allergic reaction to previous medication.
- 24. Blood or plasma donation within 30 days of randomization, or planned donations or elective surgery during the study or during the 60 days following the study.
- 25. Subjects who, in the opinion of the Investigator, are not suitable candidates for the study.


26. Individuals who are currently enrolled in or have participated in a clinical trial (i.e., received study drug) involving an investigational product within 60 days or within five half-lives of the investigational product (whichever is longer) prior to Baseline.

# 5.4. Subject Withdrawal from the Study

A subject may be withdrawn from the study at any time at the discretion of the Investigator.

Justifiable reasons to discontinue a subject from the study may include, but are not limited to, safety, ability or willingness to comply with conditions of the protocol, withdrawal of consent, lost to follow-up, Investigator discretion, Sponsor decision, or premature termination of the study.

The reason(s) for premature discontinuation will be documented on the subject's CRF.

Any AEs or SAEs that lead to study discontinuation should be followed as appropriate until the AE has resolved or stabilized (in the opinion of the Investigator and Sponsor Medical Monitor).

Subjects who prematurely discontinue after receiving a dose of study drug, should continue to be followed for scheduled safety assessments according to the SOE (Table 2), if possible. At a minimum, every attempt should be made to complete the Week 4 / Premature Discontinuation procedures; however, subjects are free to withdraw consent from participation in the study at any time, without prejudice to their medical care.

If a subject is lost to follow-up (i.e., fails to return for study visits), all reasonable efforts should be made to contact the subject and complete the Week 4 / Premature Discontinuation procedures.

Should it be discovered after a subject has begun study treatment that the subject did not meet all inclusion and exclusion criteria, or if during the study a subject ceases to meet all inclusion and exclusion criteria, the subject's continued participation in the study will be discussed with the Medical Monitor.

# 5.5. Premature Termination of the Study

If the study is prematurely terminated, written notification, documenting the reason for study termination, will be promptly provided by the Sponsor to the regulatory authorities. The Investigator will be responsible for informing the IRB.

The Sponsor reserves the right to terminate the study for any reason at any time.

# 

Version: 4.0 - 26 May 2021

# 6. STUDY TREATMENTS, MATERIALS, AND MANAGEMENT

# 6.1. Description of Study Drug

The study drug code name is SP-624. SP-624 is intended for the treatment of MDD.

The clinical trial material for this study will consist of capsules, each containing 10 mg of SP-624 API. Matching placebo capsules identical in shape and color to the active capsules will also be used.

# **6.2.** Acquisition of Study Drug Supplies

After the research site has submitted all approved regulatory and study start-up documents, the Sponsor will initiate a requisition for an initial shipment of study kits to be delivered to the site via the Sponsor's distribution facility.

All manufacturing, packaging, and labeling operations for the supplied study drug materials will be performed according to Good Manufacturing Practice (GMP) and GCP guidelines, as well as local regulations.

Storage and retest information will be provided for all supplied materials.

Upon receipt of the materials, the Investigator or designee will examine the package container, labeling, and appearance of the packaged materials to confirm the packaged materials were received in good condition.

All study materials will be stored at the study site in a restricted-access, securely locked area, under controlled temperature and humidity conditions in accordance with the manufacturer's instructions (see Section 6.7).

# **6.3.** Subject Treatment Assignment

When the decision is made to randomize a subject, the Investigator should pick the next randomization number from the study drug kits assigned to the site. The subject randomization number will be recorded in the CRF.

# 6.4. Study Drug Administration

Each dose of SP-624 will be supplied as two capsules, each containing 10 mg of API. Matching placebo capsules identical in shape and color to the active capsules will also be used. Following successful completion of the Baseline Visit, subjects will be randomized in a 1:1 ratio to one of two treatment groups:

- <u>Treatment Group #1:</u> Two 10 mg capsules SP-624 each morning for 4 weeks
- Treatment Group #2: Two capsules placebo each morning for 4 weeks

Each study drug dose should be taken orally, once daily at approximately the same time each morning. Study drug doses should be taken on an empty stomach before breakfast, and no food should be consumed for at least 1 hour after dosing. High fat foods at breakfast (e.g., bacon,

Sirtsei Pharmaceuticals, Inc. Protocol No: SP-624-201

Amendment 3


cheese, eggs, etc.) should be avoided. Morning liquids such as coffee or tea are allowed without any additives (eg, cream, sugar, etc).

If dosing on an empty stomach is not practical or not well tolerated, then a low fat, low calorie breakfast 2 hours before dosing, or 30-60 minutes after dosing, is acceptable. If dosing remains not well tolerated, then subjects should dose 30 minutes after a low fat, low calorie meal.

Study drug will be packaged in subject kits and each kit will contain four weekly blister cards with each card containing 20 capsules of study drug (two capsules per dose for seven days of dosing, plus three extra days of dosing as a provision for study visit scheduling). Each subject kit will be labeled with a 3-part label that specifies the randomization number, cautionary statement, and storage conditions. Each blister card will have a one-part label that specifies the randomization number, week, number of capsules, cautionary statement, and storage conditions.

Study drug will be dispensed as follows:

- Baseline Visit one blister card for Week 1
- Week 1 Visit one blister card for Week 2
- Week 2 Visit one blister card for Week 3
- Week 3 Visit one blister card for Week 4

Subjects will be instructed to return study drug at the Week 1, Week, 2, Week 3, and Week 4 (or Premature Discontinuation) Visits.

If the two capsule dose, is not well tolerated, the dose can be decreased to one capsule per dose after Week 1.

# **6.5.** Treatment Compliance

Study drug accountability will be recorded by study site staff, and any deviations from the administration instructions or dosing schedule will be entered into the subject's CRF.

# 6.6. Study Drug Accountability

The Investigator (or designee) is responsible for the accountability, reconciliation, and record maintenance of all study drug receipt, use, and disposition. In accordance with all applicable regulatory requirements, the Investigator or designated study personnel must maintain study drug accountability and storage records throughout the study. Unused drug will be returned to the investigative site and to the Sponsor or designee at the end of the study for destruction. No study drug usage outside the protocol will be allowed.

When a kit is assigned to a subject, the Investigator will tear off a 2 part segment of the label that contains a tamper-evident covered disclosure panel to be used for unblinding in case of emergency and affix the 2-part segment to the drug dispensing record. The drug dispensing record will be collected for the sponsor's files at the end of the study. This will serve to connect the unique randomization number to the unique subject identification number assigned at Screening.


# 6.7. Study Drug Storage and Stability

All study materials will be stored at the study site in a restricted-access, securely locked area, under controlled temperature and humidity conditions in accordance with the manufacturer's instructions.

The storage conditions for the study drug will be indicated on the label.

All supplied study drug materials will be stored at the study site in a restricted-access, securely locked area at the long-term refrigerated storage condition, 2-8°C. After a study drug kit has been assigned to a subject, the study drug kit and weekly blister cards dispensed to study subjects may be stored under room temperature conditions, 25°C (77°F), with excursions permitted between 15°C and 30°C (59°F-86°F).

In the solid state, the SP-624 drug substance is stable for at least 18 months when stored at 5°C and for at least 6 months when stored at 25°C/60% relative humidity.

SP-624 drug product stability is expected to directly correlate with that of the drug substance, since the drug product is neat drug substance filled into capsules. A 24-month stability program will be initiated for these capsules once manufacturing is completed, with storage conditions at 2-8°C and 25°C/60% relative humidity. Retest date information for the study drug will be provided.

At the Week 1, Week 2, Week 3, and Week 4 Visits, subjects will return the previously used blister cards, including any unused study drug. The used study drug kits will be maintained at the site under room temperature storage conditions until returned to the Sponsor or designee.

### **6.8.** Prior and Concomitant Medications

Medications taken within 28 days before Day 1 will be documented as prior medications. Medications taken any time on or after Day 1 and until completion of the Week 4 / Premature Discontinuation Visit will be documented as concomitant medications. Medications that started after the date of the last dose of study drug will not be considered concomitant but will be considered post-treatment.

The use of all prior, concomitant, and post-treatment medications will be recorded in the subject's CRF, including the drug name, dose, route of administration, dates of administration, and indication.

Once all Screening assessments have been completed, any current psychoactive medications and supplements must be discontinued. Subjects should consult with the Investigator before taking any medications, including over-the-counter products.

Subjects may be treated with anti-depressant medications according to physician recommendations after completion of the Week 5 Visit unless a clinically significant lab value is identified at the Week 4 Visit. If a clinically significant lab value is identified at the Week 4 Visit, consult with the Medical Monitor to determine if the lab value needs to be followed prior to initiating new therapy.

Previous medications for medical, non-psychiatric illnesses, as well as oral contraceptives and contraceptive devices, are permitted.

Medications such as non-steroidal anti-inflammatories, antacids, and non-psychoactive allergy medications, may be given at the discretion of the Investigator.

A list of restricted and prohibited medications is included in Table 4:

**Table 4: Restricted and Prohibited Medications** 

| <b>Medication Class</b> | Examples <sup>1</sup> | Comment |
|---|---|---|
| Antidepressants | Trazodone<br>TCAs<br>SSRIs<br>SNRIs<br>MAOIs | All prohibited Any anti-depressants being taken at the time of Screen must be discontinued within a time period prior to Baseline corresponding to at least five half-lives of the medication in question. |
| Antipsychotics | Aripiprazole Brexpiprazole Haloperidol Olanzapine Risperidone | All prohibited If an antipsychotic was used to treat the current episode of depression, the subject should be excluded. |
| Anxiolytics | Benzodiazepines | Restricted Subjects on a stable dose of lorazepam (2 mg/day), or equivalent dose of another benzodiazepine (e.g., diazepam 15 mg), for anxiety at the time of Screening may continue with the current treatment regimen. The dose should remain consistent throughout the study. Should a benzodiazepine be required for increased anxiety during the study in a subject who had not been taking a consistent dose prior to Screening, lorazepam 2 mg/day, or an equivalent dose of another benzodiazepine (e.g., diazepam 15 mg), is limited to two days or less per week. Use the night before or the day of a study visit (prior to the visit) is prohibited. Any need to exceed this amount must be discussed with the Medical Monitor. |
| Hypnotics | Zolpidem<br>Temazepam<br>Sedating<br>antihistamines | Restricted Zolpidem being taken daily for sleep at the time of the Screening visit is permitted for severe insomnia. The dose should remain consistent throughout the study. If zolpidem is being taken as needed at the time of Screening, use is limited to three nights or less per week and use the night before a study visit is prohibited. Prohibited All other hypnotics |

Amendment 3

| <b>Medication Class</b> | Examples <sup>1</sup> | Comment |
|---|---|---|
| Mood stabilizers | Lithium | All prohibited |
| and anticonvulsants | Valproate<br>Lamotrigine<br>Gabapentin | Any mood stabilizers or anticonvulsants being taken at the time of Screening must be discontinued within a time period prior to Baseline corresponding to at least five half lives of the medication in question. |
| Muscle relaxers | Carisoprodol Cyclobenzaprine Metaxalone Baclofen | Restricted Use of muscle relaxants during the study is limited to episodic use for an acute situation (e.g., back injury during the study) and must be discussed with the Medical Monitor. |
| Opioid analgesics | Oxycodone<br>Morphine<br>Tramadol<br>Codeine | Restricted Use of opioids during the study is limited to episodic use for an acute situation (e.g., back injury during the study) and must be discussed with the Medical Monitor. |
| Stimulants | Amphetamine Dextroamphetami ne Pemoline Methylphenidate | All prohibited Any stimulants being taken at the time of Screening must be discontinued within a time period prior to Baseline corresponding to at least five half-lives of the medication in question. |
| Herbal and nutritional supplements St. John's Wort Ginkgo Biloba S-Adenosyl methionine (SAM-e) Omega-3 supplements Cannabidiol products Melatonin | | Restricted Only multivitamins that do not contain any of the example ingredients are allowed during the study. |

<sup>&</sup>lt;sup>1</sup> Medications including, but not limited to, examples provided.

###  Version: 4.0 – 26 May 2021

### 7. STUDY PROCEDURES AND ASSESSMENTS

### 7.1. Schedule of Events

The SOE for participants in the study is provided in Table 2.

The actual dates of study drug administration and all study visits and assessments will be recorded in the subject's CRF. If a study visit or assessment occurs outside the specified time point and allowed time window (if applicable), then the reason for the deviation will be noted. Every attempt should be made to ensure that subsequent visits and assessments are performed on-time.

The Screening Period may be extended for extenuating circumstances, such as when additional time is needed for medication taper/washout or to repeat laboratory testing, with the approval of the medical monitor.

Study visits during the Treatment Period can be scheduled within  $a \pm 3$  day window relative to the Baseline Visit (i.e., the Week 1 Visit can be scheduled  $7 \pm 3$  days relative to the completion of the Baseline Visit, the Week 2 Visit can be scheduled  $14 \pm 3$  days relative to the completion of the Baseline Visit, the Week 3 Visit can be scheduled  $21 \pm 3$  days relative to the completion of the Baseline Visit, etc.).

The Week 5 Visit can be scheduled  $7 \pm 3$  days relative to the Week 4 / Premature Discontinuation Visit and the Week 6 Visit can be scheduled  $14 \pm 3$  days relative to the Week 4 / Premature Discontinuation Visit.

Whenever ECGs, vital signs, and a blood draw for PK and/or safety labs are scheduled on a given day, the ECG and vital signs should be completed in the sequence of procedures either prior to the blood draw (preferred) or after the blood draw, such that the blood draw does not interfere with the ECG and vital sign recordings.

In addition to the study visits and assessments described in the SOE, unscheduled visits/assessments may be performed or repeated at the discretion of the Investigator if required to further evaluate laboratory parameters or the subject's clinical safety.

# 7.2. Study-Specific Procedures

### 7.2.1. Informed Consent

The Investigator must inform each prospective subject of the nature of the study, explain the potential risks, and obtain written informed consent from the subject prior to performing any study-related Screening procedures. Once written informed consent is obtained, prospective subjects will be screened for eligibility into the study based on the inclusion and exclusion criteria detailed in Section 5.

# 7.2.2. Demographic Information, Medical History/Current Medical Conditions, and Treatment History

Demographic information (e.g., date of birth, sex, race, ethnicity) will be collected and a detailed medical history, including review of past and ongoing medical conditions or procedures will be


obtained during the Screening Period as specified in the SOE (Table 2). Additionally, treatment history for the current depressive episode will also be collected.

### 7.2.3. Mini International Neuropsychiatric Interview

Subjects must meet DSM-5 criteria for moderate to severe MDD, as confirmed by the MINI (Sheehan et. al, 1998). Subjects with a diagnosis of co-morbid GAD may be included if MDD is the primary diagnosis. The MINI should only be completed by Sponsor approved raters. Raters will be approved by the Sponsor based on education and experience conducting the MINI in subjects with MDD.

Current DSM-5 diagnoses of depression with peripartum onset, panic disorder, obsessive compulsive disorder, post-traumatic stress disorder, anorexia nervosa, or bulimia nervosa are exclusionary.

A history of or current DSM-5 diagnosis of MDD with psychotic features, any schizophrenia spectrum and other psychotic disorders, bipolar disorder, or personality disorder are exclusionary.

### 7.2.4. Assessment of Efficacy

Efficacy assessments will be conducted by individuals with sufficient experience conducting the below rating scales who have received centralized rater training and have been approved by the PI and Sponsor. Whenever possible, the same rater should assess the same subject throughout the study.

The schedule of these safety assessments is provided in the SOE (Table 2), and the study-specific procedures for completion of these assessments are detailed below.

Assessments should not be performed on subjects who have missed two or more consecutive study drug doses immediately before the Week 1, Week 2, Week 3, or Week 4 / Premature Discontinuation visits.

### 7.2.4.1. Montgomery-Asberg Depression Rating Scale

Efficacy will be assessed using the MADRS – Structured Interview Guide Version (SIGMA) (Appendix A). The MADRS is a 10-item depression rating scale. The MADRS will be completed at study visits as specified in the SOE (Table 2). In order to qualify for the study, subjects must have a MADRS total score  $\geq$  27 at both Screening and Baseline.

### 7.2.4.2. Clinical Global Impression – Severity

The CGI-S is completed by the Investigator and measures the severity of illness (Appendix B). The CGI-S is used to rate subjects on a 7-point scale ranging from "Normal" to "Among the most extremely ill patients.".

### 7.2.4.3. Hamilton-Depression Rating Scale (17-item)

The Hamilton-Depression Rating Scale is a 17-item depression rating scale (Appendix C). The HAM-D-17 – Structured Interview Guide Version (SIGH-D) will be completed at study visits as specified in the SOE (Table 2).

### 7.2.4.4. Sheehan Disability Scale

The SDS is a brief, subject-completed questionnaire that assesses functional impairment in work/school, social life, and family life/home responsibilities (Appendix D).

### 7.2.4.5. Quick Inventory of Depressive Symptomology – Self Report

The QIDS-SR is a subject-completed 16-item depression rating scale (Appendix E).

### 7.2.4.6. Quality of Life Enjoyment and Satisfaction Questionnaire – Short Form

The Q-LES-Q-SF is a subject-completed 16-item questionnaire that assesses life satisfaction over the past week (Appendix F). Each question is rated on a 5-point scale from 1 (Very Poor) to 5 (Very Good).

### 7.2.5. Assessment of Safety

Each subject will be closely monitored for safety throughout their study participation. Study-specific safety assessments will include the following:

- Physical examinations
- Vital signs (blood pressure, pulse rate, and oral body temperature)
- Body weight
- 12-lead ECGs
- Clinical safety laboratory tests (serum chemistry [including thyroid function], hematology, coagulation, and urinalysis tests)
- C-SSRS
- AEs

The schedule of these safety assessments is provided in the SOE (Table 2), and the study-specific procedures for completion of these assessments are detailed below.

### 7.2.5.1. Physical Examination

Physical examinations will be performed as specified in the SOE (Table 2).

Physical examinations will include a review of the following body systems: general appearance, skin and extremities, ears/eyes/nose/throat, head/neck, heart/chest, abdomen, musculoskeletal, and neurological.

Clinically significant findings on the Screening and Baseline physical examination will be evaluated to confirm the subject remains eligible for study participation. New clinically significant abnormalities or exacerbations that occur after the Screening visit will be captured as AEs.


### 7.2.5.2. Vital Signs, Height, and Weight Measurements

Vital sign measurements will be taken at the time points specified in the SOE (Table 2). Height will be measured (in centimeters) at Screen only; weight (in kilograms) will be measured at Screen and all other scheduled time points indicated in the SOE (Table 2).

Vital sign measurements will include systolic and diastolic blood pressure, pulse rate, and oral body temperature.

At each timepoint, vital signs will be assessed with the subject in the sitting position after approximately three minutes or more of quiet sitting.

Abnormal vital signs may be repeated twice for confirmatory purposes. Confirmed abnormal vital signs will be further categorized as clinically significant or not clinically significant by the Investigator based on his/her clinical judgement.

Subjects with confirmed clinically significant abnormal vital signs at the Screening or Baseline Visits should be excluded from the study. New clinically significant abnormalities or exacerbations that occur after the Screening Visit will be captured as AEs.

### 7.2.5.3. 12-lead Electrocardiograms

A 12-lead ECG will be obtained at the study site during the time points specified in the SOE (Table 2) using an ECG machine provided by the central ECG monitoring vendor. The central ECG vendor will supply the ECG quantitative and qualitative data. The ECG will be reviewed by medically qualified site personnel. The Investigator will review the ECG report for abnormalities and/or clinically significant changes from previous readings.

ECGs will be performed only after the subject is positioned supine, resting, and quiet for a minimum of three minutes.

Subjects with clinically significant abnormal ECG findings at the Screening or Baseline Visits should be excluded from the study as specified in the study inclusion/exclusion criteria (Section 5.2 and Section 5.3). Criteria for reporting abnormal ECG findings as AEs are provided in Section 8.1.1.

ECGs may be repeated once at both Screening and Baseline for confirmatory purposes.

The following quantitative ECG data will be recorded: heart rate (bpm), PR interval (msec), QRS duration (msec), QT interval (msec), and QTcF interval (msec).

The following qualitative ECG data will be documented: Overall interpretation (normal or abnormal) and if abnormal, comment describing the abnormality. Abnormal ECG results will be further categorized as clinically significant or not clinically significant by the Investigator.

### 7.2.5.4. Pregnancy Test

A serum pregnancy test for all females will be performed as indicated in the SOE (Table 2). A serum pregnancy test is required at the Screening and Week 4 / Premature Discontinuation Visit. A urine pregnancy test is to be performed at Day -1 as indicated in the SOE. If the urine pregnancy test at Day -1 is positive, a confirmatory serum pregnancy test will be conducted. If pregnancy is confirmed, the subject will be excluded from the study. If the urine pregnancy test is positive, randomization should be postponed until serum pregnancy test results can be


obtained and pregnancy definitively ruled-out. Any occurrence of pregnancy exposure (i.e., pregnancy in a female subject or the female partner of a male subject who has received study drug) must be reported to the Sponsor as summarized in Section 8.1.6.

# 7.2.5.5. Clinical Safety Laboratory Assessments

Blood samples for clinical safety laboratory tests will be collected as indicated in the SOE (Table 2) and analyzed at an accredited central laboratory approved by the Sponsor. The Clinical Laboratory Manual should be referenced for specific procedures with regards to sample collection, handling, labeling, storage, and shipping.

Clinical safety laboratory tests will include the following laboratory test panels: serum chemistry (including thyroid function), hematology, coagulation, and urinalysis.

A summary of the analytes included in each test panel is provided in Table 5.

Any value outside of the current reference ranges for the laboratory performing the test will be flagged on the laboratory results report.

Laboratory tests showing abnormal or exclusionary values at Screening may be repeated no more than once. After dose administration, abnormal laboratory test results may be repeated as often as deemed clinically necessary by the Investigator until the test values return to clinically acceptable limits or until an explanation other than drug effect is given.

Laboratory test results will be assessed in accordance with the reference ranges provided by the clinical laboratory. Abnormal laboratory results will be further categorized as clinically significant or not clinically significant by the Investigator. Subjects with clinically significant abnormal lab results at the Screening Visit should be excluded from the study. If subjects present with clinically significant lab results collected at the Baseline Visit, continued subject participation should be discussed with the Medical Monitor. New clinically significant abnormalities or exacerbations that occur after the Screening Visit will be captured as AEs.

An estimation of the total blood collection volume per subject is provided in Section 7.2.5.6 and Table 6.

### 7.2.5.6. Blood Volume Collection Summary

An estimation of the total blood collection volume per subject required for the Screening, Baseline, Treatment Period, and Follow-up Period, is provided in Table 6.

• A total of approximately 139.0 mL (about ½ of a cup) of blood is estimated to be drawn from subjects in the study over a period of about 70 days (depending on the length of the Screening period).


**Table 5:** Clinical Safety Laboratory Analytes

| Thyroid Function | Fasting Serum Chemistr | ry <sup>1</sup> | Hematology | Urinalysis <sup>2</sup> | Urine Drug Test |
|---|---|---|---|---|---|
| TSH T3 – Screen only T4 – Screen only Coagulation PT PTT INR | Albumin Alkaline Phosphatase ALT AST BUN Calcium Chloride CO <sub>2</sub> Creatinine eGFR <sup>3</sup> GGT Glucose LDH Magnesium Phosphorus | Potassium Sodium Total Bilirubin; if elevated obtain Direct Bilirubin Total Protein Uric Acid Total Cholesterol HDL Cholesterol LDL Cholesterol Triglycerides Creatine Phosphokinase Serum βhCG (all females) <sup>4</sup> | RBC (Erythrocyte) Count Hemoglobin Hematocrit Platelet Count WBC Count with differential (Absolute and %: Basophils, Eosinophils, Lymphocytes, Monocytes, and Neutrophils) MCV MCH MCHC RDW MPV Reticulocyte Count (Absolute and %) | pH Blood/ RBCs Protein Glucose Ketones Bilirubin Color Leukocytes or WBCs Nitrite Specific Gravity Urobilinogen Microscopic Exam Urine βhCG (all females) <sup>5</sup> | Amphetamines Barbiturates Cannabinoids Benzodiazepines Methadone Opiates Cocaine Phencyclidine |

All protocol scheduled Serum Chemistry samples should be collected with the subject in a fasting state (i.e., no food for a minimum of eight hours prior to sample collection).

ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; CBC=complete blood count; CO2=carbon dioxide or bicarbonate; eGFR=estimated glomerular filtration rate; GGT=gamma glutamyl transferase; hCG= human chorionic gonadotropin; HDL=high density lipoprotein; LDH=lactate dehydrogenase; LDL=low density lipoprotein; MCH=mean corpuscular hemoglobin; MCHC=MCH Concentration; MCV=mean cell volume; MPV=mean platelet volume; Premature D/C=Premature Discontinuation from treatment; PT=prothrombin time; PTT=partial thromboplastin time; RBC=red blood cell; RDW=RBC distribution width; TSH=thyroid stimulating hormone; WBC=white blood cell

<sup>&</sup>lt;sup>2</sup> If urine is positive for blood, leukocyte esterase, nitrite, or protein, then will default to reflex microtesting.

<sup>&</sup>lt;sup>3</sup> Cockcroft-Gault Method of calculation – subject weight is required for calculation

<sup>&</sup>lt;sup>4</sup> Serum pregnancy test at Screen and Week 4/Premature D/C

<sup>&</sup>lt;sup>5</sup> Urine pregnancy test at the Baseline Visit

Table 6: Estimation of Blood Volumes Required from Screening through the End of the Follow-up Period


| | Estimated | Study Day | | | | | | Estimated | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Tests | Blood<br>Draw<br>Volume/<br>Sample<br>(mL) | Screen<br>(Day -2<br>8 to -2) | Day -<br>1<br>(Pre-<br>Dose) | Week<br>1 | Week 2 | Week<br>3 | Week 4/ Prema ture D/C | Week<br>5 | Week<br>6 | Total<br>Blood<br>Draw<br>Volume<br>(mL) |
| Serum<br>Chemistry | | | | | | | | | | |
| Serum<br>Pregnancy<br>(females<br>only) | 7.5 | 7.5 | 7.5 | | 7.5 | | 7.5 | 7.5 | | 37.5 |
| TSH/T3/T4 | 5.0 | 5.0 | 5.0 | | 5.0 | | 5.0 | 5.0 | | 25.0 |
| Hematology | 3.0 | 3.0 | 3.0 | | 3.0 | | 3.0 | 3.0 | | 15.0 |
| Coagulation | 2.7 | 2.7 | 2.7 | | 2.7 | | 2.7 | 2.7 | | 13.5 |
| PK | 6.0 | | 6.0 | 6.0 | 6.0 | | 6.0 | | | 24.0 |
| Estimated T<br>Blood D | | 18.2 | 30.2 | 6.0 | 30.2 | 0.0 | 30.2 | 24.2 | 0.0 | 139.0 mL |

Abbreviations: PK=Pharmacokinetics; Premature D/C=Premature Discontinuation from treatment

###  Version: 4.0 – 26 May 2021

### 7.2.5.7. Columbia-Suicide Severity Rating Scale

The C-SSRS (Appendix G and Appendix H) will be administered by a trained site staff member during the Screening Period (Baseline/Screening Version) and the Treatment and Follow-up Periods (Since Last Visit Version) as specified in the SOE (Table 2). Subjects who pose a current or future suicidal risk in the Investigator's opinion, or have a history of suicidal behavior within the past 12 months, and/or answers "yes" to "Suicidal Ideation" Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment during the six months prior to the Screening period and/or at Baseline will not be eligible for study enrollment.

Subjects who at any time during this study spontaneously report AEs of suicidal ideation or suicidal behavior, either as an outpatient or during visit interviews, must be assessed by the PI or designee and referred for further mental health evaluation as clinically indicated.

### 7.2.6. Assessment of Pharmacokinetics

### 7.2.6.1. Pharmacokinetics

The population PK of SP-624 will be assessed.

A total of four blood samples (6 mL) will be collected from each subject for the measurement of plasma concentrations of SP-624 at the following visits:

- Visit 2 (Day -1)
- Visit 3 (Week 1): Pre-Dose
- Visit 4 (Week 2): Pre-Dose or approximately 2 to 10 hours post-dose (whichever is more convenient for the subject)
- Visit 6 (Week 4): approximately 2 to 10 hours post-dose

If a subject missed the dose the day before a scheduled "pre-dose" sample collection, study personnel should instead collect a post-dose sample at that visit. Should a subject inadvertently dose prior to a scheduled "pre-dose" sample collection at Week 1 or Week 2, study personnel should collect a post-dose sample.

In the event that samples cannot be conveniently collected for a given subject according to the scheduled sampling times specified above, study personnel should attempt to collect at least one pre-dose sample and at least one post-dose sample during the course of the study.

Plasma samples will be analyzed for SP-624 concentration using a validated bioanalytical method.

An aliquot of each subject's post-dose samples may be pooled by the bioanalytical laboratory for metabolite profiling. Potential metabolites will be identified using mass spectrometry techniques; and if conducted, these data will be summarized in a separate bioanalytical report.

Labels on blood sample collection tubes and vials will include the protocol code number, subject identification code number, and visit number.

Samples will be stored at the study center until shipment under appropriate conditions to the Sponsor-designated bioanalytical laboratory for analysis. The bioanalytical lab will analyze the samples for plasma concentrations of SP-624 using a validated LC-MS method.

Detailed instructions for all blood sampling, processing, storage, and shipment procedures will be provided in a separate study guidance document.

An estimation of the total blood collection volume per subject is provided in Section 7.2.5.6 and Table 6.




# 8. ADVERSE EVENTS, SERIOUS ADVERSE EVENTS, AND OTHER REPORTABLE EVENTS

### **8.1.** Adverse Events

An AE is any untoward medical occurrence in a clinical study subject, whether or not the event is considered causally related to the study drug. An AE can be a new occurrence or an existing process that increases significantly in intensity or frequency.

All AEs must be recorded in the appropriate section of the CRF.

Adverse event monitoring for each subject begins upon Screening and continues until study completion. Abnormalities present at Screening are considered AEs only if they reoccur after resolution or worsen in intensity or frequency during the study.

Each AE is to be classified as serious or non-serious, and categorized with regard to relationship to study drug, and intensity.

### 8.1.1. Clinical Safety Assessment Abnormalities

Abnormal findings on clinical safety assessments, including clinical safety laboratory test results, vital sign measurements, ECGs, and physical examinations, will be assessed by the Investigator as clinically significant or not clinically significant. Clinically significant abnormalities that are new or exacerbate after the Screening Visit will be reported as AEs. Classification of seriousness, relationship to study drug, and intensity should use the guidelines provided in Section 8.1.2, Section 8.1.4.3 and Section 8.1.4.4, respectively.

### 8.1.2. Serious Adverse Event (SAE)

An AE is serious, regardless of whether or not it is considered related to the study drug, if the event meets one or more of the following criteria:

- Results in death.
- Is life threatening; per the Investigator, the subject was at immediate risk of death from the event at the time that the event occurred. It does not include an event that hypothetically might have caused death if it had occurred in a more severe form.
- Requires in-patient hospitalization; initial or prolonged, meaning that a hospital admission and/or prolongation of a hospital stay was required for the treatment of the AE, or occurred as a consequence of the event. It does not include a pre-planned elective hospital admission for treatment or diagnostic procedures.
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- Congenital anomaly or birth defect that occurs in the offspring of a subject exposed to the study drug.
- Important medical event that, although does not result in one of the other serious outcomes, requires medical or surgical intervention in order to prevent one of the other serious outcomes listed above. Examples of such medical events include

Amendment 3

allergic bronchospasm requiring intensive treatment in the emergency room or at home, blood dyscrasias, or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

All SAEs that occur after any subject has been enrolled, before treatment, during treatment, or within 28 days following the Week 4 Visit, whether or not they are related to the study, must be recorded on forms provided by Sirtsei Pharmaceuticals.

#### 8.1.3. **Suspected and Unexpected Serious Adverse Reactions**

A suspected and unexpected serious adverse reaction (SUSAR) is defined as an SAE that meets both of the following criteria with respect to study drug:

- Suspected: is assessed as probably or possibly related to study drug (see Section 8.1.4.3)
- Unexpected: in comparison to drug-related AEs described in the Investigator's Brochure, the event meets any of the following criteria:
  - The event was not previously described; or is now characterized more specifically (e.g., an event of "interstitial nephritis" in a subject receiving an agent previously described as associated with "acute renal failure"); and/or
  - The event is now characterized as more severe (see Section 8.1.4.4).

#### 8.1.4. **Evaluation of Adverse Events**

Adverse events spontaneously reported by the subject and/or in response to an open question from the study personnel (i.e., how are you feeling?) or revealed by observation will be recorded during the study at the investigational site.

All AEs/SAEs will be recorded in the CRF and will include a concise AE term/diagnosis, date and time of event onset and resolution, relationship to study drug, intensity, action taken, and outcome as described in Section 8.1.4.1 through Section 8.1.4.6.

Abnormalities in vital signs, laboratory results, and other safety assessments will be recorded as an AE if they meet the definition of an AE (Section 8.1.1).

Events that are considered symptoms of MDD should not be recorded as medical history or AEs. Lack of efficacy should not be considered an AE.

#### 8.1.4.1. **Adverse Event Term/Diagnosis**

The diagnosis or description of the AE will be as specific and complete as possible (i.e., "lower extremity edema," rather than just "edema").

Whenever possible, signs, symptoms, and laboratory abnormalities due to a common etiology will be reported as an integrated diagnosis; for example, cough, runny nose, sneezing, sore throat, and head congestion would be reported as "upper respiratory infection." The AE term should be reported in standard medical terminology when possible.

A medical or surgical procedure is not an AE; rather the condition leading to the procedure should be recorded as the AE. If the condition is not known, the procedure may be reported as


Amendment 3

an AE instead. Similarly, death is not an AE, but is rather the outcome of the AE(s) that resulted in death. If the AE(s) leading to death are not known, then death will be reported as an AE.

#### 8.1.4.2. Date and Time of Adverse Event Onset and Resolution

The time, if available, and date at which the AE was first apparent will be recorded as the event onset. The date and time of onset of symptoms may be appreciably earlier than the date and time the Investigator becomes aware of the event. Some events may be apparent to the subject and Investigator independently, and information from each may contribute to the final report. The date and time of resolution of the event will be recorded when they are available.

#### 8.1.4.3. **Relationship to Study Drug**

A causality assessment (i.e., assessment of relationship to study drug) must be provided for all AEs. This assessment must be made by a physician Investigator and recorded on the CRF. The definitions for the causality assessment are provided below.

- **Probably Related:** an event that (1) follows a reasonable temporal sequence from administration of the drug, (2) follows a known or expected response pattern to the drug, (3) is improved/resolved by stopping or reducing the dosage of the drug, and/or (4) could not be reasonably explained by the known characteristics of the subject's clinical state.
- Possibly Related: an event that follows a reasonable temporal sequence from administration of the drug and where a causal relationship between drug administration and event is a reasonable possibility, even if the event could readily have been produced by a number of other factors. The expression "reasonable possibility" is meant to convey in general that there are facts (evidence) or arguments to suggest a causal relationship.
- Not Related: an event that is unlikely to have any relationship to the study drug even if such relationship cannot be definitely ruled out.

If the relationship between the AE/SAE and the study drug is determined to be "possible" or "probable" the event will be classified as "related" to the study drug for the purposes of expedited regulatory reporting.

#### 8.1.4.4. **Intensity Categorization**

The intensity of all AEs will be assessed by the Investigator using the following criteria:

- Mild: An AE that is transient, requires minimal or no treatment, and does not interfere with the subject's daily activities.
- **Moderate:** An AE that is usually alleviated with specific therapeutic intervention. The event causes some interference with usual activities of daily living, causing discomfort, but poses no significant or permanent risk of harm to the research participant.
- **Severe:** An AE that is incapacitating, prevents usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention.


It is important to distinguish between serious and severe AEs. Intensity is a measure of severity whereas seriousness is defined by the criteria under Section 8.1.2. An AE of severe intensity may not be considered serious (e.g., a headache can be severe but not serious – e.g., is not life threatening, or does not result in hospitalization).

### **8.1.4.5.** Action Taken for Adverse Event

Adverse events will be followed and managed by the Investigator, including obtaining any supplemental tests or assessments needed to define the nature and/or cause of the event (e.g., laboratory tests, diagnostic procedures, consultation with other health care professionals, etc.).

For each AE, the Investigator will categorize one or more actions taken to manage the AE as follows:

- **Discontinuation:** Scheduled study procedures and/or study drug dosing (if applicable) were stopped due to the AE.
- **Study drug dose reduction:** The study drug dose is decreased from two capsules per day to one capsule per day.
- **Concomitant medication:** One or more medications (prescription or over the counter) were started or increased in dosage.
- Study drug dose taken with food: The study drug dose is taken  $\leq 2$  hours following a meal or a meal is eaten  $\leq 1$  hour after taking a dose.
- Other action: Non-medication action(s) were ordered as management of the AE (e.g., bed placed in Trendelenburg position, warm compresses applied to intravenous access site, etc.).
- **No action:** No actions were ordered for management of the AE.

### 8.1.4.6. Outcome of Adverse Event

If possible, AEs will be followed until resolved (i.e., recovered, recuperated, or ended) either with or without sequelae, or the Investigator and Sponsor Medical Monitor assess them as chronic or stable, and no longer requiring follow-up.

The outcome of each event (including time if available, and date) will be described using the following categories:

- **Recovered:** The event resolved, and subject returned to Baseline.
- **Recovered with Sequelae:** The event resolved but the subject is left with residual problems (e.g., functional deficits, pain).
- **Not Recovered:** At the last observation, the event was ongoing.
- **Death (Fatal):** To be used for the one AE which, in the judgment of the Investigator, was the primary cause of death.
- **Unknown:** There were no observations after the onset (initial observation or report) of the event, or subject is lost-to-follow-up and outcome of AE is unknown.

A subject who is discontinued from study drug because of an AE must be followed by the Investigator until clinical recovery is complete and laboratory results have returned to normal, or


until progression has been stabilized. Follow-up may need to continue after the subject has discontinued from the study, and additional investigations may be requested by the Investigator.

#### 8.1.5. **Reporting of Serious Adverse Events**

The Investigator will review each SAE and evaluate the severity and the causal relationship of the event to study drug. Serious AEs that occur after the last study visit and come to the attention of the Investigator must be reported only if there is (in the opinion of the Investigator) reasonable causal relationship with the study drug. Serious AE reporting contact information is provided in Table 1.

The Investigator is responsible for providing notification to the Sponsor (Table 1) of any SAE, within 24 hours of when he or she became aware of the event, whether deemed study drug related or not.

An SAE report form template will be provided to the Investigator by the Sponsor (or designee) prior to study initiation, with the preferred format for reporting SAEs.

As a minimum requirement, the initial notification should include the following information:

- Study number
- Subject number
- Name of Investigator
- AE term
- Criterion for classification as 'serious'
- Study drug name
- Causality assessment (if sufficient information is available to make this classification)
- Identifiable reporter of event

If clarification is requested by the Sponsor for omitted or discrepant information in the initial notification, the Investigator or an authorized delegate is responsible for sending the requested information within 24 hours.

Initial reports of SAEs must be followed later with detailed descriptions, including clear copies of other documents as necessary (e.g., hospital reports, consultant reports, autopsy reports), with the study subject's personal identifiers removed. Additional information on the SAE may be requested, which the Investigator or an authorized delegate must send to the SAE reporting contact (Table 1).

The Sponsor is responsible for expedited reporting of qualifying events to relevant regulatory authorities. It is the Investigator's responsibility to notify the IRB of all SAEs that occur at his or her site. Investigators will also be notified by the Sponsor of all unexpected, serious, drugrelated events [Investigational New Drug (IND) safety reports; also known as SUSARs] that occur during the clinical trial from any other studies or study sites. The Investigator is responsible for notifying its IRB of these events.

Sirtsei Pharmaceuticals, Inc.


Amendment 3


### 8.1.6. Other Reportable Events

Certain events that occur in the absence of an AE should be reported to the Sponsor. These include the following events:

- Pregnancy Exposure (subject or subject's partner becomes pregnant at any time during study participation and through 30 days post-dose).
  - Should a female subject or partner of a male subject become pregnant during the study, the subject will inform the Investigator.
  - The subject will be asked to follow up with the study site to report the eventual outcome of the pregnancy. The information will be tracked by the Sponsor.
  - The outcome of all pregnancies (spontaneous miscarriage, elective termination, normal birth or congenital abnormality) must be followed up and documented even if the subject was discontinued from the study.
  - Pregnancy in itself is not regarded as an AE.
  - All reports of congenital abnormalities/birth defects are SAEs. Spontaneous miscarriages should also be reported and handled as SAEs. Elective abortions without complications should not be handled as AEs.
- Lactation Exposure (subject was taking study drug while nursing an infant).
- Accidental Exposure (someone other than the study subject was exposed to study drug).
- Overdose of Study Drug (defined as dosing > 4 capsules in a 24-hour period) as a result of a dosing amount error should be reported. Any adverse outcomes of the overdose should be recorded as AEs/SAEs according to the procedures described in Section 8.1 through Section 8.1.5. Intentional overdose of study drug should be evaluated as a potential AE/SAE and reported accordingly.
- Other medication errors that potentially place subjects at greater risk of harm than was previously known or recognized (i.e., study drug was administered via an incorrect route).

Amendment 3


### 9. STATISTICS

Following are proposed statistical analyses. A separate Statistical Analysis Plan (SAP) will be generated and finalized prior to analysis. The SAP will specify the details of all statistical analyses, including all efficacy and safety analyses to be performed.

# 9.1. Determination of Sample Size

Recent studies of MDD using change from Baseline in MADRS total scores suggest that placebo will yield an approximately nine unit decrease over four weeks with a SD of around 9.2. SP-624 is expected to yield at least a 12 unit decrease in MADRS total score over four weeks with a similar SD of around 9.2. A minimum of 150 subjects per treatment arm (300 total) would be needed to detect a treatment difference of three units with 80% statistical power. The sample size was estimated using NQuery 8 (V8.5.2.0) two group test of equal means (MTT0-1: www.statsols.com).

# 9.2. Analysis Populations

Within each population, analyses will be performed comparing subjects and by-treatment assignment (SP-624 vs placebo).

- All Subjects Population all subjects who sign informed consent and are assigned a unique subject identification number. This population will be used to summarize disposition.
- Modified Intent-to-Treat (mITT) Population all subjects who are randomized to receive treatment, receive at least one dose of study drug, and have a Baseline and at least one post-dose efficacy assessment. This population will be the primary population used to summarize demographics, baseline characteristics, medical history, treatment history, and all efficacy outcomes. Subjects will be analyzed according to randomized treatment group.
- Per Protocol (PP) Population All subjects in the mITT population who received assigned study drug as randomized, completed the Week 4 assessments without any major protocol violations, and have 75-125% compliance. The PP population will be used as an additional population for summaries of efficacy outcomes.
- Safety Population all subjects in the mITT population who receive at least one dose of study drug. Safety subjects will be summarized according to the treatment they actually received, in case they received a different treatment than assigned at randomization. This population will be used to summarize all safety assessments.
- PK Population all subjects who receive active study drug and have evaluable PK
  data based on actual treatment received, protocol compliance, adequate numbers of
  samples, and successful sample assays.


# 9.3. Description of Statistical Methods

### 9.3.1. General Approach

All data will be provided in listing files. Study results and information will be displayed in descriptive summary tables. Inferential tests are identified below. For measurements that have multiple intermediate visits, results for observed data will be summarized for each time.

When comparisons between groups are performed, two-sided tests at a 0.05 level of significance ( $\alpha$ =0.05) will be used. The null hypothesis for all analyses is that there is no difference between the SP-624 and placebo treatment groups. There is only one primary outcome for analysis, and there will be no adjustment for multiplicity for secondary endpoints.

All summaries, statistical analyses, and individual subject data listings described below will be completed using Version 9.4 or later of the SAS Statistical Analysis System (SAS Institute, Inc. Cary, NC).

Subjects who are randomized but not treated and those who are treated but have no post-treatment follow-up assessments or data will be listed, but not analyzed.

### 9.3.2. Interim Analysis

No formal interim analyses are planned for this study.

# 9.3.3. Summary of Demographics, Baseline Characteristics, Medical History, and Treatment History

Listings and summaries of demographics, baseline characteristics, medical history, and treatment history will be provided for the mITT and safety populations. Categorical variables will be assessed for homogeneity across the treatment arms using a Fisher's exact test and numeric variables will be compared using a Wilcoxon rank-sum test. If there are any ordered categorical variables, the homogeneity of the treatment arms will be evaluated using a CMH row-mean score test calculated with modified ridit ranks. This summary will be provided for the mITT population.

### 9.3.4. Summary of Efficacy

Efficacy analyses will be conducted using the mITT population.

### 9.3.4.1. Primary Efficacy Endpoint Analysis

The MADRS is a 10-item scale whose total score can range from 0 to 60. The primary efficacy variable is change from Baseline in MADRS total score at Week 4, for testing superiority of SP-624 vs. placebo in adults with major depressive disorder. The analysis will be completed using observed data without imputation. Scores will be taken at 4 weeks regardless of subject discontinuation from treatment. Subjects will not be treated with any other antidepressant medication until at least the completion of the Week 5 visit.

The change from Baseline in MADRS total score at Week 4 will be analyzed from the difference in least square mean change using MMRM, with change from Baseline in MADRS total score at each visit as the response variable. The MMRM model will include age, weight, and baseline

Sirtsei Pharmaceuticals, Inc. Protocol No: SP-624-201

Amendment 3


MADRS total score as covariates, with factors for treatment, visit (Weeks 1, 2, 3, and 4; as a categorical variable), treatment by visit interaction term, gender, and site as a fixed effect. An unstructured covariance matrix will be used for the within-subject correlation. Kenward-Rogers approximation will be used to calculate the denominator degrees of freedom. The primary efficacy endpoint will be calculated using an estimate statement. Subjects from low enrolling sites may be pooled in order to help with model convergence.

In the event of a model which fails to converge, additional strategies to address convergence may be required such as alternative covariance structures, using a maximum likelihood versus restricted maximum likelihood (REML) estimation, or dropping variables.

The protocol may include approximately 40 sites and sites with less than 10 subjects will be pooled to obtain at least 10 subjects. Sites would be pooled in order of the site number and, if necessary, the last un-pooled site will be pooled with the last set of sites pooled.

Additional variables of interest that may be evaluated as covariates will be identified in the SAP, such as age of onset of depression and number of lifetime episodes.

Additionally, results from the primary outcome will be summarized for the PP population.

### 9.3.4.2. Secondary Efficacy Endpoint Analysis

Seven secondary efficacy endpoints will be analyzed using both the mITT and PP populations. These include:

- Change from Baseline to Weeks 1, 2, and 3 in MADRS total score for SP-624 vs. placebo. The outcome will be analyzed using the same methods as the primary outcome.
- CGI-S is measured on a 7-point scale where 1 represents "normal" and 7 represents "most extremely ill". A summary of percentage of subjects with each score at Baseline and at Weeks 1, 2, 3, and 4 will be presented. The change from Baseline in CGI-S can take on interval values between -6 (improvement from 7 to 1) and 6 (worsening from 1 to 7). Treatment comparison of change from Baseline to Weeks 1, 2, 3, and 4 in CGI-S scores will be performed using an MMRM model similar to that of the primary efficacy variable.
- Change from Baseline to Week 5 and change from Week 4 to Week 5 will be assessed using descriptive statistics for the MADRS and CGI-S.
- The HAM-D-17 is a 17-item scale whose total score can range from 0 to 52. Change from Baseline to Week 2 and Week 4 in the 17-item Hamilton Depression Rating Scale (HAM-D-17) total score will be assessed for treatment differences using an MMRM model similar to that of the primary efficacy variable.
- The Sheehan Disability Scale (SDS) is a 3-part scale that measures the degree of disruption on work, social and family life using an 11-point scale where 0 represents "no disruption" and 10 represents "extreme disruption". In addition to the 11-point scale, subjects are asked to indicate the number of days in the past week that were "lost" and numbers of days that were "unproductive". The results of these questions have a range from 0 to 7. A total global functioning impairment score can be utilized by summing the scores from work, social and family life scales for a value range from 0 to 30. Treatment

Sirtsei Pharmaceuticals, Inc.


Amendment 3

difference in change from Baseline to Week 2 and Week 4 for both global functioning impairment and days lost/unproductive will be assessed using an MMRM model similar to that of the primary efficacy variable. Change in days lost will be analyzed separately from change in unproductive days.

- The Quick Inventory of Depressive Symptomology Self Report (QIDS-SR), is a 16-item self-reported scale where each item has a 4-point scale where 0 represents least impact scores while 3 represents greatest impact scores. Scale 6 and 7 are linked such that only one of these will be scored. Likewise, scales 8 and 9 are linked such that only one of them will be scored. Nine domains are scored based on the highest score of items within that domain. The total score from all domains can take a value ranging from 0 to 27. Treatment difference in change from Baseline to Week 2 and Week 4 in the QIDS-SR will be assessed using an MMRM model similar to that of the primary efficacy variable.
- The Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) is a 16-item satisfaction scale where each item has a 5-point scale. A score of 1 represents "very poor satisfaction", while a score of 5 represents "very good satisfaction". Only the first 14 items are summed for a total score that ranges from 14 to 70 and is expressed as a percentage based on the maximum total score of the items completed (0–100). Treatment difference in the change from Baseline to Week 2 and Week 4 in total scores will be assessed using an MMRM model similar to that of the primary efficacy variable. The last two items pertaining to satisfaction with medications and overall contentment will be summarized separately by treatment group.

### 9.3.5. Sensitivity Analyses

A dropout rate of 20-30% is typically seen in MDD studies. The mechanisms that cause missing data may be missing at random (MAR) or may be missing not at random (MNAR). The MMRM model (especially as implemented within the PROC MIXED procedure in SAS) used in the primary analysis of the primary efficacy endpoint relies on the assumption of MAR. Hence, a sensitivity analysis for the primary endpoint and secondary endpoints will be performed using a pattern-mixture modeling approach (Kenward, et al 2003).

Additionally, subjects will be grouped by the visit at which they had their last MADRS total score measured. This will result in five categories of discontinuation: Week 1 dropouts, Week 2 dropouts, Week 3 dropouts, Week 4 dropouts, and completers. Mean change from Baseline in MADRS total score will be plotted by the dropout category and by reason for discontinuation, in order to assess whether this efficacy measure appears to be correlated with study dropout.

If missing data are greater than 25% or the pattern-mixture model provides a different interpretation of the treatment comparison for the primary endpoint, a multiple imputation analysis may also be performed using a fully conditional specification (FCS) approach using variables identified in the SAP.

### 9.3.6. Summary of Pharmacokinetics

Plasma concentration data for SP-624 will be listed and summarized using descriptive statistics.

Sirtsei Pharmaceuticals, Inc. Protocol No: SP-624-201 Amendment 3  Version: 4.0 – 26 May 2021

If data allow, results will be used for other analyses (e.g., PopPK) which will be presented in a separate report.

The population PK analysis of SP-624 will be performed using a nonlinear mixed effects model (NONMEM). This analysis will provide estimates of population PK parameters such as CL/F, Vz/F, etc. and a measure of their variability. Pharmacokinetic parameters of individual subjects (e.g., AUC[0-tau], Cavg, Cmax) may be estimated and their correlation with relevant covariates (e.g., body weight, gender, concomitant medications) will be explored. The population PK analysis plan will be prepared separately.

Plasma concentration data will remain blinded until the unblinding of the clinical database at the end of the study.

### 9.3.7.

### 9.3.8. Concomitant Medications

Concomitant medications will be coded using the most current version of the World Health Organization (WHO) drug dictionary available.

Any medications taken during the course of the study with a start date on or after the date of the first dose of study drug and on or before the date of the last dose of study drug, or with a start date prior to, and an end date on or after, the date of the first dose of study drug, or marked as ongoing, will be considered concomitant medications. Medications that ended prior to the date of the first dose of study drug will be considered prior medications. Medications that started after the date of the last dose of study drug will not be considered concomitant but will be considered post-treatment. Prior and concomitant medications will be summarized for the number and percentage of subjects using each medication by treatment and by the drug class and preferred name for the safety population.

### 9.3.9. Summary of Safety and Tolerability

All summaries of safety and tolerability will be performed on the safety population.

Laboratory parameters, vital sign data, and ECG results will be summarized by treatment group and presented in tabular and graphic formats where appropriate. Appropriate change from Baseline calculations will be provided to detect any significant changes in laboratory parameters, vital sign values, ECG results, and C-SSRS results, but no formal statistical tests are planned.

### 9.3.9.1. Adverse events

Summaries of the number and percentage of subjects in the safety population with at least one treatment-emergent AE (TEAE), classified according to preferred term and/or body system using the MedDRA dictionary, will be provided overall and by treatment group for:

- Overall summary
- All TEAEs
- TEAEs by relationship (not related, possibly related, probably related)

Sirtsei Pharmaceuticals, Inc.


Amendment 3


- TEAEs by severity (mild, moderate, severe)
- SAEs
- TEAEs leading to withdrawal from the study
- TEAEs leading to study drug dose reduction
- TEAEs leading to study drug dose taken with food
- Analyses of AEs with time of onset beginning 24 hours after the final dose through up to 28 days after the final dose.

No formal statistical tests are planned for AE data.

### 9.3.9.2. Vital Signs and ECGs

Vital signs and ECG results will be summarized by treatment group and presented in tabular and graphic formats where appropriate. Appropriate change from Baseline calculations will be provided to detect any significant changes in vital sign values or ECG results, but no formal statistical tests are planned. Any abnormal finding or clinically significant changes will be captured as AEs.

### 9.3.9.3. Clinical Laboratory Assessments

Clinical laboratory test results for chemistry (including thyroid function), hematology, coagulation, and urinalysis will be summarized by treatment group and presented in tabular and graphic formats where appropriate. Appropriate change from Baseline calculations will be provided to detect any significant changes in laboratory parameters, but no formal statistical tests are planned. Any abnormal finding or clinically significant changes will be captured as AEs.

### 9.3.9.4. Physical Exams

Physical examination findings will be listed for each subject at each assessment period. Clinically significant new findings and adverse changes in physical examination findings will be captured as AEs, therefore eliminating the need to summarize over time.

### 9.3.9.5. C-SSRS

Frequency and severity of suicidal ideation and suicidal behavior as measured by the C-SSRS will be summarized by treatment for each visit.

###  Version: 4.0 – 26 May 2021

### 10. SPONSOR'S AND INVESTIGATOR'S RESPONSIBILITIES

# 10.1. Sponsor's Responsibilities

- The Sponsor and its representatives will undertake the management of the study in compliance with all applicable national and local regulations, as well as the global standard International Council for Harmonisation (ICH) GCP E6 Guideline.
- The Sponsor will ensure that all local regulatory authority requirements of the Sponsor are met before the start of the study including receipt of regulatory authority approvals and/or compliance with the appropriate wait-time required prior to release of the study drug for shipment to the site
- Sponsor ensures that suitable clinical study insurance coverage is in place prior to the start of the study. An insurance certificate will be supplied as needed.
- When required by national law, Sponsor will post appropriate study information on government websites which may include Investigator name and contact information for participating sites.
- Sponsor representatives will make periodic visits to participating sites to review subjects' medical records/source documents, study drug accountability records, and site regulatory documents.

# 10.2. Investigator's Responsibilities

- The Investigator will conduct the study in compliance with all applicable national and local regulations, as well as the global standard ICH GCP E6 Guideline.
- The Investigator agrees to personally oversee the study, delegate study-related tasks to qualified personnel, and meet with Sponsor representatives during on-site visits.
- The Investigator must permit representatives of Sponsor, the IRB and national, local, and foreign regulatory authorities to have direct access to original source documents/medical records, regardless of media, relevant to the study.
- The Investigator is required to maintain all study records according to the ICH GCP E6 Guideline and may not destroy any records until the mandated record retention period is over. Note: Investigators are encouraged to consult with the Sponsor before record destruction to ensure that all retention requirements have been satisfied.


### 11. ETHICS

# 11.1. Ethical Conduct of the Study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICH GCP and applicable regulatory requirements.

### 11.2. Ethics Review

The final study protocol, including the final version of the ICF, must be approved in writing by an IRB as appropriate. The Investigator must submit written approval to the Sponsor before he or she can enroll any subject into the study.

The Investigator is responsible for informing the IRB of any amendment to the protocol in accordance with local requirements. In addition, the IRB must approve all advertising used to recruit subjects for the study. The protocol must be re-approved by the IRB upon receipt of amendments and annually, as local regulations require.

The Investigator is also responsible for providing the IRB with reports of any reportable serious adverse drug reactions from any other study conducted with the study drug. The Sponsor will provide this information to the Investigator.

Progress reports and notifications of serious adverse drug reactions will be provided to the IRB according to local regulations and guidelines.

### 11.3. Written Informed Consent

The Investigator will ensure that the subject is given full and adequate oral and written information about the nature, purpose, possible risk, and benefit of the study. The subject must also be notified that they are free to discontinue from the study at any time. The subject should be given the opportunity to ask questions and allowed time to consider the information provided.

The subject's signed and dated ICF must be obtained before conducting any study procedures.

The Investigator must maintain the original, signed ICF. A copy of the signed ICF must be given to the subject.


### 12. DATA HANDLING AND RECORD KEEPING

# 12.1. Data Collection and Recording

The Investigator or personnel designated by the Investigator will perform primary data collection based on original hospital or clinic records or other source documentation. All required study information must be reported on the appropriate CRF. The study monitor will review CRFs for accuracy and completeness to ensure maximum data integrity. In addition, as the person ultimately responsible for the accuracy of all CRF data, the Investigator will provide endorsement that the data on the CRFs are accurate and complete.

Data processed outside the study site at a central laboratory (e.g., safety lab, ECG, bioanalytical data, etc.) may be transferred electronically.

### 12.2. Retention of Records

The Investigator must maintain all documentation relating to the study for a period of two years after the last marketing application approval, or if not approved, two years following the discontinuance of the study drug for investigation. The Investigator agrees that any study documentation will be promptly disclosed to the Sponsor or the regulatory authority upon request for review.

### 12.3. Protocol Deviations

A protocol deviation is any non-compliance with the clinical study protocol, including compliance requirements and agreements. Examples include an Investigator's decision to deviate from the protocol, a subject's lack of adherence to the protocol, or external/environmental factors (e.g., severe weather or holidays) that change the conduct of a protocol from that which was planned.

The Sponsor will review the protocol deviations that occur during the study. A determination will be made as to which deviations are major – e.g., deviations that impact the study results, data integrity, subject safety, subject consent, or admission criteria.

Further details about the handling of protocol deviations will be included in the Sponsor Study Monitoring and Data Management Plans. The Investigator is responsible for complying with IRB protocol deviation/violation reporting requirements, as applicable.

# **12.4.** Publication Policy

The publication policy is provided in a separate agreement between the Sponsor and those parties contracted to perform services for this study. In summary, all information received and developed in connection with this protocol is considered confidential by the Sponsor. Such information may only be disclosed as deemed appropriate and necessary by the Sponsor. The publication or presentation of data from this study is not allowed without prior agreement with the Sponsor.


# 12.5. Data Quality Assurance

Standard operating procedures (SOPs) are available for all activities performed by the investigational site relevant to the quality of this study. Designated personnel of the investigational site will be responsible for implementing and maintaining quality assurance (QA) and quality control systems to ensure that the study is conducted, and that data are generated, documented and reported in compliance with the study protocol, GCP and Good Laboratory Practice (GLP) requirements, as applicable, as well as applicable regulatory requirements and local laws, rules and regulations relating to the conduct of the clinical study.

CRFs will be 100% source data verified by a Sponsor study monitor against the source notes for identification and clarification of any discrepancies.

The Investigator must make study data accessible to the study monitor, to other authorized representatives of the Sponsor, and to the appropriate regulatory authority inspectors. Audits for QA of the database may be performed according to relevant SOPs from the contract research organization (if applicable) or at the request of the Sponsor.

# 12.6. Data Management

Following are proposed data management activities. A separate Data Management Plan (DMP) will be generated and finalized prior to initiating data management activities. The DMP will specify the details of all data management activities.

Sirtsei Pharmaceuticals, or their designee, will generate the CRFs. An electronic CRF will be used. Sirtsei Pharmaceuticals clinical and safety monitors will review entered data and ensure that they correspond to data kept by the site in source documents. Data management activities such as query management and coding of AE terms will be performed by Sirtsei Pharmaceuticals or their designee.

Each CRF will be reviewed and signed by the PI at each site, as applicable. A detailed DMP will be prepared by the assigned data manager and approved by the Sponsor.

All clinical data will undergo a quality control check prior to clinical database lock. Edit checks are performed for appropriate databases as a validation routine using SAS® or comparable program to check for missing data, data inconsistencies, data ranges, etc. Corrections will be made prior to database lock.

###  Version: 4.0 – 26 May 2021

### 13. LIST OF REFERENCES

### 13.1. Publications Referenced

American Psychiatric Association. Depressive Disorders. In: Diagnostic and Statistical Manual of Mental Disorders. 5th ed. Washington, DC: American Psychiatric Association; 2013. https://dsm-psychiatryonline-

org.ahecproxy.ncahec.net/doi/full/10.1176/appi.books.9780890425596.dsm04

Ionescu DF, Rosenbaum JF, Alpert JE. Pharmacological Approaches to the Challenge of Treatment-Resistant Depression. Dialogues Clin Neurosci. 2015 Jun;17(2):111-26.

Kenward MG, Molenberghs G, Thijs H. Pattern-Mixture Models with Proper Time Dependence. Biometrika, 2003;90(1):53-71.

Lieber A. Major Depression. https://www.psycom.net/depression.central.major.html. Updated January 7, 2020. Accessed July 7, 2020.

Sheehan DV, Lecrubier Y, Harnett-Sheehan K, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar G. The Mini International Neuropsychiatric Interview (M.I.N.I.): The Development and Validation of a Structured Diagnostic Psychiatric Interview. J. Clin Psychiatry, 1998;59(suppl 20): 22-33.

http://www.psychiatrist.com/JCP/article/Pages/1998/v59s20/v59s2005.aspx

# 13.2. Sponsor Documents and Study Reports Referenced

### 13.2.1. Investigator's Brochure

[SP-624 Investigator's Brochure 2020] Investigator's Brochure for SP-624. 2<sup>nd</sup> ed. Sirtsei Pharmaceuticals, Inc.; Release date 11 June 2020.


# 14. APPENDICES


#  Version: 4.0 – 26 May 2021

# APPENDIX A. MONTGOMERY-ASBERG DEPRESSION RATING SCALE


SIGMA 2011, v. 1.2

#### STRUCTURED INTERVIEW GUIDE FOR THE MONTGOMERY AND ASBERG DEPRESSION RATING SCALE (SIGMA)

Janet B.W. Williams, Ph.D. and Kenneth A. Kobak, Ph.D.

INTERVIEWING GUIDELINES: The questions in bold for each item should be asked exactly as written unless the information has been previously obtained, in which case it is appropriate to restate the information for confirmation. Follow-up questions are provided for use when further exploration or additional clarification of symptoms is necessary. The specified questions should be asked until you have enough information to rate the item confidently. In some cases, you may also have to add your own follow-up questions to obtain necessary information. Note that questions in parentheses are optional, for use, for example, if information is unknown. Statements in ALL CAPITALS are interviewer instructions and should not be read to the subject.

RATING GUIDELINES. Ratings should be based on the subject's condition as observed in the past week (past 7 days). As specified in the item descriptions, three of the items, Reduced Sleep, Reduced Appetits, and Inability to Feel, are rated as present only when they reflect a change from before the depression began (EUTHYMIC BASELINE). The interviewer should attempt to identify the most recent 2-month period of non-depressed functioning and use this as a reference point. In some cases, such as when the subject has dysthymia, the referent should be to the last time the subject falt shight (i.e., not depressed or high) for at least a few weeks. When a clear outlymic baseline cannot be established because of chronic depressive symptoms, these three items should be rated as observed over the past 7 days instead of comparing to a previous time point.

This interview guide is based on the Montgomery-Asberg Depression Rating Scale (MADRS) (Montgomery SA, Asberg M: A new depression scale designed to be sensitive to change. <u>Br. J. Prochestry</u>; 1979 134: 382-9). The scale itself has been retained in its original form, except for reversing the order of the first two items. This guide adds interview questions to aid in the assessment and application of the MADRS. Previous versions of this guide appeared in 1988, 1992, 1996, 2005 and 2008.

©2008, 2011 The Royal College of Psychiatrists. The SIGMA may be copied by individual researchers or clinicians for their own use without seeking parmission from the publishers. The scale must be copied in full and all copies must acknowledge the following source: Williams IBW, Kobak KA. Development and reliability of a structured interview guide for the Montgomery-Asberg Depression Rating Scale (SIGMA). Br. J. Psychiatry 2008;192:52-58. Brianne Brown, PsyD, contributed to this revision. Written permission must be obtained from the Royal College of Psychiatrist for copying, distribution to others, for replacion (in print, online or by any other medium), and translations. Scientific correspondence should be addressed to Dr. Janet Williams at journay/@gmail.com. To inform an ongoing survey, researchers and clinicians are asked to notify Dr. Williams of their instantion to use the SIGMA.

SIOMA 2011, v. 1.2

#### STRUCTURED INTERVIEW GUIDE FOR THE MONTGOMERY AND ASBERG DEPRESSION RATING SCALE (SIGMA)

| PISINITIALS: PISID: | TIME BEGAN SIGMA: AM / PM |
|---|---|
| INTERVIEWER: | DATE: |
| OVERVIEW: I'd like to ask you some questions about the past week. How IF OUTPATIENT: Have you been working? (What kind of we IF NOT WORKING OR WORKING LESS, CLARIFY WHY. | r have you been fedling since last (DAY OF WEEK)?<br>rk do you do? Have you been able to work your normal hours?) |
| In the past week, have you been feeling sad or<br>unhappy? (Depressed at all?) IF YES: Can you describe<br>what this has been like for you? (IF UNKNOWN: How<br>had has that been?) | <ol> <li>REPORTED SADNESS. Representing reports of depressed<br/>mood, regardless of whether it is reflected in appearance or not.<br/>Includes low spirits, despondency or the feeling of being beyond<br/>help and without hope. Rute according to intensity, duration, and<br/>the extent to which the mood is reported to be inflammed by<br/>events.</li> </ol> |
| IF DEPRESSED: Does the feeting lift at all if something good happens? How much does your mood lift? Does the feeting ever go savey completely? (How often have you had lift in your mood this week? What things have made you feel better?) | 0 - Occasional aschess in keeping with the circumstances. 1 - 2 - Sad or low but brightens up without difficulty. 3 - 4 - Pervasive feelings of sadness or gloominess. The mood is still influenced by external circumstances. |
| How often did you feel (depressed/OWN BQUIVALENT)<br>this past week? (IF UNCNOWN: How many days this<br>week did you feel that way? How much of each day?) | 5 – 6 – Continuous or unvarying audness, misery, or despondency. |
| In the past week, how have you been fielding about the future? (Have you been discouraged or peasamistic?) What have your thoughts been? How (discouraged or postimistic) have you been? How often have you felt that way? Do you think things will ever get better for you? | |
| ESTABLISH EUTHYMIC BASELINE: When was the last time you were well, not depressed at all, for at least 2 months? | |
| I | 1 |

© 2011, v.1.2, The Royal College of Psychiatrists Confidential and Proprietary 

 Version: 4.0 - 26 May 2021

### SIOMA 2011, v. 1.2

| RATING BASED ON OBSERVATION DURING INTERVIEW AND THE FOLLOWING QUESTIONS. In the past week, do you think you have looked sad or depressed to other people? Did anyone say you looked and or down? How about when you've looked in the mirror; did you look gloomy or depressed? IF YES: How and or depressed do you think you have looked? How much of the time over the past week do you think you have looked? How much of the time over the past week do you think you have looked depressed or down? Has it been hard for you to laugh or smile in the past week? | APPARENT SADNESS. Representing despondency, gloom and despair. (More than just ordinary transient low spirits) reflected in speech, facial expressions, and posture. Rate by depth and inability to brighten up. No nadness The spirits of the spirits |
|---|---|
| Have you felt tense or edgy in the last week? Have you felt anxious or nervous? IF YES: Can you describe what that has been like for you? | <ol> <li>INNER TENSION. Representing feelings of ill-defined<br/>discomfort, edginess, inner turnoil, mental tension mounting to<br/>either partic, dread, or anguish. Rate according to intensity,<br/>frequency, duration and the extent of reassurance called for.</li> </ol> |
| How bad has it been? | 0 - Placid. Only fleeting inner tension. |
| What about feding fearful that something bad is about<br>to happen? | Cocasional feelings of edginess and ill-defined discomfort. 3 – |
| How much of the time have you felt (amious/tense/OWN<br>EQUIVALENT) over the past week? | Continuous feelings of inner tension or intermittent panic<br>which the patient can only master with some difficulty. S – |
| Have you felt panicky in the past week? IF YES: Can<br>you describe this feeling? How often have you felt this<br>way? | 6 - Unrelenting dread or anguish. Overwhelming panic. |
| IF YES TO ANY TENSION SYMPTOM: How hard has it<br>been to control these feelings? (What has it taken to help<br>you feel calmer? Has anything worked to calm you down?) | |
| How has your sleeping been in the last week? (How<br>many hours have you been sleeping, compared to<br>usual?) | <ol> <li>REDUCED SLEEP. Representing the experience of reduced<br/>duration or depth of sleep compared to the subject's own normal<br/>pattern when well.</li> </ol> |
| Have you had trouble falling askep? (How long has it<br>been taking you to fall seleep this past week? How many<br>nights?) | Sleeps as usual. Slight difficulty dropping off to sleep or slightly reduced, light, or fitful sleep. |
| Have you been able to stay askeep through the night?<br>(Have you been waking up at all in the middle of the night?<br>How long does it take you to fall back to sleep? How many<br>nights?) | 3 - Sleep reduced or broken by at least 2 hours. 5 - 6 - Less than 2 or 3 hours sleep. |
| Have there been any mornings this past week when you have awakened earlier than (EUTHYMIC BASELINE)? | |
| IF UNKNOWN: Has your sleeping been restless or<br>disturbed? | |

© 2011, v.1.2, The Royal College of Psychiatrists Confidential and Proprietary 

SIOMA 2011, v. 1.2

 REDUCED APPETITE. Representing the feeling of a loss of appetite compared with when well. Rate by loss of desire for food or the need to force oneself to est. How has your appetite been this past week? (What about compared to your usual appetite?) IF NOT REDUCED: Have you been less interested in food? (How much less?) 0 - Normal or increased appetite.

Does food taste as good as usual? IF LESS: How much less? Does it have any taste at all?

(Have you had to push yourself to est or have other people had to urge you to est?)

- 2 Slightly reduced appetite.
- 4 No appetite. Food is tasteless
- 6 Needs persuasion to est at all.

Have you had trouble concentrating or collecting your thoughts in the past week? (How about at home or at work?) If YES: Can you give me some examples? (Have you been able to concentrate on reading a book or on the computer? Do you need to read things over and over again? Are you able to follow movies or television?)

How often has that happened in the past week? Has this caused any problems for you?

Have you had any trouble following a conversation? (IF YES: How had has that been? How often has that happened this past week?)

NOTE: ALSO CONSIDER BEHAVIOR DURING INTERVIEW.

6. CONCENTRATION DIFFICULTIES. Representing difficulties in collecting one's thoughts mounting to incapaci lack of concentration. Rate according to intensity, frequency, and degree of incapacity produced.

- 0 No difficulties in concentration.
- 2 Occasional difficulties in collecting one's thoughts.
- 4 Difficulties in concentrating and sustaining thought which reduces ability to read or hold a conversation.
- 6 Unable to read or convene without great difficulty

Have you had any trouble getting started at things in the past week? IF YES: What things? How bad has that born? Have you had difficulty getting started at simple routine

everyday things (like getting dressed, brushing your teeth, showering)?

Are you OK once you get started at things or is it still more of an effort to get something done?

Has there been anything that you needed to do that you were unable to do? Have you needed help to do things? IF YES: What things? How often?

Have you done everyday things more slowly than usual? IF YES: Like what, for example? How bad has that been? LASSITUDE. Representing a difficulty getting started, or slowness initiating and performing everyday activities.

- 0 Hardly any difficulty in getting started. No sluggishness.
- 2 Difficulties in starting activities.
- 3 4 Difficulties in simple routine activities, which are carried out with effort.
- 6 Complete lassitude. Unable to do anything without help.

© 2011, v.1.2, The Royal College of Psychiatrists Confidential and Proprietary


SIOMA 2011, v. 1.2

SIOMA 2011, v. 1.2

Have you been less interested in things around you, or in activities you used to enjoy? IF YES: What things? How much less interested in (those things) are you now compared to (EUTHYMC BASELINE)?

What things have you enjoyed this week? How much did you enjoy them?

Has there been any change in your ability to feel emotions in the past week? (Do you feel things less intensely than you used to, things like anger, grief, pleasure?) IF YES: Can you tell me more about that? (IF UNKNOWN: Are you able to feel any emotions at all?)

Have your feelings towards family and friends changed at all since (EUTHYMIC BASELINE)? IF YES: Do you feel less towards them than you used to?

Have you been putting yourself down, or feeling that you're a fallare in some way, ever the past week? (Eave you been blanning yourself for things that you've done, or not done?) IF YES: What have your thoughts been? How often have you felt that way.

In the past week have you been feeling guilty about anything? What about feeling as if you have done something bad or sinful? IF YES: What have your thoughts been? How often have you felt that way?

ALSO CONSIDER RESPONSES TO QUESTIONS ABOUT PESSIMISM FROM ITEM 1.  INABILITY TO FEEL. Representing the subjective experience of reduced interest in the surroundings, or activities that normally give pleasure. The ability to react with adequate emotion to circumstances or people is reduced.

- 0 Normal interest in the surroundings and in other people.
- 2 Reduced shility to enjoy usual interests.
- 4 Loss of interest in the surroundings. Loss of feelings for friends and acquaintances.
- 6 The experience of being emotionally paralyzed, inability to feel anger, grief or pleasure, and a complete or even painful failure to feel for close relatives and friends.

 PESSIMISTIC THOUGHTS. Representing thoughts of guilt, inferiority, self-reproach, sinfulness, remorse, and ruin.

- 0 No pessimistic thoughts.
- 1-
- Pluctuating ideas of failure, self-reproach, or self-depreciation.
- 4 Persistent self-accusations, or definite but still national ideas of
- guilt or sin. Increasingly pessimistic about the future.
- 6 Delusions of ruin, remone, or unredomable sin. Selfaccusations which are about and unshakeable.

This past week, have you felt like life isn't worth living? (IF NO: What about feeling as if you're tired of living?) IF YES: Tell me about that. How often have you felt that way?

This week, have you thought that you would be better off dead? IF YES: Tell me about that. How often have you felt that way?

Have you had thoughts of hurting or even killing yourself this past week? IF YES: What have you thought abous? How often have you had these thoughts? How long have they lasted? Have you actually made plans? IF YES: What are these plans? Have you made any reparamions to carry out these plans? (Have you told anyone about it?)

10. SUICIDAL THOUGHTS. Representing the feeling that life is not worth living, that a natural death would be welcome, saticidal thoughts, and preparation for suicide. Suicidal attempts should not in themselves influence this rating.

- 0 Enjoys life or takes it as it comes
- 2 Weary of life. Only fleeting suicidal thoughts.
- 4- Probably better off dead. Suicidal thoughts are common, and suicide is considered so a possible solution, but without specific plans or intention.
- 5 Explicit plans for suicide when there is an opportunity. Active preparations for suicide.

| TIME ENDED SIGMA: | AM/PM |
|--------------------------|-------|
| TOTAL MADRS SCALE SCORE: | |

# APPENDIX B. CLINICAL GLOBAL IMPRESSION – SEVERITY

# Clinical Global Impression - Severity (CGI-S)

Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?

| 0 = Not assessed |
|-----------------------------|
| 1 = Normal, not at all ill |
| 2 = Borderline mentally ill |

- 3 = Mildly ill
- 4 = Moderately ill
- 5 = Markedly ill
- 6 =Severely ill
- 7 = Among the most extremely ill patients


#  Version: 4.0 – 26 May 2021

# APPENDIX C. 17-ITEM HAMILTON DEPRESSION RATING SCALE


SIGH-D-17 Feb. 2013

# STRUCTURED INTERVIEW GUIDE FOR THE HAMILTON DEPRESSION RATING SCALE - 17 ITEM VERSION (SIGH-D-17)

Janet B.W. Williams, PhD

#### INTERVIEWER

The first question for each item should be asked exactly as written. Often this question will elicit enough information about the severity and frequency of a symptom for you to rate the item with confidence. Follow-up questions are provided for use when further exploration or additional clarification of symptoms is necessary. The specified questions should be asked until you have enough information to rate the item confidently. In some cases, you may also have to add your own follow-up questions to obtain necessary information. You should ask for examples for any symptoms acknowledged as present (e.g., "Can you give me an example of that?"). For some of the HAM-D items, you may find you have already asked about some of the symptoms (for a previous item). You do not need to repeat questions about these symptoms unless you need additional information to rate their severity.

<u>Time period</u>. The interview questions indicate that the ratings should be based on the subject's condition in the past week.

Administration method. This version includes interview questions to help the clinician rate psychomotor agitation and psychomotor retardation, when the interview is administered by telephone. Several research studies have demonstrated that depression scale scores are equivalent whether the scale is administered face-to-face, by telephone, or by video (Williams JBW and Kobak KA: Development and Reliability of a Structured Interview Guide for the Montgomery-Asberg Depression Rating Scale. Br J Psychiatry 192, 52-59, 2008; Kobak KA: A comparison of face-to-face and remote administration of the Hamilton Depression Rating Scale via videoconferencing. J Telemed Telecare 10, 231-235, 2004).

Referent of "usual" or "normal" condition. In the HAM-D, most items are rated positive only if they represent a change from usual functioning. For this reason, several of the interview questions in the HAM-D refer to the subject's usual or normal functioning. The referent should be to the last time they felt okay (i.e., not depressed or high and normal interest in things) for at least two months. When no clear euthymic baseline can be established, one should rate symptomatic behavior as one sees it, even if it is not a change from the subject's usual dysphoric

This instrument provides an interview guide for the Hamilton Depression Scale (Hamilton, Max.: A rating scale for depression, <u>J. Neurol. Neurosurp. Psychiat.</u> 23.56-61, 1960). The anchor point descriptions for all items except Helpiesoness, indepleasness, and Worthlessness, with very inmormodications, have been taken from the ECDEU. Assessment Manual (Guy, Williams, have been taken from the ECDEU. Assessment Manual for <u>Psychopharmacology</u>, Revised 1976, DHEW Publication No. (ADM) 76-398). The loss of weight ten has been simplified to eliminate the section for radings by ward staff. A reliability study of the SIGH-ID (interview guide for the HAM-ID alone) was published in the <u>Archives of General Psychiatry</u> (1988;45-742-747). Additional designators were added in perentheses to the anchor points by Kobaku, Lipstiz and Williams to further standardize rating and the province of the standardize rating and the standardize rating

For further information and permission to use or translate the SIGH-D, contact Mapi Research Trust (Internet: https://eprovide.mapi-trust.org).


Version 2013.1 ⊚ Janet B.W. Williams, 1988. All Rights Reserved SIGH-D\_Utiled States/English – Original version SIGH-D\_AUZO\_eng-USon

SIGH-D-17 Feb. 2013 STRUCTURED INTERVIEW GUIDE FOR THE HAMILTON DEPRESSION RATING SCALE - 17 ITEM VERSION (SIGH-D-17) SUBJECT'S INITIALS: \_\_\_\_\_ TIME BEGAN SIGH-D: \_\_\_\_ INTERVIEWER: \_\_\_\_\_\_ DATE: \_\_\_\_/ \_\_\_/ OVERVIEW: I'd like to ask you some questions about the past week. How have you been feeling since last (DAY OF WEEK)? IF OUTPATIENT: Have you been working? IF NOT: Why not? 1. DEPRESSED MOOD (sadness, hopeless, What's your mood been like this past week helpless, worthless) (compared to when you feel okay)? Have you been feeling down or depressed? 0 Absent Indicated only on questioning (occasional, mild IF YES: Can you describe what this feeling has been depression) like for you? How bad is the feeling? Spontaneously reported verbally (persistent, mild to moderate depression) Does the feeling lift at all if something good happens? Communicated non-verbally, i.e., facial expression, posture, voice, tendency to weep How are you feeling about the future? (persistent, moderate to severe depression) VIRTUALLY ONLY those feeling states reported IF UNKNOWN: Have you been feeling discouraged in spontaneous verbal and non-verbal or pessimistic? communication (persistent, very severe depression, with extreme hopelessness or IF YES: What have your thoughts been? tearfulness) In the last week, how often have you felt (OWN EQUIVALENT FOR DEPRESSED MOOD)? On how many days? For how long each day? Have you been crying at all? How often? IF SCORED 1-4 ABOVE, ASK: How long have you been feeling this way (OWN EQUIVALENT FOR DEPRESSED MOOD)?


© Janet B. W. Williams, 1988. All Rights Reserved SIGH-D – United States/English – Original version SIGH-D\_AUZ0\_eng-USon


#### SIGH-D-17 Feb. 2013

| week (when not at work)? | 0 | No difficulty |
|---|---|---|
| Have you felt interested in doing (THOSE THINGS),<br>or do you feel you have to push yourself to do them?<br>How much less interested in these things have you<br>been this past week compared to when you're not | 1 | Thoughts and feelings of incapacity, fatigue<br>or weakness related to activities, work or<br>hobbies (mild reduction in interest or<br>pleasure; no clear impairment in functioning) |
| over this pass week compared to when you're not depressed? How hard to do you have to push yourself to do them? Have you stopped doing anything you used to do? (What about hobbles?) IF YES: Why? | 2 | Loss of interest in activity, hobbies or work-<br>by direct report of the patient or indirect in<br>listlessness, indecision and vacilitation (feels<br>he has to push self to work or activities)<br>(clear reduction in interest, pleasure or<br>functioning) |
| About how many hours a day do you spend doing things that interest you? Is there anything you look forward to? IF WORKING (IN OR OUT OF THE HOME): Have | 3 | Decrease in actual time spent in activities or decrease in productivity. In hosp., pl. spends less than 3 hrs./day in activities (hospital job or hobbles) exclusive of ward chores (profound reduction in interest, pleasure, or functioning) |
| you been able to get as much (work) done as you<br>usually do?<br>How much less productive or efficient are you<br>compared to before you were depressed? | 4 | Stopped working because of present illness.<br>In hospital, no activities except ward chores,<br>or fails to perform ward chores unassisted<br>(unable to work or fulfill primary role because<br>of illness, and total loss of interest) |


Version 2013.1 ⊕ Janet B. W. Williams, 1988. All Rights Reserved SIGH-D – United States/English – Original version SIGH-D\_AU20\_eng-USon

#### SIGH-D-17 Feb. 2013

| During the past week, have you been waking up in the middle of the night? IF YES: Do you get out | 4. IN | SOMNIA MIDDLE: |
|---|---|---|
| of bed? What do you do? (Only go to the | 0 | No difficulty |
| bathroom?)<br>When you get back in bed, are you able to fall right | 1 | Complains of being restless and disturbed during the night (or occasional difficulty, i.e., 2-3 nights, 30 minutes or more) |
| back asleep? How long does it take you to fall back<br>asleep?<br>Do you wake up more than once during the night? | 2 | Waking during the night; any getting out of bed (except to void) (often, i.e., 4 or more nights of difficulty, 30 minutes or more) |
| (IF YES: How long does it take for you to fall back to sleep each time?) | | The state of the s |
| Have you felt your sleeping has been restless or<br>disturbed some nights? | | |
| How many nights this week have you had that kind of trouble? | | |
| What time have you been waking up in the morning for the last time, this past week? | 5. IN | SOMNIA LATE (TERMINAL INSOMNIA): |
| | 0 | No difficulty |
| IF EARLY: Is that with an alarm clock, or do you just<br>wake up yourself? What time do you usually wake up<br>(that is, when you feel well)? | 1 | Waking in early hours of morning but goes back to sleep (occasional, i.e., 2-3 nights difficulty) |
| How marry mornings this past week have you<br>awakened early? | 2 | Unable to fall asleep again if gets out of bed (often, i.e., 4 or more nights difficulty) |
| Sometimes, along with depression or anxiety, people might lose interest in sex. This week, how has your interest in sex been? (I'm not asking about actual sexual activity, but about your interest in | | ENITAL SYMPTOMS (such as loss of libido, strual disturbances): Absent |
| sex.) | 1 | Mild (somewhat less interest than usual) |
| Has there been any change in your interest in sex<br>(from when you were feeling OK)? | 2 | Severe (a lot less interest than usual) |
| IF YES: How much less interest do you have compared to when you're not depressed? (Is it a little | | |


7. SOMATIC SYMPTOMS GASTROINTESTINAL:

Loss of appetite but eating without encouragement (appetite somewhat less

significantly less than usual)

Difficulty eating without urging (appetite

than usual)

2

© Janet B.W. Williams, 1988. All Rights Reserved SIGH-D – United States/English – Original version SIGH-D\_AUZ0\_eng-USori

How has your appetite been this past week? (What about compared to your usual appetite?)

Have other people had to urge you to eat? (Have you skipped meals?)

IF LESS: How much less than usual?

Have you had to force yourself to eat?


#### SIGH-D-17 Feb. 2013

| Have you lost any weight since this (DEPRESSION) began? | 8. LC | DSS OF WEIGHT |
|---|---|---|
| | Rate | by history: |
| IF YES: Did you lose any weight this last week? (Was it because of feeling depressed or down?) How | _ | I |
| much did you lose? | 0 | No weight loss |
| | 1 | Probable weight loss due to current<br>depression |
| IF NOT SURE: Do you think your clothes are any | 1 2 | Definite (according to patient) weight loss |
| looser on you? | ^ | due to depression |
| FOLLOW-UP: Have you gained any of the weight back? IF YES: How much? | | |
| How has ∨our energy been this past week? | 9. 50 | DMATIC SYMPTOMS GENERAL: |
| , | | |
| IF LOW ENERGY: Have you felt tired? (How much of the time? How bad has it been?) | 0 | None |
| , | 1 | Heaviness in limbs, back, or head.<br>Backaches, muscle aches. Loss of energy |
| This week, have you had any aches or pains? (What | Ш | and fatigability (somewhat less energy than |
| about backaches or muscle aches?) (How much of the time? How bad has it been?) | II | usual; mild, intermittent loss of energy or |
| | - | muscle aches/heaviness) |
| Have you felt any heaviness in your limbs, back, or<br>head? | 2 | Any clear-cut symptoms (persistent,<br>significant loss of energy or muscle<br>aches/heaviness) |
| Have you been putting yourself down this past<br>week, feeling you've done things wrong, or let | 10. F | EELINGS OF GUILT: |
| others down? | 0 | Absent |
| IF YES: What have your thoughts been? | 1 | Self-reproach; feels he has let people down |
| | 2 | Ideas of guilt or rumination over past errors |
| Have you been feeling guilty about anything that | | or sinful deeds (feelings of guilt, remorse or |
| you've done or not done? | II 🖵 | shame) |
| IF YES: What have your thoughts been? | 3 | Present illness is a punishment; delusions<br>of guilt (severe, pervasive feelings of guilt) |
| What about things that happened a long time ago? | 4 | Hears accusatory or denunciatory voices |
| venial about things that happened a long time ago? | 11 | and/or experiences threatening visual |
| Have you thought that you've brought (THIS | | hallucinations |
| DEPRESSION) on yourself in some way? | | |

 © Janet B.W. Williams, 1988. All Rights Reserved SIGH-0 – United States/English – Original version sith-0\_AUZ\_paydon SIGH-D-17 Feb. 2013

| This past week, have you had thoughts that life is not worth living? | 11.5 | UICIDE: |
|---|---|---|
| • | 0 | Absent |
| What about thinking you'd be better off dead? | 1 | Feels life is not worth living |
| Have you had thoughts of hurting or killing yourself? | 2 | Wishes he were dead or any thoughts of<br>possible death to self |
| IF YES: What have you thought about? Have you | 3 | Suicidal ideas or gesture |
| actually done anything to hurt yourself? | 4 | Attempts at suicide |
| Have you been feeling anxious or tense this past week? | 12. A | NXIETY PSYCHIC: |
| IF YES: Is this more than is normal for you? | 0 | No difficulty |
| Have you been feeling irritable this past week? | 1 | Subjective tension and irritability (mild, occasional) |
| (IF YES): Can you give me some example? How<br>bad has it been? | 2 | Worrying about minor matters (moderate, causes some distress) |
| Have you been worrying a lot about little things, | 3 | Apprehensive attitude apparent in face or<br>speech (severe; significant impairment in<br>functioning due to anxiety) |
| things you don't ordinarily worry about?<br>IF YES: Like what, for example? | 4 | Fears expressed without questioning<br>(symptoms incapacitating) |
| How about worrying about big problems more than you need to? | | |
| you need to: | | |
| How much of the time has that happened this week? | | |


Pai © Janet B. W. Williams, 1988, All Rights Reserved SIGH-D – United States/English – Original version SIGH-D\_WZD\_eng-Uson


#### SIGH-D-17 Feb. 2013

| Tell me if you've had any of the following physical symptoms in the past week. (READ LIST) FOR EACH SX ACKNOWLEDGED AS PRESENT: How much has (THE SX) been bothering you this past week? [How bad has if gotten? How much of the time, or how often, have you had it? Did (the symptom) interfere at all with your functioning or your susual activities?] | ANXIETY SOMATIC (physiologic concomitants of anxiety, such as GI - dry mouth, gas, indigestion, diarrhea, stomach cramps, belching CV - heart palpitations, headaches Resp - hyperventilating, sighing Urinary frequency Sweating): |
|---|---|
| | 0 Not present |
| NOTE: DO NOT RATE SXS THAT ARE CLEARLY<br>RELATED TO A DOCUMENTED PHYSICAL<br>CONDITION. | 1 Mild (symptom(s) present only infrequently, no impairment, minimal distress) |
| CONDITION. | 2 Moderate (symptom(s) more persistent, or<br>some interference with usual activities,<br>moderate distress) |
| | 3 Severe (significant impairment in functioning) |
| | 4 Incapacitating |
| In the last week, how much have your thoughts<br>been focused on your physical health or how | 14. HYPOCHONDRIASIS: |
| been focused on your physical health or how | |
| been focused on your physical health or how<br>your body is working (compared to your normal<br>thinking)? (Have you worried a lot about being or<br>becoming physically iii? Have you really been<br>preoccupied with this?) | Not present Self-absorption (bodily) (some inappropriate worry about his/her health OR slightly concerned despite reassurance) |
| been focused on your physical health or how<br>your body is working (compared to your normal<br>thinking)? (Have you worried a lot about being or<br>becoming physically ill? Have you really been<br>precoccupied with this?) Have you worried a lot that you have a specific<br>medical illness? | Not present Self-absorption (bodily) (some inappropriate worry about his/her health OR |
| been focused on your physical health or how<br>your body is working (compared to your normal<br>thinking)? (Have you worried a lot about being or<br>becoming physically sli? Have you really been<br>preoccupied with this?) Have you worried a lot that you have a specific | Not present Self-absorption (bodily) (some inappropriate worry about his/her health OR slightly concerned despite reassurance) Preoccupation with health (often has excessive worries about his/her health OR definitely concerned has specific liliness |
| been focused on your physical health or how your body is working (compared to your normal thinking)? (Have you worried a lot about being or becoming physically lil? Have you really been preoccupied with this?) Have you worried a lot that you have a specific medical illness? Do you complain much about how you feel physically? Have you seen a doctor about these problems? | Not present Self-absorption (bodily) (some inappropriate worry about his/her health OR slightly concerned despite reassurance) Preoccupation with health (often has excessive worries about his/her health OR definitely concerned has specific illiness despite medical reassurance) Frequent complaints, requests for help, etc. (is certain there is a physical problem which the doctors cannot confirm, exaggerated or unrealistic concerns about body and physical health) Hypochondriacal delusions |
| been focused on your physical health or how your body is working (compared to your normal thinking)? (Have you worried a lot about being or been decided with this?) Have you worried a lot that you have a specific medical illness? Do you complain much about how you feel physically? Have you seen a doctor about these problems? FYES: What did the doctor say? | Not present Self-absorption (bodily) (some inappropriate worry about his/her health OR slightly concerned despler reassurance) Preoccupation with health (often has excessive worries about his/her health OR definitely concerned has specific illness despler medical reassurance) Frequent complaints, requests for help, etc. (is certain there is a physical problem which the doctors cannot confirm; exaggerated or unrealistic concerns about body and physical health) |
| been focused on your physical health or how your body is working (compared to your normal thinking)? (Have you worried a lot about being or been decided with this?) Have you worried a lot that you have a specific medical illness? Do you complain much about how you feel physically? Have you seen a doctor about these problems? FYES: What did the doctor say? | Not present Self-absorption (bodily) (some inappropriate worry about his/her health OR slightly concerned despite reassurance) Preoccupation with health (often has excessive worries about his/her health OR definitely concerned has specific illiness despite medical reassurance) Frequent complaints, requests for help, etc. (is certain there is a physical problem which the doctors cannot confirm, exaggerated or unrealistic concerns about body and physical health) Hypochondriacal delusions |
| been focused on your physical health or how your body is working (compared to your normal thinking)? (Have you worried a lot about being or becoming physically ill? Have you really been preoccupied with this?) Have you worried a lot that you have a specific medical illness? Do you complain much about how you feel physically? Have you seen a doctor about these problems? | Not present Self-absorption (bodily) (some inappropriate worry about his/her health OR slightly concerned despite reassurance) Preoccupation with health (often has excessive worries about his/her health OR definitely concerned has specific liliness despite medical reassurance) Frequent complaints, requests for help, etc. (is certain there is a physical problem which the doctors cannot confirm; exaggerated or unrealistic concerns about body and physical health) Hypochondriacal delusions 15. INSIGHT: |


Pai ⊕ Janet B. W. Williams, 1988. All Rights Reserved SIGH-D – United States/English – Original version SIGH-D, 2022, proju/Sai SIGH-D-17 Feb. 2013

| RATING BASED ON OBSERVATION DURING INTERVIEW | 16. AGITATION: |
|---|---|
| | 0 None |
| IF INTERVIEWING BY PHONE: | 1 Fidgetiness (slight agitation or mild restlessness) |
| During this interview have you been fidgeting a lot or<br>moving around a lot in your chair? | 2 Playing with hands, hair, etc. (moderate to marked restlessness or agitation) |
| Have you had trouble sitting still? | <li>Moving about, can't sit still (cannot remain seated)</li> |
| Have you been shaking your legs or playing with your<br>hair or your hands? | Hand-wringing, nail biting, hair-pulling, biting of lips (interview cannot be conducted; severe agitation) |
| | 17. RETARDATION (slowness of thought and speed impaired ability to concentrate; decreased motor activity): |
| RATING BASED ON OBSERVATION DURING INTERVIEW IF INTERVIEWING BY PHONE: | impaired ability to concentrate; decreased motor activity): |
| INTERVIEW IF INTERVIEWING BY PHONE: During this interview have you been moving slowly, reacting slowly, or speaking more slowly than usual | impaired ability to concentrate; decreased motor activity): 0 |
| INTERVIEW IF INTERVIEWING BY PHONE: During this interview have you been moving slowly, | impaired ability to concentrate; decreased motor activity): 0 Normal speech and thought |
| INTERVIEW IF INTERVIEWING BY PHONE: During this interview have you been moving slowly, reacting slowly, or speaking more slowly than usual | impaired ability to concentrate; decreased motor activity): 0 |

| TIME ENDED SIGH-D-17: | AM / PM |
|-----------------------|---------|
| TOTAL HAM-D-17 SCORE: | |


Pai © Janet B. W. Williams, 1988, All Rights Reserved SIGH-D – United States/English – Original version SIGH-D\_WZD\_eng-Uson


# APPENDIX D. SHEEHAN DISABILITY SCALE


# SHEEHAN DISABILITY SCALE

### A BRIEF, PATIENT RATED, MEASURE OF DISABILITY AND IMPAIRMENT

Please mark ONE circle for each scale.

## In the past (timeframe):







### DAYS LOST

On how many days in the last week did your symptoms cause you to miss school or work or leave you unable to carry out your normal daily responsibilities?

### DAYS UNDERPRODUCTIVE

On how many days in the last week did you feel so impaired by your symptoms, that even though you went to school or work or had other daily responsibilities, your productivity was reduced? \_\_\_\_\_

Copyright 1963, 2010, 2012 David V. Sheehan. All rights reserved.

Permissions: davidvsheehan@gmail.com

# APPENDIX E. THE QUICK INVENTORY OF DEPRESSIVE SYMPTOMOLOGY – SELF REPORT


QIDS-SR16 - United States/English - Original version QISARNS, ALC 1, exp. (Sec. 4)

##  Version: 4.0 – 26 May 2021

#### SELF-REPORT QUICK INVENTORY OF DEPRESSIVE SYMPTOMATOLOGY (QIDS-SRIA) 11. View of Myself: 14. Energy Level: 0 I see myself as equally worthwhile and 0 There is no change in my usual level of deserving as other people. I am more self-blaming than usual. energy. I get tired more easily than usual. 2 I have to make a big effort to start or finish my usual daily activities (for example, shopping, homework, cooking or going to work). 3 I really cannot carry out most of my usual daily 2 I largely believe that I cause problems for Please circle the one response to each item that best describes you for the past seven days. I think almost constantly about major and minor defects in myself. 1. Falling Asleep: 6. Decreased Appetite: activities because I just don't have the energy. 0 I never take longer than 30 minutes to fall There is no change in my usual appetite. 12. Thoughts of Death or Suicide I eat somewhat less often or lesser amounts of 15. Feeling slowed down: 1 I take at least 30 minutes to fall asleep, less food than usual. 2 I eat much less than usual and only with 0 I do not think of suicide or death. than half the time. I feel that life is empty or wonder if it's worth 0 I think, speak, and move at my usual rate of 2 I take at least 30 minutes to fall asleep, more personal effort. 3 I rarely eat within a 24-hour period, and only living. I think of suicide or death several times a week than half the time. I take more than 60 minutes to fall asleep. I find that my thinking is slowed down or my with extreme personal effort or when others persuade me to eat. for several minutes. 3 I think of suicide or death several times a day voice sounds dull or flat. 2 It takes me several seconds to respond to more than half the time. in some detail, or I have made specific plans for suicide or have actually tried to take my life. most questions and I'm sure my thinking is 2. Sleep During the Night: 7. Increased Appetite I am often unable to respond to questions I do not wake up at night. There is no change from my usual appetite. I feel a need to eat more frequently than usual. 13. General Interest: without extreme effort. I have a restless, light sleep with a few brief awakenings each night. I wake up at least once a night, but I go back I regularly eat more often and/or greater amounts of food than usual. 0 There is no change from usual in how 16. Feeling restless: interested I am in other people or activities. to sleep easily. 3 I awaken more than once a night and stay awake for 20 minutes or more, more than half I feel driven to overeat both at mealtime and I do not feel restless. I'm often fidgety, wringing my hands, or need to shift how I am sitting. I notice that I am less interested in people or I find I have interest in only one or two of my formerly pursued activities I have impulses to move about and am guite 3 I have virtually no interest in formerly pursued restless. At times, I am unable to stay seated and need 3. Waking Up Too Early: 8. Decreased Weight (Within the Last Two Weeks): to page around. I have not had a change in my weight. I feel as if I've had a slight weight loss. 0 Most of the time, I awaken no more than 30 minutes before I need to get up. More than half the time, I awaken more than I have lost 2 pounds or more. 30 minutes before I need to get up. 2 I almost always awaken at least one hour or so 3 I have lost 5 pounds or more To Score: before I need to, but I go back to sleep 3 I awaken at least one hour before I need to. 9. Increased Weight (Within the Last Two Weeks): Enter the highest score on any 1 of the 4 sleep items (1-4) and can't go back to sleep. I have not had a change in my weight. I feel as if I've had a slight weight gain. Item 5 4. Sleeping Too Much: I have gained 2 pounds or more. I have gained 5 pounds or more. Enter the highest score on any 1 appetite/ 0 I sleep no longer than 7-8 hours/night, without napping during the day. 1 I sleep no longer than 10 hours in a 24-hour period including naps. Item 10 I sleep no longer than 12 hours in a 24-hour Concentration/Decision Making: 6. Item 12 eriod including naps. I sleep longer than 12 hours in a 24-hour period including naps. 0 There is no change in my usual capacity to 7. Item 13 concentrate or make decisions. 8. Item 14 I occasionally feel indecisive or find that my Feeling 8ad: attention wanders. Most of the time, I struggle to focus my 9. Enter the highest score on either of the 2 psychomotor items (15 and 16) I do not feel sad attention or to make decisions. I feel sad less than half the time. I cannot concentrate well enough to read or TOTAL SCORE (Range 0-27) I feel sad more than half the time cannot make even minor decisions. I feel sad nearly all of the time. © 1986, 2000 UT Southwestern Medical Center, Dallar © 1986, 2000 UT Southwestern Medical Center, Dallar

QIDS-SR16 - United States/English - Original version QIDS-SR16\_ALD (\_eg/Chiri.sea

APPENDIX F. QUALITY OF LIFE ENJOYMENT AND SATISFACTION

QUESTIONNAIRE – SHORT FORM


| Name: | Date: |
|-------|-------|

# Quality of Life Enjoyment and Satisfaction Questionnaire – Short Form (Q-LES-Q-SF)

Taking everything into consideration, during the past week how satisfied have you been with your.......

| | Very Poor | Poor | Fair | Good | Very Good |
|---|---|---|---|---|---|
| physical health? | 1 | 2 | 3 | 4 | 5 |
| mood? | 1 | 2 | 3 | 4 | 5 |
| work? | 1 | 2 | 3 | 4 | 5 |
| household activities? | 1 | 2 | 3 | 4 | 5 |
| social relationships? | 1 | 2 | 3 | 4 | 5 |
| family relationships? | 1 | 2 | 3 | 4 | 5 |
| leisure time activities? | 1 | 2 | 3 | 4 | 5 |
| ability to function in daily life? | 1 | 2 | 3 | 4 | 5 |
| sexual drive, interest and/or performance?* | 1 | 2 | 3 | 4 | 5 |
| economic status? | 1 | 2 | 3 | 4 | 5 |
| living/housing situation?* | 1 | 2 | 3 | 4 | 5 |
| ability to get around physically<br>without feeling dizzy or unsteady<br>or falling?* | 1 | 2 | 3 | 4 | 5 |
| your vision in terms of ability to do work or hobbies?* | 1 | 2 | 3 | 4 | 5 |
| overall sense of well being? | 1 | 2 | 3 | 4 | 5 |
| medication? (If not taking any,<br>check hereand leave item<br>blank.) | 1 | 2 | 3 | 4 | 5 |
| How would you rate your overall life<br>satisfaction and contentment during<br>the past week? | 1 | 2 | 3 | 4 | 5 |

<sup>\*</sup>If satisfaction is very poor, poor or fair on these items, please UNDERLINE the factor(s) associated with a lack of satisfaction.

#  Version: 4.0 – 26 May 2021

# APPENDIX G. COLUMBIA – SUICIDE SEVERITY RATING SCALE – BASELINE/SCREENING VERSION

# RATING SCALE (C-SSRS)

Baseline/Screening Version

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

### Disdaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbio-Suidde Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suiddal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide History Form</u>, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstom B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardtand Evaluation in Clinical Practice, pp. 103 - 130, 2003)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hystene, Inc.

| SUICIDAL IDEATION | | | | | |
|---|---|---|---|---|---|
| Ada promiser ( em l 1. gland) ary magazine, processor in "Abdella" Biberian" combine. Pello mercur se<br>anniber ( la ") | | | Lifetime: Time<br>Ha'She Felt<br>Mest Subtidal | | Past<br>Months |
| <ol> <li>Wish to be Dead<br/>Subject endorse: Songita about a wish to be dead or not dive supresen<br/>Have you wished you wave dead or wished you sould go to deep and o</li> </ol> | | Y** | No. | Y** | No. |
| Eye, describe 2. Non-Specific Active Suicidal Thoughts Control one | No. 1 - 1 | Yes | No | Yes | No |
| 2. Non-Operation Active Substitute I Dissigned<br>Committee and Committee a | meaned peind. | • | • | • | |
| 3. Active Strictfal Idention with Any Methods (Not Plan)<br>Subject software thoughts of mixids and has frought of at least one on<br>specific plan with time, plan or southed details worked not (e.g., though<br>who small are, "Tempt and the contract of the contract of<br>and "small every in though with it." Maw you been distribute about how you might do this? | thed during the assessment period. This is different than a | Y== | | <b>:</b> | No |
| Nye, destile | | | | L | |
| 4. Active Statistian Ideation with Some Intent to Act, with<br>Aution sainful foundate of it ling consell on adapted open having as<br>thoughts had a defensly will not do acquiting about them.<br>Here you had those thoughts and had come intention of acting on the<br>Hym, dwarfer. | one intint to act on such thousand, as opposed to Taxon | Y= | No. | - | No |
| <ol> <li>Active Suicidal Ideation with Specific Plan and Intent<br/>Thought of tiling mount with death of Jon Fully or partially writed<br/>How you started to work out or work of out the datable of how to hill y<br/>if you, donot be</li> </ol> | d out and exhiped has some intent to early it me.<br>covered? Do you become to early out this plane? | Yes | <u>*</u> | - | No |
| INTENSITY OF IDEATION The following features should be rated with respect to the most | severe type of ideation (i.e., 1-5 from above, with I being | | | _ | |
| The following features should be raued with respect to the most the least severe and 5 being the most severe). Ask about time h <u>126stime</u> - Mont Severe Montion: "Specific) | | M<br>Ser | ost<br>esre | Mc<br>Sev | |
| The following features should be raused with respect to the most the least source and 5 being the most source). Ask about time he Lifetime. Most Source Mention: Type (3.1) Type (3.1) | wishe was feeling the most suicidal. | | | | |
| The following features should be rande with respect to the most the least source and 5 being the most source). Ask about time he lifetime. Most Severe Mention: That X Mooths - Most Severe Mention: Type 6-3: Frequency How many times have you had these thoughts? (1) Less than once a week. (2) Once a week. (3) 2.5 times in we | Withouse finding the most suicidal Benights of Matte | | | | |
| The following features should be rand with respect to the most the least source and 5 being the most source). Aid about time he Likeline.— Most Servere Meastlen: Type 10:10 Past X Months - Most Servere Meastlen: Type 10:10 Frequency How many times have you had these thoughts? (1) Less then come a west. (2) Come a west. (3) 2.5 times in we Describe. Phen you have the thoughts how long do they less? (2) Less then 1 bourbone of the time (3) Less than 1 bourbone of the time (3) Less than 1 bourbone of the time | Withouse finding the most suicidal Benights of Matte | Ser | | | |
| The following features should be rande with respect to the most be least as most award, Ask about time in Lifetime. Most Severe Montion: That X Months - Most Severe Montion: That X Months - Most Severe Idention: Trequency How many times have you had these thoughts? (I) Less than ones a week. (I) however the part of the Phenopeur Severe Idention: The property of the severe Identified the Severe Identified to the | Therefore of Market Description of Market (6) Delty or almost delty (3) Many times each day (6) Ad househood of day (5) More than 1 househows for or confinence (6) Ad househood of day (5) More than 1 househows for confinence (6) Consumers from the second tool (6) Consumers fr | Ser | - | | |
| The following features should be rande with respect to the most the least source and 5 being the most source). Ask about time he lifeting. Most Severe Mention: "Spirit (3). Past X Mooths - Most Severe Mention: "Spirit (3). Frequency How many times have you had those thoughts? (1) Less than ones work (2) You as work (3) 2.5 times in we Darration Pleasing few seconds or minutes. (2) Less than 1 best interes of the first (3) Early shift of shielding about hilling yourself or want (3) Early shift of southed thoughts (3) Can control thoughts with little difficulty Determine the density of consomining anishted? (4) Determine the fluid yourself you from attempting minisht (5) Determine the finishty output you from attempting minisht | Thereights of Status Thereights of Status Thereights of Status Thereights of Status Thereights of Status (6) this bears to dely (5) Many times each day (6) this horselment of day (5) this horselment of day (6) this horselment of day (6) this horselment of the status (6) this horselment of the status (6) the status of the status (6) the status of the status (7) this has to extend the status (8) the status of details a, pain of details) - that stayped your from wanting to (8) Determent status is the status of the stay you (9) Determent status is the stay you (1) Determent status is the stay you (1) Determent status is the stay you (1) Determent status is the stay you | Ser | - | | |
| The following features should be rande with respect to the most be least as some and 3 being the most awardy. Ask about time is 11deline. Most Severe Mention: That X Mooths - Most Severe Mention: Type (3.1) Frequency Blow many times have you had these thoughts? (1) Least has most work. (2) Cone is work. (3) 2.5 times in me Darration. Plant you have the thoughts have long do they last? (3) I who have the thoughts have long do they last? (3) I show has it to do time. (3) 1.4 houses it to time. (3) 1.4 houses it to do time. (3) I show has to do time to time. (3) 1.4 houses it to do time. (4) 1.4 houses it to do time. (5) 1.4 houses the distinct of time. (6) 1.4 h | Securities of Harden Description of Harden Description of Harden (4) Act homeostered of day (5) More than 1 homeostered or continuous ting to dis if your want to? (6) Con-montal troughs with a lot of difficulty (7) Unders to control troughs (8) On motival troughs with a lot of difficulty (9) Con-motival troughs with a lot of difficulty (9) Understood troughs (9) Description and strong or your forms wanting to (9) Con-motival troughs with a lot of pro- (9) Con-motival distribution of the pro- (9) Con-motival definitely did not steep you (9) Con-motival definitely steep yourself? What it to cond the pains motibart? Or both? | Ser | | | |

90


Version: 4.0 - 26 May 2021

| SUICIDAL BEHAVIOR (Oxeck all that apply, so long as these are separate events; must ask about all types) | | Lifetime | Past<br>Years |
|---|---|---|---|
| Actual Attempt | | Yes No | Yes No |
| A potentially self-injurious act committed with at least some wish to dis, as a result of act Debavior was in part thou | | | 00 |
| count! Inter does not have to be 100%. If there is any intercidenies to dis associated with the set, then it can be at | | | |
| attempt. There does not have to be any injury or have, just the potential for injury or have. If person pulls<br>mouth but gue in broken so no injury results, this is considered an attempt. | patter agent from the | ı | |
| Inferring Intent: From if an individual denies intent/wish to dis, it may be inferred clinically from the behavior or circ | constances. For example, a | | |
| highly lithal act that is clearly not an accident so no other intent hat mixide can be inflored (e.g., guestot to head, ju-<br>high flooristory). Also, if someone denies intent to die, but they thought that what they did could be lathel, intent ma- | mping from window of a | | |
| Have you made a suicide attempt? | y in immedia | | |
| Have you done anything to have yourself? | | Total # of | Total # of |
| Have you done anything dangerous where you could have died? What did you do? | | Attacopts | Attainets |
| Did you as a way to end your life? | | I — | l — |
| Did you want to die (even a little) when you? | | | |
| Were you trying to end your life when you? Or Did you think it was possible you could have died from? | | | |
| | and the same | | |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relic<br>get sympathy, or get something due to happen)? (hill-bijurious behavior without misidal issue)<br>it you, describe | ere serena, jest neser, | | |
| If you, describe: | | Yes No | Yes No |
| | | 0.0 | 0 0 |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | Ves No | Yes No |
| Interrupted Attempt: When the person is interrupted (by an outside obcumetance) from starting the potentially self-injurious act (if not for | that actual attenut would | | |
| have convered. | | | 0 0 |
| Overdoo: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt attempt. Shooting: Person has gon pointed toward self, gon in taken army by someone else, or is somehow prevented | cother than an interrupted | | |
| they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and t | aben down from ledge. | | |
| Hanging: Penns has notes around seek but has not yet started to hang - is stopped from doing so. Heat there been a time when you started to do nomething to end your life but someone or nometh | | Total Fof | Total # of |
| Hai there been a time when you started to do something to end your life but someone or someth | ing stopped you before | interrupted | interrupted |
| you actually did anything? You deaths | | | |
| 2 yes, describe | | _ | |
| Aborted Attempt: | | Yes No | Yes No |
| When person begins to take stape toward making a minide attempt, but stope themselves before they actually have an<br>destructive behavior. Examples are similar to interrupted attempts, except that the individual stope binchered? inste | | | |
| exactly de. | and it comes and describe | | |
| Has there been a time when you started to do something to try to end your life but you stopped y | ourself before you | Total # of | Total # of |
| actually did anything? | | aborted | aboted |
| If you, describe | | ı — | l |
| Preparatory Acts or Behavior: | | | |
| Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization | or thought, such as | | W W |
| assembling a specific method (e.g., harbourne, product or property for the state of | ng things away, writing a | Yes No | Yes No |
| Here you taken any steps towards making a suicide attempt or preparing to kill yourself (such a | e collection pills. | | |
| matter a man all the code of the common and the control of the code of | • | | |
| genting a gain, group transactor awdy or revising a national money? 2 yes, describe: | | | |
| Suicidal Behavior:<br>Suicidal behavior was present during the assessment period? | | Yes No | Yes No |
| Answer for Actual Attempts Only | | fost Lethal | NATION. |
| | | | Manuel<br>Mari |
| Actual Letta By Medical Danage. | Rear Code | Roter Code | Reter Code |
| No physical damage or very minor physical damage (e.g., surface contains). Minor statical damage (e.g., lateratic specific for damage laterate militalistics provide). | | | |
| <ol> <li>Minor physical damage (e.g., lethargic speech; first-dagme horse; milt blacking; spraine).</li> <li>Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-de</li> </ol> | gree | | |
| bons, bleeding of major vessel). | | | |
| <ol> <li>Moderately serves physical damage, medical hospitalization and likely intensive care required (e.g., constons wit<br/>intact, third-degree horse less than 20% of body, extensive blood less but can recover, major fractures).</li> </ol> | The Personal Property of the Personal Property | | |
| 4. Severe situated damage, made of homitalization with intensive care required (e.g., constone without reflexes; this | rd-degree | | |
| burns over 20% of body, extensive blood loss with unstable vital eight, major damage to a vital area). | | | |
| 5. Duch Peterdal Lethnity: Only Assess If Actual Lethnity=0 | | | |
| Petrodial Lithelity: Only Assesse If Actual Lithelity-9<br>Likely inhality of actual attempt if no medical damage (the following examples, while having no actual medical dam | age, had Ener Code | Enter Code | Enter Code |
| potential for very serious lethality: put gue in mouth and pulled the trigger but gue fails to fire so no medical damage. | Laying | | |
| on train tracks with oncoming train but pulled away before run over). | | | |
| 6 = Tedantion not likely to result in injury | | | |
| 1 = Relativitor likely to menit in injury but not likely to cause death 2 = Relativitor likely to menit in death despite available medical care | | | |
| 2 * Heliantor Many to most in death daught available medical care C 2008 Research Provideline for Medic Hygiens, Inc. C 2008 Research Provideline for Medic Hygiens, Inc. | | | Page 2 of 2 |
| Comp control (Venice 1/400) | | | 100 2 01 2 |

# APPENDIX H. COLUMBIA – SUICIDE SEVERITY RATING SCALE –

SINCE LAST VISIT VERSION


# RATING SCALE (C-SSRS)

Since Last Visit

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.;
Burke, A.; Oquendo, M.; Mann, J.

#### Disdaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbio-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide History Form</u> developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD). New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk (factors for suicidal behavior utility and limitations of research instruments. In M.B. First [Ed.] Standardzad Evaluation in Clinical Practica, pp. 103-130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerki@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc.

C-SSRS Since Last Visit - United States/English - Mapi.

| SUICIDAL IDEATION | | | |
|---|---|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suic | tidal Behavior "section. If the answer to question 2 is "yes", | Since | Last |
| ask questions 3, 4 and 5. If the answer to question 1 and/or 2 | ts "yes", complete "Intensity of Ideation" section below. | Vi | nit |
| 1. With to be Dead | | | |
| Subject endorses thoughts about a wish to be dead or not allies asymory, or | with to full salesp and not wake up. | Yes | No |
| Subject endorses thoughts about a wish to be dead or not allow asymous, or wish to fall aslessp and not wake up. How you wished you were dead or wished you could go to slessy and not walks up? | | | |
| If you, describe: | | | |
| 2. Non-Specific Active Suicidal Thoughts | | | |
| General non-specific thoughts of wasting to end one's life/commit mixide) | (e.g., "I've thought about killing myself") without thoughts of ways to kill | | No |
| onself associated methods, intent, or plan during the assumment period. How you extendly had any thoughts of killing yourself? | | - | |
| If you, describe: | | | |
| 3. Active Suicidal Ideation with Any Methods (Not Plan) wi | thout Intent to Act | _ | |
| Subject endorses thoughts of minide and has thought of at least one method | during the assessment period. This is different than a specific plan with time, | Yes | No |
| place or method details worked out (e.g., thought of method to kill self but o | during the assessment period. This is different than a specific plan with time, not a specific plan). Includes person who would say, "I thought about taking as | l 🗖 | |
| overdose but I never made a specific plan as to when, where or how I would | f actually do itand I would never go through with it". | ı – | _ |
| Have you been thinking about how you might do this? | | l | |
| If you, describe: | | | |
| 4. Active Suicidal Ideation with Some Intent to Act, without | | 20.0 | - |
| | intent to act on such thoughts, as opposed to "I have the thoughts hat I definitely | | No |
| will not do anything about them".<br>Here you had these thoughts and had some intention of acting on them? | | | |
| If you, describe: | | | |
| 5. Active Suicidal Ideation with Specific Plan and Intent | | Yes | No |
| Thoughts of killing consolf with details of plan fally or partially worked out<br>How you started to work out or worked out the details of how to hill yours | and subject has some extent to carry it out. | | |
| ,,,,,,, | 4. 1. / 2. 2 | - | |
| If you, describe: | | | |
| INTENSITY OF IDEATION | | | |
| ETIETO DE IDELITOR | | | |
| | ore type of ideation (i.e., i-5 from above, with 1 being the least severe | | |
| | are type of Iduation (i.e., 1-3 from above, with 1 being the least severe | M | and . |
| The following flutures should be rated with respect to the most are<br>and 3 being the most severe). | are type of kination (i.e., i-5 from above, with $l$ being the least severe | | cet |
| The following features should be rated with respect to the most are<br>and 3 being the most arvers). Most Severe Ideation: | | | |
| The following flustures should be rated with respect to the most are and 5 being the most areas). Most Severe Ideation: Type # (1-5) | ere type of ideation (i.e., i-3 from above, with I being the least severe Description of Ideation | | |
| The following features should be rated with respect to the most are and 5 being the most arrens). Most Severe Ideation: Type 6 (1-5) Frequency | | | |
| The following flustures should be rated with respect to the most are and 5 being the most areas). Most Severe Ideation: Type # (1-5) | Description of Ideation | | |
| The following features should be rated with respect to the most area and 3 being the most areas). Most Severe Ideation: Type # (1-5) Frequency (b) Less than most a well: (2) Once a weel; (2) 2-5 time in weel; Duration | Description of Ideation | | |
| The following features should be rated with respect to the most are and 3 being the most arrent). Most Severe Ideation: Type 8 (1-5) Frequency How many times have you had these thoughts? (3) Last bean case a well. (2) Once a well. (3) 2-5 time in well. When you have the thoughts how long do they last? | Description of Ideation (6) Daily or almost daily (5) Many times such day | | |
| The following features should be rated with respect to the most area and 3 being the most areas). Most Severe Ideation: Type 8 (1-5) Frequency (1) Law then coop a week (2) Once a week (3) 2-5 times in week Duration When you have the thoughth for long do they leat? (3) Rotting—the woods or minute. | Description of Idention (4) Daily or almost daily (5) Many time each day (6) 4-8 house/most of day | | |
| The following features should be rated with respect to the most are and 3 being the most are send 3 being the most are send 3 being the most are send 3 being the most are send 4 feat for the send 5 features. Type # (3-5) Frequency How many times here you had these thoughts? (3) Loss the mose a walk. (2) Conca wask. (3) 2-5 times in wask. Duration When you have the thoughts how long do they last? (3) Rating -few seconds or minutes. (2) Loss then I bourtones of the time. | Description of Ideation (6) Daily or almost daily (5) Many times such day | | |
| The following features should be rated with respect to the most area and 3 being the most areas). Most Severe Ideation: Type 8 (1-5) Frequency (1) Law then coop a week (2) Once a week (3) 2-5 times in week Duration When you have the thoughth for long do they leat? (3) Rotting—the woods or minute. | Description of Idention (4) Daily or almost daily (5) Many time each day (6) 4-8 house/most of day | | |
| The following features should be rated with respect to the most are and 3 being the most areas). Most Severe Ideation: Type # (1-5) Frequency (b) Less than none a welt. (2) Once a west. (2) 2-5 times in west Duration When you have the thought how long do they least? (1) Floring-low accords or minutes. (2) Less then I hourisons of the time. (3) Less then I hourisons of the time. (3) Less than I hourisons of the time. (4) Less than I hourisons of the time. (5) Less than I hourisons of the time. | Description of Idention (4) Daily or almost daily (3) Many times each day (4) 44 house/most of day (5) Man than 8 house/penisted or continuous to dat if your want to? | | |
| The following features should be rated with respect to the most are and 3 being the most areas). Most Severe Ideation: Type # (1-5) Frequency (b) Less than none a welt. (2) Once a west. (2) 2-5 times in west Duration When you have the thought how long do they least? (1) Floring-low accords or minutes. (2) Less then I hourisons of the time. (3) Less then I hourisons of the time. (3) Less than I hourisons of the time. (4) Less than I hourisons of the time. (5) Less than I hourisons of the time. | Description of Idention (4) Daily or almost daily (3) Many times each day (4) 44 house/most of day (5) Man than 8 house/penisted or continuous to dat if your want to? | | |
| The following features should be rated with respect to the most area and 3 being the most areas). Most Severe libration: Type 8 (1-5) Frequency (b) Law then coop a week (2) Once a week (2) 2-5 times in week Duration When you have the thoughth four long do they leat? (1) Hosting—low acoust or minima. (2) Law then I bourbone of the time (3) Law then I bourbone of the time (3) Law then I bourbone of the time (4) Law then I bourbone of the time (5) Law then I bourbone of the time (6) Law then I bourbone of the time (7) Law then I bourbone of the time (8) Law then I bourbone of the time (9) Law then I bourbone of the time (10) Law then I bourbone of the time (11) Law the I bourbone of the time (12) Law then I bourbone of the time (3) Law then I bourbone of the time (4) Law the content thoughts with the difficulty | Description of Idention (4) Daily or almost daily (3) Many from each day (4) 44 home/most of day (5) More than 8 home/penistent or continuous for die if your want for? (6) On control thoughts with a lot of difficulty (5) Dailelet to control thoughts | | |
| The following features should be rated with respect to the most are and 3 being the most areas). Most Severe Ideation: Type # (1-5) Frequency (b) Less than none a welt. (2) Once a west. (2) 2-5 times in west Duration When you have the thought how long do they least? (1) Floring-low accords or minutes. (2) Less then I hourisons of the time. (3) Less then I hourisons of the time. (3) Less than I hourisons of the time. (4) Less than I hourisons of the time. (5) Less than I hourisons of the time. | Description of Idention (4) Daily or almost daily (3) Many times each day (4) 44 house/most of day (5) Man than 8 house/penisted or continuous to dat if your want to? | | |
| The following features should be rated with respect to the most area and 3 being the most areas). Most Server libration: Type 8 (1-5) Frequency. Type 8 (1-5) Frequency. (b) Lass than coop a week. (2) Once a week. (2) 2-5 times in week Duration When you have the thoughth flow long do they leat? (1) Bosting—free mosted or minutes. (2) Lass then I hourisons of the time. (3) Last have I have been a minute. (b) Last you have the thoughth flow long do they leat? (c) Eastly all less to convent or minute. (c) Last you not a stop thinking about killing yourself or wanting. (i) Eastly alls to convert thoughts. (i) Can control thoughts with some lifficulty. (i) Can control thoughts with some lifficulty. Determined. | Description of Idention (4) Daily or almost daily (3) Many times each day (4) 4-4 homes/most of day (5) More than 8 homes/penistent or continuous for die if your want for? (6) One most of thoughts with a lot of difficulty (5) Daile to control thoughts (9) Done not attauge to control thoughts | | |
| The following funtures should be rated with respect to the most are and 5 desig the most arread. Most Server Identice: Type 8 (3-5) Frequency How many times have you had these thoughts? (1) Last has none a wak. (2) Once a week. (3) 2-5 times in week. Duration When you have the thoughts how long do they lest? (1) Roting -few encode or minutes. (2) Loss the 1 hourisms of the time. (3) Last has 1 hourisms of the time. (4) Early list to control thoughts. (5) Early list to control thoughts. (5) Early list to control thoughts. (5) Control thoughts of the control thoughts of control thoughts of control thoughts of thoughts. (5) Early lists to control thoughts. (5) Early lists to control thoughts. (5) Early lists to control thoughts. (5) Control control thoughts with some fiftiently. Determined. Are there things - suprone or ampthing (e.g., family, religion, potengals). | Description of Ideation (4) Daily or almost daily (3) Many from each day (4) 44 home/most of day (5) More than 8 home/penisted or continuous (to die if your want to? (4) One control thoughts with a lot of difficulty (5) Dailes to control thoughts (9) Dailes to control thoughts size of death) - that stopped you from wanting to die or acting on | | |
| The following features should be rated with respect to the most sensed 3 being the most sensed 5 being the most sensed 5 being the most sensed 5 being the most sensed 60 being the following times have you had these thoughts? (1) It has then one a welk (2) Ones a welk (3) 2-5 time in welk Duration When you have the thoughts how long do they lead? (3) Floring - fees encode or minima (3) Len then 1 bourbons of the time (3) Len then 1 bourbons of the time (3) Len's yellow to differ the fees (4) Len's the 1 bourbons of the time (3) Len's yellow to differ the fees (4) Len's yellow to differ the fees (5) Len's yellow to consider the galaxy (5) Concentration the galaxy (6) Concentration the galaxy of the galaxy o | Description of Idention (4) Daily or almost daily (5) Many times each day (4) 44 house/most of day (5) Mars than 8 house/particular or conditiones to die if you want to? (6) On control daughts with a lot of difficulty (6) Does not attempt to control thoughts (6) Does not attempt to control thoughts (6) Determine most likely 66 not stay you (6) Determine most likely 66 not stay you | | |
| The following features should be rated with respect to the most sensed 3 being the most sensed 5 being the most sensed 5 being the most sensed 5 being the most sensed 60 being the following times have you had these thoughts? (1) It has then one a welk (2) Ones a welk (3) 2-5 time in welk Duration When you have the thoughts how long do they lead? (3) Floring - fees encode or minima (3) Len then 1 bourbons of the time (3) Len then 1 bourbons of the time (3) Len's yellow to differ the fees (4) Len's the 1 bourbons of the time (3) Len's yellow to differ the fees (4) Len's yellow to differ the fees (5) Len's yellow to consider the galaxy (5) Concentration the galaxy (6) Concentration the galaxy of the galaxy o | Description of Idention (4) Daily or almost daily (5) Many times each day (4) 44 house/most of day (5) Mars than 8 house/particular or conditiones to die if you want to? (6) On control daughts with a lot of difficulty (6) Does not attempt to control thoughts (6) Does not attempt to control thoughts (6) Determine most likely 66 not stay you (6) Determine most likely 66 not stay you | | |
| The following funtures should be rated with respect to the most are and 5 desig the most arread. Most Server Identice: Type 8 (3-5) Frequency How many times have you had these thoughts? (1) Last has none a wak. (2) Once a week. (3) 2-5 times in week. Duration When you have the thoughts how long do they lest? (1) Roting -few encode or minutes. (2) Loss the 1 hourisms of the time. (3) Last has 1 hourisms of the time. (4) Early list to control thoughts. (5) Early list to control thoughts. (5) Early list to control thoughts. (5) Control thoughts of the control thoughts of control thoughts of control thoughts of thoughts. (5) Early lists to control thoughts. (5) Early lists to control thoughts. (5) Early lists to control thoughts. (5) Control control thoughts with some fiftiently. Determined. Are there things - suprone or ampthing (e.g., family, religion, potengals). | Description of Ideation (4) Daily or almost daily (3) Many from each day (4) 44 home/most of day (5) More than 8 home/penisted or continuous (to die if your want to? (4) One control thoughts with a lot of difficulty (5) Dailes to control thoughts (9) Dailes to control thoughts size of death) - that stopped you from wanting to die or acting on | | |
| The following finances should be rated with respect to the most sense and 3 being the most sense. Most Severe Ideation: Type 8 (1-5) Frequency: (1) Last than one a week. (2) Ones a week. (3) 2-5 time in week Duration When you have the thoughts how long do they last? (3) Rosting-free associal or minima. (3) Last than 1 houstones of the time. (3) Last than 1 houstones of the time. (4) Last than 1 houstones of the time. (5) Last than 1 houstones of the time. (6) Last than 1 houstones of the time. (7) Last than 1 houstones of the time. (8) Last than 1 houstones of the time. (9) Last than 1 houstones of the time. (1) Early side to most of the time. (1) Early side to most of the side. (2) One content doughts with some difficulty. (2) One content doughts with some difficulty. (3) Determine defaulty stoped you from attempting mixide. (1) Determine the delayed supped you. (2) Determine the delayed supped you. (3) Thouston that delayed supped you. (4) Thouston that delayed supped you. (5) Thouston that delayed supped you. (6) Thinking about wanting. | Description of Ideation (4) Daily or almost daily (5) Many times each day (4) 4-8 home/most of day (5) More than 8 home/particular or condinuous to die if your want to? (6) The control thoughts with a lot of difficulty (5) Under to control thoughts (6) Date not attempt to control thoughts (6) Date not attempt to thought some of entirely on the control thoughts (6) Datements and finitely did not stop you (5) Datements and distributed the control thoughts (6) Datements and finitely did not stop you (6) Datements definitely did not stop you (6) Datements definitely did not stop you (6) Datements definitely did not stop you (6) Datements definitely did not stop you (6) Datements definitely did not stop you (7) Datements definitely did not stop you (8) Datements definitely did not stop you (9) Datements definitely did not stop you (9) Datements definitely did not stop you | | |
| The following funtures should be rated with respect to the most are and 3 being the most are sent 3 being the most are sent 3 being the most are sent as the following following | Description of Ideation (4) Daily or almost daily (5) Many times each day (4) 4-8 home/most of day (5) More than 8 home/particular or condinuous to die if your want to? (6) The control thoughts with a lot of difficulty (5) Under to control thoughts (6) Date not attempt to control thoughts (6) Date not attempt to thought some of entirely on the control thoughts (6) Datements and finitely did not stop you (5) Datements and distributed the control thoughts (6) Datements and finitely did not stop you (6) Datements definitely did not stop you (6) Datements definitely did not stop you (6) Datements definitely did not stop you (6) Datements definitely did not stop you (6) Datements definitely did not stop you (7) Datements definitely did not stop you (8) Datements definitely did not stop you (9) Datements definitely did not stop you (9) Datements definitely did not stop you | | |
| The following features should be rated with respect to the most sensed 3 being the most served. Most Severe Ideation: Type 8 (1-5) Frequency: (1) Last than one a welk. (2) Once a welk. (2) 2-5 time in welk Duration When you have the thoughts how long do they lead? (3) Floring-free mosted or minima. (2) Last than 1 hourisons of the time. (3) Last than 1 hourisons of the time. (3) Last than 1 hourisons of the time. (4) Last than 1 hourisons of the time. (5) Last than 1 hourisons of the time. (6) Last than 1 hourisons of the time. (7) Last than 1 hourisons of the time. (8) Last than 1 hourisons of the time. (9) Last than 1 hourisons of the time. (1) Last than 1 hourisons of the time. (1) Last than 1 hourisons of the time. (1) Last than 1 hourisons of the time. (2) Concentration than the time time of time time, religion, p. thoughts of committing raticular? (1) Intervent and delable support you from attempting mixide. (1) Intervent that there will enough you. Reasons for Ideation. Reasons for Ideation. What not of greatment all you have for thinking about wanting you were feeling (in other worth you couldn't go on living well recomes or a reaction from others? Or books? | Description of Idention (4) Daily or almost daily (5) Many lines each day (4) 44 house/most of day (5) Man than Ehouse/particular or condimens to die if you want to? (6) The control thoughts with a lot of difficulty (5) Theirs to control thoughts (6) Their is to control thoughts (6) Date and ethnical to control thoughts (6) Date and ethnical to control thoughts (6) Dateman and likely did not stop you (5) Dateman definitely did not stop you (6) Dateman definitely did not stop you (6) Date and applically did not stop you (7) Date and applically did not stop you (8) Date and application of the pain or stop the way to this pain or how you were feelingly or was it to get attention. | | |
| The following features should be rated with respect to the most sensed 3 being the most served. Most Severe Ideation: Type 8 (1-5) Frequency: (1) Last than one a welk. (2) Once a welk. (2) 2-5 time in welk Duration When you have the thoughts how long do they lead? (3) Floring-free mosted or minima. (2) Last than 1 hourisons of the time. (3) Last than 1 hourisons of the time. (3) Last than 1 hourisons of the time. (4) Last than 1 hourisons of the time. (5) Last than 1 hourisons of the time. (6) Last than 1 hourisons of the time. (7) Last than 1 hourisons of the time. (8) Last than 1 hourisons of the time. (9) Last than 1 hourisons of the time. (1) Last than 1 hourisons of the time. (1) Last than 1 hourisons of the time. (1) Last than 1 hourisons of the time. (2) Concentration than the time time of time time, religion, p. thoughts of committing raticular? (1) Intervent and delable support you from attempting mixide. (1) Intervent that there will enough you. Reasons for Ideation. Reasons for Ideation. What not of greatment all you have for thinking about wanting you were feeling (in other worth you couldn't go on living well recomes or a reaction from others? Or books? | Description of Idention (4) Daily or almost daily (5) Many times each day (6) 4-8 house/most of day (7) Many times each day (8) 6-8 house/most of day (9) Man than I house/moistent or continuous to dair if your want to? (6) Das sound thoughts with a lot of difficulty (5) Table to control thoughts (5) Table to thoughts (6) Date and thoughts with a lot of difficulty (6) Date and many to control thoughts with of death) - that stopped you from wanting to die or acting on (6) Datemonts defaultely did not stop you (9) Datemonts defaultely did not stop you (9) Datemonts day for the position or stop the way to this pain or know you were feelingly or was it to get attention, (6) Matrix to and or stop the pain (you couldn't you on living with the pain (or | | |
| The following features should be rated with respect to the most sensed 3 being the most served. Most Severe Ideation: Type 8 (1-5) Frequency (b) Last than one a welk. (2) Once a welk. (3) 2-5 time in welk Duration When you have the thoughts how long do they lead? (1) Floring-free accords or minima. (2) Last than 1 hourisons of the time. (2) Last than 1 hourisons of the time. (2) Last than 1 hourisons of the time. (3) Last yellow to conside the spile. (4) Early allow to only the spile. (5) Early allow to only the spile. (6) Can control thoughts with some difficulty. (7) Can control thoughts with some difficulty. (8) Can control thoughts with some difficulty. (9) Can control thoughts with some difficulty. Determine the spile of the spile of the spile of conveniency excited? (1) Determine whethy the spile of the spile of the spile. (1) Determine whethy the spile of the spi | Description of Ideation (4) Daily or sinuest daily (3) Many firms each day (4) 44 house/most of day (5) More than 8 house/penisted or continuous (4) 64 house/most of day (5) Dailes to most of house/most one (6) Dailes control changins with a lot of difficulty (5) Dailes to most of house/most of difficulty (5) Dailes to most of house/most of difficulty (6) Dailes not stating to most of display (6) Dailes not stating to most of day from wanting to die or acting on (6) Dailes not defailedly did not stay you (5) Dailes not defailedly did not stay you (6) Dailes not defailedly did not stay you (7) Dailes not defailedly did not stay you (8) Most not defailedly did not stay you (9) Most not defailedly did not stay you (9) Most not defailedly did not stay you (9) Most not defailedly on the your were feelingly or was it to get aftersion. (4) Mostly to not or stay the pain (you couldn't go on Eving with the pain or how you were feelingly | | |
| The following funtures should be rated with respect to the most sensed? Seting the most served. Most Server Ideation: Type 8 (1-5) Frequency (1) Last than one a welk. (2) Ones a welk. (3) 2-5 time in welk Duration When you have the thoughts how long do they last? (1) Floring-free mosteds or minima. (2) Last than 1 hourisms of the time. (2) Last than 1 hourisms of the time. (2) Last than 1 hourisms of the time. (3) Last than 1 hourisms of the time. (4) Last than 1 hourisms of the time. (5) Last than 1 hourisms of the time. (6) Last than 1 hourisms of the time. (7) Last than 1 hourisms of the time. (8) Last than 1 hourisms of the time. (9) Last than 1 hourisms of the time. (10) Last than 1 hourisms of the time. (11) Last than 1 hourisms of the time. (12) Concentration than the time time of time time, religion, p. thoughts of committee quicker? (1) Datarwaits solubly copyed you (2) Bastowns solubly copyed you (3) Bastown that determine includes you from strongting mixide. (3) Bastown that determine includes you for the strongton of the time of the time to the plant of the time you have for thinking about wanting you were feeling (in other worth you couldn't go on living well revenues or a reaction from others? Or books? | Description of Idention (4) Daily or almost daily (5) Many times each day (6) 4-8 house/most of day (7) Many times each day (8) 6-8 house/most of day (9) Man than I house/moistent or continuous to dair if your want to? (6) Das sound thoughts with a lot of difficulty (5) Table to control thoughts (5) Table to thoughts (6) Date and thoughts with a lot of difficulty (6) Date and many to control thoughts with of death) - that stopped you from wanting to die or acting on (6) Datemonts defaultely did not stop you (9) Datemonts defaultely did not stop you (9) Datemonts day for the position or stop the way to this pain or know you were feelingly or was it to get attention, (6) Matrix to and or stop the pain (you couldn't you on living with the pain (or | | |

Research Foundation for Mental Hygimus, Inc. C 398.3—Since Last Visit (Venico 14 609)


| SUICIDAL BEHAVIOR | |
|---|---|
| (Check all that apply, so long as these are separate events; must ask about all types) | Last Visit |
| Actual Attempt: A potentially self-injection act committed with at least some wish to dis, as a result of act. Behavior was in part thought of as method to bill seased! Intest does not have to be 100%. If there is any intestibilisis to dis associated with the act, then it can be considered an actual existin strategy. There does not have to be any interpret a harm to be any interpret harm to be any interpret a harm to be any interpret and are to be any interpret and are part and a potential for highey or harm. If passes pulls trigger while gas is in most but gas is broken so so highey counts, this is considered as attempt. | Yes No |
| Informing Inters: From if an individual domine interstwish to tile, it may be informed clinically from the behavior or circumstances. For example, a highly behavior at leastly yet an excitate a non-order interst to mission on both informed (e.g., general to be bed, jumping from window of a high filter/strony). Also, if someone domine inters to tile, but they founder that what they fild could be lethed, intere may be informed. Here you readed a mission of surprise property. Here you readed a mission of surprise for the property of the pr | |
| Hare you done anything to harm yourself? Hare you done anything dangerous where you could have died? | Total # of<br>Attempts |
| What did you do? Did you are a way to end your life? Did you went to die (even a little) when you ? | - |
| Were you trying to end your life when you 7 Or Did you think it was possible you could have died from 7 | |
| Or did you do it purely for other remota / without ANY intention of killing yourself (like to relieve stress, feel better, get sympathy, or get constituing also to happen? (Solf-injuina Valuries without advisal insus) ## 194, Manifes | |
| Has subject ensured in Non-Sokidal Self-Inturious Behavior? | Yes No |
| Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have convend. | Yes No |
| Overflow: Penne has pills in hard but is emport from ingusting. Once they inquire my pills, this become an actuary traffer than a timerquist attempt. Interior: Penne has gas pointed record off, gas in their army by assessment also, or is assessed prevented from pringing trigger. Once they pill their gas, ease if the gas falls to fire, it is an attempt. Imaging: Penne is goined to jump, is grabbed and takes down from Indge, Hanging Penne has access around such better as one extends to have, it adopted from following the contract to have, or adopted from following the contract to have, or adopted from following the contract to have, or adopted from following the contract to have, or adopted from following the contract to have present the contract to the con | |
| Has there been a time when you started to do something to end your life but someone or something stopped you before you actually did anything? If yo, double. | Total # of<br>interrupted |
| Aborted Attempt: Who peans hope to take steps troud making a mixide attempt, but steps fameables below they actually have suggested in any self-destructive belavior. Framples are similar to interrupted attempt, except that the individual steps limitated (I being stopped by something site. Has there been a time when you started to do nomething to try to end your life but you stopped yourself before you actually did amphing? If you, describe: | Yes No |
| Preparatory Acts or Behavior: Acts or population towark imminently saking a minite attauge. This can include anything beyond a verbalization or thought, each as assembling a quotific method, e.g., bejong pilit, purchasing a gua) or proposing the ear's death by minite (e.g., ghing things enery, writing a minite sate). Here you taken any steps towards making a minite attempt or preparing to kill yourself (such as collecting pills, getting a guan, giving valuables away or writing a minite note)? Eyes, describe: | Yes No |
| Suicidal Behavior:<br>Suicidal behavior was present during the assessment period? | Yes No |
| Suicide: | Yes No |
| Answer for Actual Attempts Only | Most Lethal<br>Attaunt<br>Date |
| Actual Lethality/Medical Damage: 0. No physical desage or very minor physical damage (e.g., surface scenthes). | Steer Code |
| <ol> <li>More physical damage (e.g., inflampic speech, first-degree burne; solid blanding species).</li> <li>Mohente physical damage, medical attaction sended in ag, consenies but temps, somewhat responsive, second-degree burne; blanding of major vessel).</li> <li>Mohentarity servers physical damage, medical benjakitation and Blady intensive cares required (e.g., consates with reflexus intext; third-degree burne last that 20°th of logic extensive blood less but can envery major financies.</li> <li>Sower physical damage, medical benjakitation with intensive care required (e.g., consutes without reflexus; third-degree burne over 20% of body; extensive blood loss but can envery major financies.</li> <li>Sower physical damage, medical benjakitation with intensive can required (e.g., consutes without reflexus; third-degree burne over 20% of body; extensive blood loss with untable vide degree, major demage to vital about 10°th.</li> </ol> | _ |
| 5. Duch Potential Lethality: Only Answer if Actual Lethality=0 | Enter Code |
| Likely ideality of actual extensit if no medical damage (the following examples, while lawing no actual medical damage, had possed for very serious<br>lethelity; put gas in meeth and pulled the trigger but gas fails to five so no medical damage, keying on train trades with encoming train but pulled every<br>lettless ma coust). | |
| 0 = Balanties and Hady to result in injury 1 = Balanties Hady to result in injury but not Hady to cause duath 2 = Balanties Hady to result in death duajob available multical case | |

© 2008 Research Foundation for Meetal Hygima, Inc

C-898.9—Since Last Visit (Venion 1/1409)

Page 2 of 2
